



## STATISTICAL ANALYSIS PLAN

Project Number: GLPG0634

Study Number: GLPG0634-CL-309

Study Title: Combined Phase 3, Double-blind, Randomized, Placebo-Controlled

Studies Evaluating the Efficacy and Safety of Filgotinib in the

Induction and Maintenance of Remission in Subjects with Moderately

to Severely Active Crohn's Disease

Development Phase: 3

Status: Final

Version: 2.0 Date: 15-Jan-2023

EudraCT: 2016-001367-36 IND: 02914561

Sponsor: Galapagos NV, Generaal De

Wittelaan L11 A3, 2800

Mechelen, Belgium

Biostatistician: PPD

Medical Leader: PPD

#### **Confidentiality Statement**

The information contained in this document is privileged and confidential. It is the property of Galapagos NV and may not be used, disclosed, reproduced or otherwise disseminated within your organization or communicated to any third parties without the express written authorization of Galapagos NV.

## **TABLE OF CONTENTS**

| TA | BLE OF | F CONTENTS | 2 |
|---|---|---|---|
| LIS | T OF I | N-TEXT TABLES | 4 |
| | | N-TEXT FIGURES | |
| | | BBREVIATIONS | |
| PH | ARMA | COKINETIC ABBREVIATIONS | 8 |
| 1. | INTR | ODUCTION | 9 |
| | 1.1. | Study Objectives | 9 |
| | | 1.1.1. Primary Objectives | |
| | | 1.1.2. Secondary Objectives | 10 |
| | | CCI | |
| | 1.2. | Study Design | |
| | | 1.2.1. Induction Studies (Cohort A and B) | |
| | | 1.2.2. Maintenance Study | |
| | | 1.2.4. Schedule of Assessments. | |
| | 1.3. | Sample Size and Power | |
| 2 | | OF PLANNED ANALYSIS | |
| 2. | TYPE | | |
| | 2.1. | Data Monitoring Committee (DMC) Analyses | 20 |
| | | 2.1.1. Safety Analyses | 20 |
| | 2.2 | 2.1.2. Cohorts A and B End-of-Induction Analysis | |
| | 2.2. | Final Analysis | 20 |
| 3. | GENI | GENERAL CONSIDERATIONS FOR DATA ANALYSES | |
| | 3.1. | Analysis Sets | 21 |
| | 3.1. | 3.1.1. All Randomized Analysis Sets | |
| | | 3.1.2. Full Analysis Sets. | |
| | | 3.1.3. Safety Analysis Sets | |
| | | 3.1.4. Pharmacokinetic Analysis Sets | |
| | | 3.1.5. Pharmacokinetic Substudy Analysis Sets | 22 |
| | | CCI | |
| | 3.2. | Subject Grouping | |
| | 3.3. | Strata and Covariates | |
| | 3.4.<br>3.5. | J U 1 | |
| | 3.3. | 3.5.1. EU-Specific | |
| | | 3.5.2. Other (non-EU) | |
| | 3.6. | Missing Data and Outliers | |
| | | 3.6.1. Missing Data | |
| | | 3.6.2. Outliers | |
| | 3.7. | Data Handling Conventions and Transformations | 32 |
| | 3.8. | Analysis Visit Windows | 34 |
| | | 3.8.1. Definitions | |
| | | 3.8.2. Analysis Visit Windows | 35 |
| | | 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit | 20 |
| | 3.9. | Window | |
| | J.J. | ASSESSMENT OF COLUMANITUS DISCASE 2017 HIPPACE | |

| 4. | SUBJ | ECT DISE | POSITION | 41 |
|---|---|---|---|---|
| | 4.1. | Subject | Enrollment and Disposition | 41 |
| | 4.2. | | of Study Drug Exposure and Adherence | |
| | | 4.2.1. | Duration of Exposure to Study Drug | |
| | | 4.2.2. | Adherence to Study Drug | |
| | 4.3. | Protoco | 1 Deviations | |
| | 4.4. | | and Virtual Visits due to COVID-19 | |
| 5. | BASELINE CHARACTERISTICS | | | |
| | 5.1. | Demogr | raphics and Other Baseline Characteristics | 46 |
| | 5.2. | Baseline | Disease Characteristics | 46 |
| | 5.3. | Medical | l History | 49 |
| 6. | EFFI | CACY AN | IALYSES | 51 |
| | 6.1. | General | Considerations | 51 |
| | | 6.1.1. | Calculation of CDAI and PRO2 Scores | |
| | | 6.1.2. | Calculation of SES-CD and Other Endoscopy Endpoints | |
| | | 6.1.3. | COVID-19 Impact on Primary Efficacy Endpoints | |
| | 6.2. | Primary | Efficacy Endpoints | |
| | | 6.2.1. | Definition of the Primary Efficacy Endpoints | |
| | | 6.2.2. | Statistical Hypotheses for the Primary Efficacy Endpoints | |
| | | 6.2.3. | Estimands for the Primary Efficacy Endpoints | |
| | | 6.2.4. | Primary Analysis of the Primary Efficacy Endpoints | |
| | | 6.2.5. | Sensitivity Analyses for the Primary Efficacy Endpoints | |
| | | 6.2.6. | Analysis of the Primary Efficacy Endpoints for Japan Submission | |
| | | 6.2.7. | Subgroup Analyses for the Primary and key secondary Efficacy | |
| | | | Endpoints | 66 |
| | 6.3. | Seconda | ary Efficacy Endpoints | 68 |
| | | 6.3.1. | Definition of the Secondary Efficacy Endpoints | 68 |
| | | 6.3.2. | Analysis of the Secondary Efficacy Endpoints | 69 |
| | CCI | | | |
| | 6.5. | Cohorte | A and B End-of-Induction Analysis | 76 |
| | 6.6. | · | | |
| 7. | | | LYSES | |
| | 7.1. | | Events and Deaths | |
| | | 7.1.1. | Adverse Event Dictionary | |
| | | 7.1.2. | Adverse Event Severity | |
| | | 7.1.3. | Relationship of Adverse Events to Study Drug | |
| | | 7.1.4. | Serious Adverse Events | |
| | | 7.1.5. | Treatment-Emergent Adverse Events | |
| | | 7.1.6.<br>7.1.7. | Summaries of Adverse Events and Deaths Adverse Events of Interest | |
| | 7.2 | | | |
| | 7.2. | 7.2.1. | ory Evaluations | |
| | | 7.2.1.<br>7.2.2. | • | |
| | | | Graded Laboratory Values | |
| | | 7.2.3.<br>7.2.4. | Liver-Related Laboratory Evaluations | |
| | | 7.2.4.<br>7.2.5. | Shifts Relative to the Baseline Value | |
| | 7.3. | | Veight and Vital Signs | |
| | 7.3.<br>7.4. | | d Concomitant Medications | |
| | / .T. | TITOL all | Concomment Productions | |

| | 7.4.1. | | |
|---|---|---|---|
| | 7.4.2. | Concomitant Medications. | 90 |
| | 7.5. Electr | ocardiogram Results | 91 |
| | | Safety Measures | |
| | 7.7. Chang | ges from Protocol-Specified Safety Analyses | 91 |
| 8. | PHARMACO | KINETIC ANALYSES | 92 |
| CCI | | | |
| 10. | REFERENCE | SS | 94 |
| 11. | SOFTWARE | | 95 |
| 12. | 2. SAP REVISION | | |
| 13. | APPENDIX | | 101 |
| | | | 100 |
| | Appendix 1. | Schedule of Assessments | |
| | Appendix 2. | List of Biologics for CD Treatment | 107 |
| | Appendix 3. | Crohn's Disease Activity Index (CDAI) and Patient Reported Outcomes – 2 items | 100 |
| | Appandix 4 | (PRO2) | |
| | Appendix 4. Appendix 5. | • • | |
| | Appendix 6. | Simple Endoscopic Score for Crohn's Disease (SES-CD) Study Treatment Failure Rules | |
| | Appendix 6. Appendix 7. | Determining Missing and Virtual Visits due to COVID-19 | |
| | Appendix 8. | SAS Programming for Tipping Point Analysis for Binary Endpoint | |
| | Appendix 9. | MST lists for AEs of Interest. | |
| | Appendix 10. | | |
| | | LIST OF IN-TEXT TABLES | |
| | Table 1-1. | Re-Randomization of Induction Cohorts A and B to Maintenance Study | |
| | Table 3-1. | Analysis Visit Windows for Induction Study: CDAI, PRO2, CCI SES-CD, PGIS, | |
| | T 11 2 2 | PGIC and CC | 35 |
| | Table 3-2. | Analysis Visit Windows for Induction Study: Weight, Vital Signs, ECG, | |
| | CCI | Hematology, Chemistry, Lipid Profile, Serum Immunoglobulin, CCl | |
| | Table 3-4. | Analysis Visit Windows for Maintenance Study: CDAI, PRO2, CC SES-CD, | |
| | | PGIS and PGIC | 37 |
| | Table 3-5. | Analysis Visit Windows for Maintenance Study: | 37 |
| | Table 3-6. | Analysis Visit Windows for Maintenance Study: Weight, Vital Signs, ECG, | |
| | | Hematology, Chemistry, Lipid Profile, Serum Immunoglobulin and CC | |
| | CCI | | |
| | Table 6-1. | Definitions of Selected Efficacy Endpoints | |
| | Table 6-2. | Composite Estimand 1 (Primary Analysis) for Clinical Remission by PRO2 | |
| | Table 6-3. | Composite Estimand 2 (Sensitivity Analysis) for Clinical Remission by PRO2 | |
| | Table 6-4. | Composite Estimand 1 (Primary Analysis) for Clinical Remission by CDAI | |
| | Table 6-5. | Composite Estimand 2 (Sensitivity Analysis) for Clinical Remission by CDAI | |
| | Table 6-6. | Composite Estimand 1 (Primary Analysis) for Endoscopic Response | |
| | Table 6-7. | Composite Estimand 2 (Sensitivity Analysis) for Endoscopic Response | |
| | Table 13-1.<br>Table 13-2. | Calculation of Total CDAI Score | |
| | Table 13-2. | Calculation of PRO2 Components Calculation of Total PRO2 score | |
| | 1 aut 13"3. | Carculation of Total Livoz score | 103 |

| Table 13-4. | Calculation of CDAI Patient-Reported Outcome Components and PRO2 Scores at | |
|---|---|---|
| | Screening | 110 |
| Table 13-5. | Calculation of CDAI Patient-Reported Outcome Components and PRO2 Scores at | |
| | Post-Screening Visits | 113 |
| Table 13-6. | Sources of Information for Calculating CDAI and PRO2 Scores | 115 |
| Table 13-6. | Examples of Search Terms for "COVID-19" and "Virtual" Used to Identify Missed and Virtual Visits | |
| Figure 1-1 | LIST OF IN-TEXT FIGURES Study Schema | 14 |
| Figure 1-1. | Study Schema | 14 |
| Figure 3-1. | Induction Studies (Cohorts A and B): Testing Strategy for the Primary and Key Secondary Hypotheses | 25 |
| Figure 3-2. | Maintenance Study: Testing Strategy for the Primary and Key Secondary | 20 |
| | Hypotheses | 27 |
| Figure 3-3. | Induction Studies (Cohorts A and B): Testing Strategy for the Primary and Key | |
| | Secondary Hypotheses | 29 |
| Figure 3-4. | Maintenance Study: Testing Strategy for the Primary and Key Secondary | |
| | Hypotheses | 31 |

#### LIST OF ABBREVIATIONS

6-MP 6-mercaptopurine AE adverse event

AEI adverse event of interest
ALT alanine aminotransferase
ANCOVA analysis of covariance
AST aspartate aminotransferase

ASTE arterial systemic thromboembolism BLQ below the limit of quantitation

BMI body mass index CD Crohn's disease

CDAI Crohn's Disease Activity Index

CI confidence interval

COVID-19 Cochran-Mantel-Haenszel covoravirus disease 2019

CCI

CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

DMC data monitoring committee

ECG electrocardiogram

eCRF electronic case report form(s)

JUI

CCI

ET early termination
EU European Union
FAS Full Analysis Set

FWER family-wise type I error rate

CCI

Gilead Gilead Sciences

CCI

HDL high-density lipoprotein HLGT high-level group term

HLT high-level term

CCI

IBD inflammatory bowel disease

CCI

ID identification
Ig immunoglobulin

IWRS interactive web response system

LDL low-density lipoprotein
LLOQ lower limit of quantitation

LLT lower-level term

LOCF last observation carried forward

LOQ limit of quantitation

LS least squares

LTE long-term extension

MACE major adverse cardiovascular events

M-Day maintenance study day

MedDRA Medical Dictionary for Regulatory Activities

MH Mantel-Haenszel
MI myocardial infarction

MICE multivariate imputation by chained equations

CCI

MST MedDRA search term

MTX methotrexate

NCEP National Cholesterol Education Program

NLP natural language processing

CCI

PGIC Patient Global Impression Change PGIS Patient Global Impression Severity

PK pharmacokinetic

PKAP Pharmacokinetic analysis plan

PRO2 patient reported outcome consisting of 2 items: abdominal pain severity and liquid stool

frequency

PT preferred term
PTM placebo-to-match
Q1 first quartile
Q3 third quartile

CCI

SAE serious adverse event
SAP statistical analysis plan
SD standard deviation
SE standard error

SES-CD Simple Endoscopic Score for Crohn's Disease

CCI

SMQ Standardised MedDRA Query

SOC system organ class

T-Day subject activation date on the electronic diary device during screening

TEAE treatment-emergent adverse event

TFLs tables, figures, and listings TNF- $\alpha$  tumor necrosis factor-alpha

ULN upper limit of normal

US United States V-Day visit day

VAS visual analogue scale
VTE venous thromboembolism
WHO World Health Organization



## PHARMACOKINETIC ABBREVIATIONS

AUC area under the concentration versus time curve

AUC<sub>tau</sub> area under the concentration versus time curve over the dosing interval

C<sub>max</sub> the maximum observed concentration of drug in plasma

CL<sub>ss</sub>/F apparent oral clearance at steady state

C<sub>tau</sub> observed drug concentration at the end of the dosing interval

 $T_{max}$  the time (observed time point) of  $C_{max}$ 

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes all statistical analyses methods required to address both the EU and non-EU specific objectives. It also describes all tables, figures, and listings (TFLs) to be included in the clinical study report (CSR) for Study Protocol GS-US-419-3895/GLPG0634-CL-309.

This SAP is based on the study protocol Amendment 9 dated 02 December 2021 and the electronic case report forms (eCRF). The SAP will be approved before database finalization of the final analysis. Any changes made after the finalization of the SAP will be documented in the CSR.

#### 1.1. Study Objectives

The overall objective of the study is to evaluate the effect of treatment with filgotinib on the induction and maintenance of clinical remission and endoscopic response in subjects with moderately to severely active Crohn's disease (CD). Subjects who are biologic-naive or biologic-experienced will be enrolled in Cohort A and subjects who are biologic-experienced will be enrolled in Cohort B, respectively. Treatment assignments will be randomized within each cohort.

## 1.1.1. Primary Objectives

The primary objectives are:

## Induction Studies (Cohorts A and B) (EU-specific)

- To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical remission by Patient Reported Outcome (PRO2) at Week 10
- To evaluate the efficacy of filgotinib as compared to placebo in establishing endoscopic response at Week 10

## Induction Studies (Cohorts A and B) (other: non-EU)

• To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical remission by Crohn's Disease Activity Index (CDAI) at Week 10

To evaluate the efficacy of filgotinib as compared to placebo in establishing endoscopic response at Week 10

#### Maintenance Study (EU-specific)

- To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical remission by PRO2 at Week 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing endoscopic response at Week 58

## Maintenance Study (other: non-EU)

- To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical remission by CDAI at Week 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing endoscopic response at Week 58

#### 1.1.2. Secondary Objectives

The key secondary objectives are:

#### Induction Studies (Cohorts A and B) (EU-specific)

- To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical remission by Crohn's Disease Activity (CDAI) at Week 10
- To evaluate the efficacy of filgotinib as compared to placebo in establishing both clinical remission by PRO2 and endoscopic response (combined into a single endpoint on a patient level at Week 10

#### Induction Studies (Cohorts A and B) (other: non-EU)

- To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical remission by Patient Reported Outcomes (PRO2) at Week 10
- To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical response by CDAI at Week 10

#### Maintenance Study (EU-specific)

- To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical remission by CDAI at Week 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing sustained clinical remission by PRO2 at Weeks 10 and 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing both clinical remission by PRO2 and endoscopic response (combined into a single endpoint on a patient level) at Week 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing 6-month corticosteroid-free remission by PRO2 at Week 58

## Maintenance Study (other non-EU)

 To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical remission by PRO2 at Week 58

- To evaluate the efficacy of filgotinib as compared to placebo in establishing clinical response by CDAI at Week 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing sustained clinical remission by CDAI at Weeks 10 and 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing 6-month corticosteroid-free remission by CDAI at Week 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing sustained clinical remission by PRO2 at Weeks 10 and 58
- To evaluate the efficacy of filgotinib as compared to placebo in establishing 6-month corticosteroid-free remission by PRO2 at Week 58

The other secondary objectives are:

#### Induction Studies (Cohorts A and B)

- To evaluate the safety and tolerability of filgotinib
- To assess the pharmacokinetic (PK) characteristics of filgotinib

## Maintenance Study

- To evaluate the safety and tolerability of filgotinib
- To assess the PK characteristics of filgotinib





| • | CCI |
|---|---|
| C | |
| | CCI |
| - | |
| - | |
| C | |
| | To evaluate the efficacy of filgotinib as compared to placebo in establishing both clinical |
| | remission by PRO2 and endoscopic response (combined into a single endpoint on a patient level) at Week 58 |
| • | CCI |
| • | CCI |
| • | CCI |



These are combined Phase 3 randomized, double-blind, placebo-controlled studies to evaluate the efficacy and safety of filgotinib in the induction and maintenance of clinical remission, as well as endoscopic response in subjects with moderately to severely active Crohn's disease. A schematic of this study is provided in Figure 1-1.

Figure 1-1. Study Schema



FIL = filgotinib; PBO = placebo; PRO = patient reported outcomes

Non-responders are subjects who achieve <u>neither</u> clinical remission (PRO2) <u>nor</u> endoscopic response at Week 10.

Subjects in the Maintenance Study that meet disease worsening criteria (see protocol Section 3.6) will be offered open-label filgotinib.

## 1.2.1. Induction Studies (Cohort A and B)

Subjects who meet protocol eligibility criteria will be assigned to the respective cohort and subsequently randomized in a blinded fashion in a 1:1:1 ratio to 1 of 3 treatments as follows:

#### **Treatment Groups (Induction Studies)**

**Treatment Group 1 (n = 220):** Filgotinib 200 mg and placebo-to-match (PTM) filgotinib 100 mg, once daily

Treatment Group 2 (n = 220): Filgotinib 100 mg and PTM filgotinib 200 mg, once daily

Treatment Group 3 (n = 220): PTM filgotinib 200 mg and PTM filgotinib 100 mg, once daily

Note: males in the US and Korea who have not failed at least 2 biologic therapies (ie, any tumor necrosis factor-alpha [TNF- $\alpha$ ] antagonist <u>and</u> vedolizumab) will be randomized in a 1:1 ratio to receive either filgotinib 100 mg or matching placebo.

Based on the interactive web response system (IWRS) design, biologic-experienced subjects will not enroll in Cohort A until the enrollment for Cohort B has been closed. For subjects enrolled in Cohort A before the closure of Cohort B enrollment, treatment assignments will be stratified according to the following factors:

## <u>Stratification Factors (Cohort A, Biologic-Naive and Biologic-Experienced Induction Study, before Closure of Cohort B Enrollment)</u>

- Concomitant use of oral, systemically absorbed corticosteroids (eg, prednisone) at Day 1, (Yes or No)
- Concomitant use of immunomodulators (eg, 6-mercaptopurine [6-MP], azathioprine, methotrexate [MTX]) at Day 1, (Yes or No)

For subjects enrolled in Cohort A after the closure of Cohort B enrollment, treatment assignments will be stratified according to the following factors:

## <u>Stratification Factors (Cohort A, Biologic-Naive and Biologic-Experienced Induction</u> Study, after Closure of Cohort B Enrollment)

- History of exposure to no biologic agent, one biologic agent, or more than one biologic agent
- Concomitant use of oral, systemically absorbed corticosteroids (eg, prednisone) at Day 1, (Yes or No)
- Concomitant use of immunomodulators (eg, 6-MP, azathioprine, MTX) at Day 1, (Yes or No)

For subjects enrolled in Cohort B, treatment assignments will be stratified according to the following factors:

## **Stratification Factors (Cohort B, Biologic-Experienced Induction Study)**

- Exposure to *one* biologic agent versus *more than one* biologic agent
- Concomitant use of oral, systemically absorbed corticosteroids (eg, prednisone) at Day 1, (Yes or No)
- Concomitant use of immunomodulators (eg, 6-MP, azathioprine, MTX) at Day 1, (Yes or No)

## **1.2.2.** Maintenance Study

Subjects in Cohorts A and B who complete the Induction Study and achieve either clinical remission by PRO2 or endoscopic response at Week 10 will be re-randomized into the following treatments in the Maintenance Study at Week 11.

Table 1-1. Re-Randomization of Induction Cohorts A and B to Maintenance Study

| Treatment Assignment in Induction Studies, Cohorts A and B | Maintenance Study Re-randomization |
|---|---|
| Treatment 1 Electivih 200 mg | Treatment 1, 200 mg |
| Treatment 1, filgotinib 200 mg | Treatment 3, placebo |
| Treatment 2 Startinit 100 ma | Treatment 2, 100 mg |
| atment 2, filgotinib 100 mg | Treatment 3, placebo |
| Treatment 3, placebo | Continue Treatment 3, placebo |

Note: Subjects receiving Treatment 1 or 2 in the Induction study will be randomized in a 2:1 ratio to either continue on the assigned filgotinib regimen or to placebo for the duration of the Maintenance Study.

For subjects enrolled in Maintenance before the closure of Induction Cohort B enrollment, treatment assignments will be stratified according to the following factors:

# <u>Stratification Factors (Maintenance Study, before the Closure of Induction Cohort B Enrollment)</u>

- Participation in Cohort A or Cohort B
- Concomitant use of oral, systemically absorbed corticosteroids (eg, prednisone) at Day 1, (Yes or No)
- Concomitant use of immunomodulators (eg, 6-MP, azathioprine, MTX) at Day 1, (Yes or No)

For subjects enrolled in Maintenance after the closure of Induction Cohort B enrollment, treatment assignments will be stratified according to the following factors:

## <u>Stratification Factors (Maintenance Study, after the Closure of Induction Cohort B</u> Enrollment)

- History of exposure to a biologic agent, (Yes or No)
- Concomitant use of oral, systemically absorbed corticosteroids (eg, prednisone) at Day 1, (Yes or No)
- Concomitant use of immunomodulators (eg, 6-MP, azathioprine, MTX) at Day 1, (Yes or No)

Subjects who achieve neither clinical remission by PRO2 nor endoscopic response at Week 10 will have the option to enter a separate, Long-Term Extension (LTE) study (GS-US-419-3896/GLPG0634-CL-310). The Maintenance Study will run from Weeks 11 to 58 with the primary efficacy assessments at Week 58. Subjects who opt out of the LTE study will return 30 days after the last dose of study drug for post-treatment safety assessments. Subjects who complete all procedures per protocol, including the endoscopy, of the 58-week study will be offered the option to continue into the LTE study. Subjects who are eligible and opt to participate in the LTE study can continue into the study without post-treatment safety assessments.

#### 1.2.3. Pharmacokinetics Substudy

An optional PK substudy will be performed in a subset of subjects (approximately 30 subjects each in Cohort A and Cohort B) who provide separate informed consent. In the PK substudy, the daily dose of study drug should be administered under supervision in the clinic (at any single visit between Week 2 and Week 10, inclusive), and PK samples should be collected predose and at 0.5, 1, 2, 3, 4, and 6 hours after dosing. If a substudy PK sample is scheduled to be collected at the same time as a sparse PK sample, only one sample should be collected.

#### 1.2.4. Schedule of Assessments

Efficacy will be assessed primarily through CDAI, PRO2, and Simple Endoscopic Score for Crohn's Disease (SES-CD). CDAI and PRO2 will be assessed at Screening, Weeks 2, 4, 6, 10, 14, 20, 26, 34, 42, 50, and 58, and ET. SES-CD will be assessed at Screening, Week 10, and Week 58.

For additional details, please see the Schedule of Assessments in Appendix 1.

## 1.3. Sample Size and Power

## **Induction Studies (Cohorts A and B)**

## **EU-specific**:

The sample size was chosen to ensure that a clinically meaningful difference in both clinical remission rate by PRO2 at Week 10 and endoscopic response rate at Week 10 could be detected when comparing filgotinib 200 mg to placebo within each Induction Study.

A sample size of 220 subjects in each treatment group (N = 660 total) will provide an overall power of 93% for a filgotinib 200 mg dose group comparison to placebo at a 2-sided 0.05 significance level to detect a treatment difference of 15% in clinical remission rate by PRO2 at Week 10 (30% on filgotinib 200 mg and 15% on placebo) and a treatment difference of 15% in endoscopic response rate at Week 10 (25% on filgotinib 200 mg and 10% on placebo). Since each endpoint needs to achieve statistical significance, the overall power of 93% is calculated as the product of the two individual powers based on each endpoint.

#### Other (non-EU)

The sample size was chosen to ensure that a clinically meaningful difference in both clinical remission rate by CDAI at Week 10 and endoscopic response rate at Week 10 could be detected when comparing filgotinib 200 mg to placebo within each Induction Study.

A sample size of 220 subjects in each treatment group (N = 660 total) will provide an overall power of 97% for a filgotinib 200 mg dose group comparison to placebo at a 2-sided 0.05 significance level to detect a treatment difference of 20% in clinical remission rate by CDAI at Week 10 (45% on filgotinib 200 mg and 25% on placebo) and a treatment difference of 15% in endoscopic response rate at Week 10 (25% on filgotinib 200 mg and 10% on placebo). Since each endpoint needs to achieve statistical significance, the overall power of 97% is calculated as the product of the two individual powers based on each endpoint.

#### **Maintenance Study**

Assuming an Induction response rate (ie, proportion of subjects achieving clinical remission by PRO2 or endoscopic response at Week 10) of 40% among subjects receiving filgotinib 200 mg or filgotinib 100 mg treatment, approximately 176 subjects from each filgotinib dose group from Cohorts A and B Induction Studies combined would be eligible to be re-randomized into the Maintenance Study.

The sample size was chosen to ensure that a clinically meaningful difference in both clinical remission rate by CDAI and endoscopic response rate at Week 58 could be detected when comparing the filgotinib 200 mg dose group to placebo in the Maintenance Study.

A sample size of 60 subjects in the placebo group and 120 subjects in the filgotinib group at the same dose level as the induction dose will provide an overall 94% power for a filgotinib 200 mg

comparison to placebo at a 2-sided 0.05 significance level to detect a treatment difference of 30% in maintenance clinical remission rate by CDAI/PRO2 at Week 58 and maintenance endoscopic response rate at Week 58 (50% on filgotinib 200 mg and 20% on placebo). Since each endpoint needs to achieve statistical significance, the overall power of 94% is calculated as the product of the two individual powers based on each endpoint.

## 2. TYPE OF PLANNED ANALYSIS

## 2.1. Data Monitoring Committee (DMC) Analyses

The DMC's role and responsibilities and the scope of analysis to be provided to the DMC are described in a mutually agreed upon charter, which defines the DMC membership, meeting logistics, and meeting frequency.

#### 2.1.1. Safety Analyses

An external multidisciplinary DMC will review the progress of the study and perform interim reviews of safety data in order to protect subject welfare and preserve study integrity. The DMC is to recommend to the sponsor whether the nature, frequency, and severity of adverse events (AEs) associated with study treatment warrant the early termination of the study in the best interests of study subjects, whether the study should continue as planned, or whether the study should continue with modifications.

The initial meeting will occur after approximately 100 subjects complete Week 10 or discontinue from the study in Cohorts A and B combined. Following this, subsequent meetings will occur approximately once every 4 months or at a frequency determined by the DMC. Additional meetings may be triggered by safety findings, predetermined or otherwise.

## 2.1.2. Cohorts A and B End-of-Induction Analysis

Efficacy and safety analyses will be performed after *all* subjects in both cohorts complete Week 10 or prematurely discontinue study drug (and complete post-treatment assessments, if applicable). Please refer to Section 6.5 for details.

## 2.2. Final Analysis

After all subjects have completed the Maintenance Study, outstanding data queries have been resolved or adjudicated as unresolvable, and the data have been cleaned and finalized, the study blind will be broken and the final analysis of the data will be performed.

#### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of subjects in each category will be presented; for continuous variables, the number of subjects (n), mean, standard deviation (SD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

By-subject listings will be presented for all subjects in the All Randomized Analysis Set. Data collected on log forms, such as AEs, will be presented in chronological order within subject. The treatment group to which subjects were randomized or initially assigned will be used in the listings.

Unless otherwise specified, for the Maintenance Study, the data will be summarized by the Induction dose (ie, filgotinib 200 mg, filgotinib 100 mg, or placebo) and respective Maintenance dose, and overall for subject disposition and baseline characteristics described in Section 4 and Section 5, respectively. The data will be summarized by the Induction dose (ie, filgotinib 200 mg, filgotinib 100 mg) and respective Maintenance dose for efficacy and described in Section 6 and Section 9, respectively. The data will be summarized by the Induction dose (ie, filgotinib 200 mg, filgotinib 100 mg or placebo) and respective Maintenance dose for safety analyses described in Section 7. The data will be summarized by Maintenance treatment group for PK analyses described in Section 8.

## 3.1. Analysis Sets

Analysis sets define the subjects to be included in an analysis. Analysis sets and their definitions are provided in this section. The analysis set will be identified and included as a subtitle of each TFL.

For each analysis set, the number and percentage of subjects eligible for inclusion, as well as the number and percentage of subjects who were excluded and the reasons for their exclusion (if available), will be summarized by treatment group.

A listing of reasons for exclusion from analysis sets will be provided by subject.

#### 3.1.1. All Randomized Analysis Sets

The All Randomized Analysis Set for each Induction Study (Cohorts A and B) includes all subjects who were randomized on Day 1 into each corresponding study.

The All Randomized Analysis Set for the Maintenance Study includes all subjects who were re-randomized into the Maintenance Study (including subjects randomized to the placebo treatment group in the Induction Studies who continued on placebo treatment in the Maintenance Study).

The All Randomized Analysis Sets are the primary analysis sets for by-subject listings.

## 3.1.2. Full Analysis Sets

The Full Analysis Set (FAS) for each Induction Study (Cohorts A and B) includes all randomized subjects who took at least 1 dose of study drug in the corresponding Induction Study.

The FAS for the Maintenance Study includes all subjects randomized to either the filgotinib 200 mg or filgotinib 100 mg treatment groups in the Induction Studies who were re-randomized in the Maintenance Study and:

- Took at least 1 dose of study drug in the Maintenance Study, and
- Achieved clinical remission by PRO2 or endoscopic response at Week 10 as specified in the SAP.

The Full Analysis Sets are the primary analysis sets for efficacy analyses.

## 3.1.3. Safety Analysis Sets

The Safety Analysis Set for each Induction Study (Cohorts A and B) includes all subjects who took at least 1 dose of study drug in the corresponding Induction Study.

The Safety Analysis Set for the Maintenance Study includes all subjects who took at least 1 dose of study drug in the Maintenance Study.

The Safety Analysis Sets are the primary analysis sets for safety analyses.

## 3.1.4. Pharmacokinetic Analysis Sets

The primary analysis set for general PK analyses will be defined separately for each individual study (Cohort A Induction, Cohort B Induction, and Maintenance). For each study, the PK Analysis Set includes all randomized subjects who took at least 1 dose of filgotinib and have at least 1 nonmissing concentration value for filgotinib and/or its metabolite GS-829845 reported by the PK laboratory.

#### 3.1.5. Pharmacokinetic Substudy Analysis Sets

The primary analysis set for intensive PK analyses will be the PK Substudy Analysis Set for each Induction Study (Cohorts A and B), which includes all randomized subjects from the corresponding Induction Study who took at least 1 dose of filgotinib, participated in the PK substudy, and have at least 1 nonmissing intensive concentration value for filgotinib and/or its metabolite GS-829845 reported by the PK laboratory. This is the primary analysis set for detailed PK analysis of intensive PK sampling.



## 3.2. Subject Grouping

For analyses based on the All Randomized Analysis Sets and FAS, subjects will be grouped according to the treatment to which they were randomized. For analyses based on the Safety Analysis Sets and CCl subjects will be grouped according to actual treatment received. The actual treatment received will differ from the randomized treatment only when their actual treatment differs from randomized treatment for the entire treatment duration.

For the PK Analysis Sets, subjects will be grouped according to the actual treatment they received.

#### 3.3. Strata and Covariates

Subjects will be randomly assigned to treatment groups via IWRS using a stratified randomization schedule into each individual study (Cohort A Induction, Cohort B Induction, and Maintenance). Details of the randomization ratio and stratification variables for each study are provided in Section 1.2.

If there are discrepancies in stratification factor values between the IWRS and the clinical database (eCRF data), the baseline values recorded in the clinical database will be used for analyses. For the derivation of concomitant medication use at Day 1, the start date of such medication should be before or on the same date of the first dose of study drug and with either the stop date of such medication being on or after the first dose of study drug or with "ongoing" status.

Stratification factors will be used as covariates in evaluating efficacy endpoints, as specified in Section 6.

## 3.4. Examination of Subject Subgroups

Subgroup analyses for the primary and key secondary efficacy endpoints are specified in Section 6.2.7.

#### 3.5. Multiple Comparisons

The graphical approach {Bretz 2009} of sequentially rejective Bonferroni-based iterative multiple test procedures will be used to control a family-wise type I error rate (FWER) at 5% (ie,  $\alpha = 0.05$ ) for hypothesis testing on co-primary and key secondary endpoints for each

individual study (Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study). This procedure strongly protects the FWER on all the primary and key secondary endpoints.

## 3.5.1. EU-Specific

#### 3.5.1.1. Induction Studies (Cohorts A and B)

The hypotheses to be tested for the Induction Studies are outlined below.

The primary null hypotheses to be tested:

- H<sub>11</sub>: The clinical remission by PRO2 rate in the filgotinib 200 mg group is equal to the clinical remission by PRO2 rate in the placebo group at Week 10
- H<sub>12</sub>: The endoscopic response rate in the filgotinib 200 mg group is equal to the endoscopic response rate in the placebo group at Week 10
- H<sub>21</sub>: The clinical remission by PRO2 rate in the filgotinib 100 mg group is equal to the clinical remission by PRO2 rate in the placebo group at Week 10
- H<sub>22</sub>: The endoscopic response rate in the filgotinib 100 mg group is equal to the endoscopic response rate in the placebo group at Week 10

The key secondary null hypotheses to be tested:

- H<sub>13</sub>: The clinical remission by CDAI rate in the filgotinib 200 mg group is equal to the clinical remission by CDAI rate in the placebo group at Week 10
- H<sub>14</sub>: The clinical remission by PRO2 and endoscopic response rate (combined into a single endpoint on a patient level) in the filgotinib 200 mg group is equal to the clinical remission by PRO2 and endoscopic response rate (combined into a single endpoint on a patient level) in the placebo group at Week 10
- H<sub>23</sub>: The clinical remission by CDAI rate in the filgotinib 100 mg group is equal to the clinical remission by CDAI rate in the placebo group at Week 10
- H<sub>24</sub>: The clinical remission by PRO2 and endoscopic response rate (combined into a single endpoint on patient level) in the filgotinib 100 mg group is equal to the clinical remission by PRO2 and endoscopic response rate (combined into a single endpoint on a patient level) in the placebo group at Week 10

Each co-primary endpoint for filgotinib 200 mg compared with placebo will be tested at 2-sided 0.05 significance level first. If it fails to reject the null hypothesis for at least one co-primary endpoint, then no further formal testing will be performed. If the null hypotheses for both co-primary endpoints are rejected, testing will proceed in two sequences as describe below:

- Key secondary endpoints for filgotinib 200 mg compared with placebo at 2-sided 0.025 significance level in a sequential order
- Each co-primary endpoint for filgotinib 100 mg compared with placebo at 2-sided 0.025 significance level. If the null hypotheses for both co-primary endpoints are rejected, then the key secondary endpoints for filgotinib 100 mg compared with placebo at 2-sided 0.025 significance level will be tested in a sequential order

If all the null hypotheses within the same sequence are rejected, then the respective alpha can be passed on to the other sequence. If an endpoint fails to reach statistical significance within the sequence, then formal testing will stop, and only nominal significance will be reported for the remaining endpoints.

A graphical illustration of the testing strategy for the primary and key secondary hypotheses in the Induction Studies is shown in Figure 3-1.

Figure 3-1. Induction Studies (Cohorts A and B): Testing Strategy for the Primary and Key Secondary Hypotheses



## 3.5.1.2. Maintenance Study

The hypotheses to be tested for the Maintenance Study are outlined below.

The primary null hypotheses to be tested:

- H<sub>11</sub>: The clinical remission by PRO2 rate in the filgotinib 200 mg group is equal to the clinical remission by PRO2 rate in the placebo group at Week 58
- H<sub>12</sub>: The endoscopic response rate in the filgotinib 200 mg group is equal to the endoscopic response rate in the placebo group at Week 58
- H<sub>21</sub>: The clinical remission by PRO2 rate in the filgotinib 100 mg group is equal to the clinical remission by PRO2 rate in the placebo group at Week 58
- H<sub>22</sub>: The endoscopic response rate in the filgotinib 100 mg group is equal to the endoscopic response rate in the placebo group at Week 58

The key secondary null hypotheses to be tested:

- H<sub>13</sub>: The clinical remission by CDAI rate in the filgotinib 200 mg group is equal to the clinical remission by CDAI rate in the placebo group at Week 58
- H<sub>14</sub>: The sustained clinical remission by PRO2 rate in the filgotinib 200 mg group is equal to sustained clinical remission by PRO2 rate in the placebo group at Weeks 10 and 58
- H<sub>15</sub>: The clinical remission by PRO2 and endoscopic response rate (combined into a single endpoint on a patient level) in the filgotinib 200 mg group is equal to the clinical remission by PRO2 and endoscopic response rate (combined into a single endpoint on a patient level) in the placebo group at Week 58
- H<sub>16</sub>: The 6-month corticosteroid-free remission by PRO2 rate in the filgotinib 200 mg group is equal to the 6-month corticosteroid-free remission by PRO2 rate in the placebo group at Week 58
- H<sub>23</sub>: The clinical remission by CDAI rate in the filgotinib 100 mg group is equal to the clinical remission by CDAI rate in the placebo group at Week 58
- H<sub>24</sub>: The sustained clinical remission by PRO2 rate in the filgotinib 100 mg group is equal to sustained clinical remission by PRO2 rate in the placebo group at Weeks 10 and 58
- H<sub>25</sub>: The clinical remission by PRO2 and endoscopic response rate (combined into a single endpoint on a patient level) in the filgotinib 100 mg group is equal to the clinical remission by PRO2 and endoscopic response rate (combined into a single endpoint on a patient level) in the placebo group at Week 58
- H<sub>26</sub>: The 6-month corticosteroid-free remission by PRO2 rate in the filgotinib 100 mg group is equal to the 6-month corticosteroid-free remission by PRO2 rate in the placebo group at Week 58

A similar approach as in the induction studies will be followed. A graphical illustration for the testing strategies for the primary and key secondary hypotheses in the Maintenance Study is shown in Figure 3-2.

Figure 3-2. Maintenance Study: Testing Strategy for the Primary and Key Secondary Hypotheses



## **3.5.2. Other (non-EU)**

#### 3.5.2.1. Induction Studies (Cohorts A and B)

The hypotheses to be tested for the Induction Studies are outlined below.

The primary null hypotheses to be tested:

• H<sub>11</sub>: The clinical remission by CDAI rate in the filgotinib 200 mg group is equal to the clinical remission by CDAI rate in the placebo group at Week 10

- H<sub>12</sub>: The endoscopic response rate in the filgotinib 200 mg group is equal to the endoscopic response rate in the placebo group at Week 10
- H<sub>21</sub>: The clinical remission by CDAI rate in the filgotinib 100 mg group is equal to the clinical remission by CDAI rate in the placebo group at Week 10
- H<sub>22</sub>: The endoscopic response rate in the filgotinib 100 mg group is equal to the endoscopic response rate in the placebo group at Week 10

The key secondary null hypotheses to be tested:

- H<sub>13</sub>: The clinical remission by PRO2 rate in the filgotinib 200 mg group is equal to the clinical remission by PRO2 rate in the placebo group at Week 10
- H<sub>14</sub>: The clinical response by CDAI rate in the filgotinib 200 mg group is equal to the clinical response by CDAI rate in the placebo group at Week 10
- H<sub>23</sub>: The clinical remission by PRO2 rate in the filgotinib 100 mg group is equal to the clinical remission by PRO2 rate in the placebo group at Week 10
- H<sub>24</sub>: The clinical response by CDAI rate in the filgotinib 100 mg group is equal to the clinical response by CDAI rate in the placebo group at Week 10

A similar approach as for the EU-specific endpoints will be followed. A graphical illustration of the testing strategy for the primary and key secondary hypotheses in the Induction Studies is shown in Figure 3-3.

Figure 3-3. Induction Studies (Cohorts A and B): Testing Strategy for the Primary and Key Secondary Hypotheses



## 3.5.2.2. Maintenance Study

The hypotheses to be tested for the Maintenance Study are outlined below.

The primary null hypotheses to be tested:

- H<sub>11</sub>: The clinical remission by CDAI rate in the filgotinib 200 mg group is equal to the clinical remission by CDAI rate in the placebo group at Week 58
- H<sub>12</sub>: The endoscopic response rate in the filgotinib 200 mg group is equal to the endoscopic response rate in the placebo group at Week 58
- H<sub>21</sub>: The clinical remission by CDAI rate in the filgotinib 100 mg group is equal to the clinical remission by CDAI rate in the placebo group at Week 58
- H<sub>22</sub>: The endoscopic response rate in the filgotinib 100 mg group is equal to the endoscopic response rate in the placebo group at Week 58

The key secondary null hypotheses to be tested:

- H<sub>13</sub>: The clinical remission by PRO2 rate in the filgotinib 200 mg group is equal to the clinical remission by PRO2 rate in the placebo group at Week 58
- H<sub>14</sub>: The clinical response by CDAI rate in the filgotinib 200 mg group is equal to the clinical response by CDAI rate in the placebo group at Week 58
- H<sub>15</sub>: The sustained clinical remission by CDAI rate in the filgotinib 200 mg group is equal to sustained clinical remission by CDAI rate in the placebo group at Weeks 10 and 58
- H<sub>16</sub>: The 6-month corticosteroid-free remission by CDAI rate in the filgotinib 200 mg group is equal to the 6-month corticosteroid-free remission by CDAI rate in the placebo group at Week 58
- H<sub>17</sub>: The sustained clinical remission by PRO2 rate in the filgotinib 200 mg group is equal to the sustained clinical remission by PRO2 rate in the placebo group at Weeks 10 and 58
- H<sub>18</sub>: The 6-month corticosteroid-free remission by PRO2 rate in the filgotinib 200 mg group is equal to 6-month corticosteroid-free remission by PRO2 rate in the placebo group at Week 58
- H<sub>23</sub>: The clinical remission by PRO2 rate in the filgotinib 100 mg group is equal to the clinical remission by PRO2 rate in the placebo group at Week 58
- H<sub>24</sub>: The clinical response by CDAI rate in the filgotinib 100 mg group is equal to the clinical response by CDAI rate in the placebo group at Week 58
- H<sub>25</sub>: The sustained clinical remission by CDAI rate in the filgotinib 100 mg group is equal to sustained clinical remission by CDAI rate in the placebo group at Weeks 10 and 58
- H<sub>26</sub>: The 6-month corticosteroid-free remission by CDAI rate in the filgotinib 100 mg group is equal to the 6-month corticosteroid-free remission by CDAI rate in the placebo group at Week 58
- H<sub>27</sub>: The sustained clinical remission by PRO2 rate in the filgotinib 100 mg group is equal to the sustained clinical remission by PRO2 rate in the placebo group at Weeks 10 and 58
- H<sub>28</sub>: The 6-month corticosteroid-free remission by PRO2 rate in the filgotinib 100 mg group is equal to 6-month corticosteroid-free remission by PRO2 rate in the placebo group at Week 58

A similar approach as for the EU-specific endpoints will be followed. A graphical illustration for the testing strategies for the primary and key secondary hypotheses in the Maintenance Study is shown in Figure 3-4.

Figure 3-4. Maintenance Study: Testing Strategy for the Primary and Key Secondary Hypotheses



## 3.6. Missing Data and Outliers

## 3.6.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified. Exceptions are presented in this document.

For missing last dosing date of study drug, imputation rules are described in Section 4.2.1. Imputation and calculation rules for missing patient diary data and other CDAI components are described in Appendix 3. Imputation and calculation rules for missing SES-CD data are described in Section 6.1.2. The handling of missing or incomplete dates for AE onset is described in Section 7.1.5.2 and for prior and concomitant medications in Section 7.4.

#### 3.6.2. Outliers

Outliers will be identified during the data management and data analysis process. All data, including outliers, will be included in the data analysis, unless otherwise specified.

## 3.7. Data Handling Conventions and Transformations

In general, age (in years) on the date of the first dose of study drug will be used for analyses and presentation in listings. If an enrolled subject was not dosed with any study drug, the randomization date will be used instead of the first dosing date of study drug. For screen failures, the date the informed consent was signed will be used for age calculation. If only birth year is collected on the eCRF, "01 July" will be used for the unknown birth day and month for the purpose of age calculation. If only birth year and month are collected, "15" will be used for the unknown birth day.

Duration of CD (years) is the number of years between the diagnosis date of CD and date of first dose of Induction study drug. The partial diagnosis date of CD (if any) will be imputed for calculation as follows:

- If day and month are missing but year is available, then the imputed day and month will be 01 Jan.
- If day is missing but the month and year are available, then the imputed day will be the first day of the month.
- Partial date will not be imputed if the year is missing.

Non-PK Data that are continuous in nature but are less than the lower limit of quantitation (LOQ) or above the upper LOQ will be imputed as follows:

- A value that is 1 unit less than the LOQ will be used for calculation of descriptive statistics if the datum is reported in the form of "< x" (where x is considered the LOQ). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used for calculation of summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used for calculation of summary statistics.
- A value that is 1 unit above the LOQ will be used for calculation of descriptive statistics if the datum is reported in the form of "> x" (where x is considered the LOQ). Values with decimal points will follow the same logic as above.
- The LOQ will be used for calculation of descriptive statistics if the datum is reported in the form of " $\leq$  x" or " $\geq$  x" (where x is considered the LOQ).

Natural logarithm transformation will be used for plasma concentrations and analysis of PK parameters. Plasma concentration values that are below the limit of quantitation (BLQ) will be presented as "BLQ" in the concentration data listing. Values that are BLQ will be treated as 0 at predose time points, and one-half the value of the LOQ at postbaseline time points.

The following conventions will be used for the presentation of summary and order statistics:

- If at least 1 subject has a concentration value of BLQ for the time point, the minimum value will be displayed as "BLQ."
- If more than 25% of the subjects have a concentration data value of BLQ for a given time point, the minimum and Q1 values will be displayed as "BLQ."
- If more than 50% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, and median values will be displayed as "BLQ."
- If more than 75% of the subjects have a concentration data value of BLQ for a given time point, the minimum, Q1, median, and Q3 values will be displayed as "BLQ."
- If all subjects have concentration data values of BLQ for a given time point, all order statistics (minimum, Q1, median, Q3, and maximum) will be displayed as "BLQ."

Pharmacokinetic parameters that are BLQ will be imputed as one-half LOQ before log transformation or statistical model fitting.

## 3.8. Analysis Visit Windows

#### 3.8.1. Definitions

#### 3.8.1.1. Induction Studies (Cohorts A and B)

<u>The First Dosing Date</u> of each Induction Study is defined as the date when subjects take the first dose of Induction study drug, as recorded in the Study Drug Administration eCRF.

<u>The Last Dosing Date</u> of each Induction Study is defined as the date when subjects take the last dose of Induction study drug as recorded in the Study Drug Administration eCRF.

Study Day will be calculated from the first dosing date of study drug and derived as follows:

- For days on or after first dosing date: Assessment Date First Dosing Date + 1
- For days prior to the first dosing date: Assessment Date First Dosing Date

Therefore, Study Day 1 is the day of the first dose of study drug administration.

<u>Baseline</u> is defined as the last available observation on or prior to the first dosing date, unless otherwise specified.

## 3.8.1.2. Maintenance Study

<u>The First Dosing Date</u> of Maintenance Study is defined as the date when subjects take the first dose of Maintenance Study drug, as recorded in the Study Drug Administration eCRF.

<u>The Last Dosing Date</u> of Maintenance Study is defined as the date when subjects take the last dose of Maintenance Study drug as recorded in the Study Drug Administration eCRF.

<u>Maintenance Study Day</u> (M-Day) will be calculated from the First Dosing Date of Maintenance Study and derived as:

- For days on or after First Dosing Date of Maintenance Study:
   Assessment Date First Dosing Date + 1
- For days prior to First Dosing Date of Maintenance Study: Assessment Date – First Dosing Date

Therefore, M-Day 1 is the first dosing date of the Maintenance Study.

<u>Re-randomization baseline</u> (henceforth referred to as maintenance baseline) is defined as the last available observation on or prior to the first dosing date of the Maintenance Study. Maintenance baseline will be considered the baseline of Maintenance Study, unless otherwise specified.

## 3.8.2. Analysis Visit Windows

Subject visits may not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.



Note: the rule for selecting on-treatment data will precede assigning records to analysis windows. Therefore, for 2 lab measurements equidistant to the target day, but only one being on-treatment, then the on-treatment measurement will be selected.

Table 3-1. Analysis Visit Windows for Induction Study: CDAI, PRO2, CC SES-CD, PGIS, PGIC and CC

| Nominal Visit | Analysis Visit | Nominal Day<br>(Study Day) | Lower Limit<br>(Study Day) | Upper Limit<br>(Study Day) |
|---|---|---|---|---|
| Screening/Day 1 | Baseline | 1 | (none) | 1 |
| Week 2 | Week 2 | 15 | 2 | 22 |
| Week 4 | Week 4 | 29 | 23 | 36 |
| Week 6 | Week 6 | 43 | 37 | 57 |
| Week 10 | Week 10 | 71 | 58 | Minimum of 85 and<br>Study Day of<br>[Maintenance<br>first dose date<br>(if applicable)] |

CDAI = Crohn's Disease Activity Index; CCI

·PGIC

<sup>=</sup> patient global impression change; PGIS = patient global impression severity; PRO2 = patient reported outcome consisting of 2 items: abdominal pain severity and liquid stool frequency; SES-CD = simple endoscopic score for Crohn's diseaseNote: For analysis purpose, PRO2 from Screening and Visit Day 1 will be calculated and both visits will be considered for the derivation of baseline, which is defined as the last available observation on or prior to the first dosing date of the study drug.

Note: PGIC at maintenance baseline will not be created.

Table 3-2. Analysis Visit Windows for Induction Study: Weight, Vital Signs, ECG, Hematology, Chemistry, Lipid Profile, Serum Immunoglobulin,

| Nominal Visit | Analysis Visit | Nominal Day<br>(Study Day) | Lower Limit<br>(Study Day) | Upper Limit<br>(Study Day) |
|---|---|---|---|---|
| Screening/Day 1 | Baseline | 1 | (none) | 1 |
| Week 2 | Week 2 | 15 | 2 | 22 |
| Week 4 | Week 4 | 29 | 23 | 36 |
| Week 6 | Week 6 | 43 | 37 | 57 |
| Week 10 | Week 10 | 71 | 58 | For subjects who entered Maintenance Study: minimum of 85 and Study Day of [Maintenance first dose date]; For other subjects: ≥ 71 |

ECG = electrocardiogram; CCl


Table 3-4. Analysis Visit Windows for Maintenance Study: CDAI, PRO2, SES-CD, PGIS and PGIC

| Nominal Visit | Analysis Visit | Nominal Day<br>(M-Day) | Lower Limit<br>(M-Day) | Upper Limit<br>(M-Day) |
|---|---|---|---|---|
| Week 10/Week 11 | Maintenance -baseline | 1 | (none) | 1 |
| Week 14 | Maintenance Week 3 | 22 | 2 | 43 |
| Week 20 | Maintenance Week 9 | 64 | 44 | 85 |
| Week 26 | Maintenance Week 15 | 106 | 86 | 134 |
| Week 34 | Maintenance Week 23 | 162 | 135 | 190 |
| Week 42 | Maintenance Week 31 | 218 | 191 | 246 |
| Week 50 | Maintenance Week 39 | 274 | 247 | 302 |
| Week 58 | Maintenance Week 47 | 330 | 303 | 358 |

CDAI = Crohn's Disease Activity Index; CC M-Day = maintenance study day; CC PGIC = patient global impression change; PGIS = patient global impression severity;

PRO2 = patient reported outcome consisting of 2 items: abdominal pain severity and liquid stool frequency; SES-CD = simple endoscopic score for Crohn's disease.

Note: For analysis purpose, PRO2 from Weeks 10 and 11 will be considered for the derivation of maintenance baseline, which is defined as the last available observation on or prior to the first dosing date of the study drug in Maintenance Study. Note: PGIC at maintenance baseline will not be created.



**Table 3-6.** Analysis Visit Windows for Maintenance Study: Weight, Vital Signs, ECG, Hematology, Chemistry, Lipid Profile, Serum Immunoglobulin and CC

| Nominal Visit | Analysis Visit | Nominal Day<br>(M-Day) | Lower Limit<br>(M-Day) | Upper Limit<br>(M-Day) |
|---|---|---|---|---|
| Week 10/Week 11 | Maintenance baseline | 1 | (none) | 1 |
| Week 14 | Maintenance Week 3 | 22 | 2 | 43 |
| Week 20 | Maintenance Week 9 | 64 | 44 | 85 |
| Week 26 | Maintenance Week 15 | 106 | 86 | 134 |
| Week 34 | Maintenance Week 23 | 162 | 135 | 190 |
| Week 42 | Maintenance Week 31 | 218 | 191 | 246 |
| Week 50 | Maintenance Week 39 | 274 | 247 | 302 |
| Week 58 | Maintenance Week 47 | 330 | 303 | ≥ 330 |

ECG = electrocardiogram; CCl M-Day = maintenance study day

Maintenance baseline will be calculated using Week 11 assessment if available. If there is no Week 11 assessment scheduled, the Week 10 assessment will be used for calculation.



M-Day = maintenance study day

Maintenance baseline will be calculated using Week 11 assessment if available. If there is no Week 11 assessment scheduled, the Week 10 assessment will be used for calculation.

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window.

If multiple, valid, nonmissing, continuous measurements exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- In general, the baseline/maintenance baseline value will be the last nonmissing value on or prior to the first dosing date of study drug for each individual Induction Study, and Maintenance Study, respectively, unless otherwise specified. If multiple measurements occur on the same day, the last nonmissing value prior to the first dose of study drug will be considered as the baseline value. If these multiple measurements occur at the same time or the time is not available, the average of these measurements (for continuous data) will be considered the baseline/maintenance baseline value.
- For postbaseline visits:
  - The record closest to the nominal day for that visit will be selected.
  - If there are 2 records that are equidistant from the nominal day, the later record will be selected.
  - If there is more than 1 record on the selected day, the average will be taken, unless otherwise specified.

If multiple, valid, nonmissing, categorical measurements exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- For baseline/maintenance baseline, the last available record on or prior to the date of the first dose of study drug for each individual study (Cohort A Induction, Cohort B Induction, and Maintenance) will be selected. If there are multiple records with the same time or no time recorded on the same day, the value with the lowest severity will be selected (eg, normal will be selected over abnormal for safety ECG findings).
- For postbaseline visits:
  - The record closest to the nominal day for that visit will be selected.
  - If there are 2 records that are equidistant from the nominal day, the later record will be selected.
  - If there is more than 1 record on the selected day, the worst severity will be taken (eg, abnormal will be selected over normal for safety ECG findings), unless otherwise specified.
  - For shift tables for safety endpoints, the worst severity within the analysis window will be used.

# 3.9. Assessment of Coronavirus Disease 2019 Impact

This study is ongoing during the coronavirus disease 2019 (COVID-19) pandemic, which has had an impact on study conduct. For example, some subjects were unable to attend onsite visits due to shelter-in-place guidelines, site closures, or other public health measures in response to the COVID-19 pandemic. Due to these restrictions, virtual visits may be conducted and alternative assessments (eg, local laboratory tests) may be used to assess subject safety and efficacy.

The assessment on the impact of the COVID-19 pandemic will be provided in the corresponding sections (mainly on subject disposition, efficacy analyses and safety analyses in Sections 4, 6, and 7, respectively) throughout this SAP.

Laboratory results from local laboratories (except hematocrit) due to COVID-19 impact will not be collected in the eCRF. Vital signs collected at home (except body weight) during virtual visits due to COVID-19 impact will not be collected in the eCRF. Hematocrit results collected from local laboratories, body weight measured at home due to COVID-19 impact will be used in CDAI calculations only, and will not be included in the safety summary (Sections 7.2. and 7.3, respectively). All laboratory and vital sign data collected will be included in listings, with a flag to indicate which records were collected at a local laboratory or at home, respectively.

# 4. SUBJECT DISPOSITION

# 4.1. Subject Enrollment and Disposition

For each individual study (Cohort A Induction, Cohort B Induction, and Maintenance), key study dates (ie, first subject screened, first subject randomized, last subject randomized, last subject last visit for each co-primary endpoint, and last subject last visit for the CSR) will be provided.

For each individual study (Cohort A Induction, Cohort B Induction, and Maintenance), a summary of subject enrollment will be provided by treatment group for each country, investigator within a country, and overall. The summary will present the number and percentage of subjects enrolled. For each column, the denominator for the percentage calculation will be the total number of subjects analyzed for that column.

For each individual study (Cohort A Induction, Cohort B Induction, and Maintenance), a similar enrollment table will be provided by randomization stratum. The denominator for the percentage of subjects in the stratum will be the total number of enrolled subjects. If there are discrepancies in the value used for stratification assignment between the IWRS and the clinical database, the value collected in the clinical database will be used for the summary. Subjects with discrepancies in the value used for stratification assignment between the IWRS and the clinical database at the time of data finalization will be summarized by treatment group and overall. A corresponding listing will also be provided.

The randomization schedule used for each individual study (Cohort A Induction, Cohort B Induction, and Maintenance) will be provided as an appendix to the CSR.

# Cohort A Induction Study and Cohort B Induction Study

A summary of subject disposition will be provided by treatment group and overall for each individual Induction study. This summary will present the number of subjects screened, the number of subjects who met all eligibility criteria but were not randomized with reasons subjects were not randomized, the number of subjects randomized, and the number of subjects in each of the categories listed below:

- Full Analysis Set
- Safety Analysis Set
- PK Analysis Set
- PK Substudy Analysis Set



- Completed study drug dosing through Week 10 (indicated in Induction Study Drug Completion eCRF)
- Continuing study drug (for analysis other than the final analysis)
- Did not complete study drug up to Week 10 with reasons for premature discontinuation of study drug
- Completed Induction Study through Week 11
- Continuing Induction Study (for analysis other than the final analysis)
- Did not complete Induction Study with reasons for premature discontinuation from the study

## Maintenance Study

A summary of subject disposition will be provided by treatment group and overall. This summary will present the number of subjects who completed the Induction Studies, the number of subjects re-randomized, and the number of subjects in each of the categories listed below:

- Full Analysis Set
- Safety Analysis Set
- PK Analysis Set
- · CCI
- Completed study drug dosing through Week 58
- Did not complete study drug with reasons for premature discontinuation of study drug as captured in the CRF.
- Completed Maintenance Study (defined as completion of protocol-planned duration of the study through Week 58)
- Did not complete Maintenance Study with reasons for premature discontinuation from the study

For the status of study drug and study completion and reasons for premature discontinuation, the number and percentage of subjects in each category will be provided. The denominator for the percentage calculation will be the total number of subjects in the Safety Analysis Set corresponding to that column in that study.

A similar summary as described for subject disposition summary will be provided for discontinuing study drug or study due to COVID-19.

The following by-subject listings will be provided by subject identification (ID) number in ascending order to support the above summary tables:

- Reasons for premature study drug or study discontinuation (a separate listing of reasons for premature study drug or study discontinuation due to COVID-19 will be created)
- Reasons for screen failure (will be provided by screening ID number in ascending order)
- Lot number and kit ID of assigned study medication

# 4.2. Extent of Study Drug Exposure and Adherence

Extent of exposure to study drug will be examined by assessing the total duration of exposure to study drug and the level of adherence to the study drug specified in the protocol.

Summaries of extent of study drug exposure and adherence will be provided for:

- Cohort A Induction Study
- Cohort B Induction Study
- Maintenance Study

A by-subject listing will be provided to support summaries.

In addition, a by-subject listing of study drug administration will be created for subjects with study drug interruption due to COVID-19 impact.

# **4.2.1. Duration of Exposure to Study Drug**

Total duration of exposure to study drug will be defined as last dosing date minus first dosing date plus 1, regardless of any temporary interruptions in study drug administration, and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks). If the last study drug dosing date is missing (for subjects that haves stopped treatment or the study as indicated by a study disposition record), the latest date among the treatment (study) disposition, clinical visit date, laboratory sample collection date, and vital sign assessment date that occurred during the ontreatment period (e.g. after exposure start date) will be used.

If month and year of the last dose are known, and the last study drug dosing date imputed above is different from the month collected, the last date of that month will be used. If only year of the last dose is known, and the last study drug dosing date imputed above is after the year collected, the last date of that year will be used; if the last study drug dosing date imputed above is before the year collected, the first date of that year will be used.

The total duration of exposure to study drug will be summarized for the following using descriptive statistics and using the number (ie, cumulative counts) and percentage of subjects exposed through the following time periods:

• Cohort A Induction Study: 1 day, 2 weeks, 4 weeks, 6 weeks, 10 weeks, and 11 weeks

- Cohort B Induction Study: 1 day, 2 weeks, 4 weeks, 6 weeks, 10 weeks, and 11 weeks
- Maintenance Study: 1 day, 3 weeks, 9 weeks, 15 weeks, 23 weeks, 31 weeks, 39 weeks, and 47 weeks

Summaries will be provided by treatment group for the Safety Analysis Set.

No formal statistical testing is planned.

# 4.2.2. Adherence to Study Drug

The total number of tablets administered will be summarized using descriptive statistics.

The presumed total number of tablets administered to a subject will be determined by the data collected on the drug accountability eCRF using the following formula. If the bottle was not returned, it is assumed that the subject took all the study drug tablets from the dispensed bottle. The number of tablets returned will be imputed as zero for the given bottle for study drug adherence calculation purpose.

The total number of tablets administered =

Total number of tables dispensed – total number of tablets returned

#### 4.2.2.1. On-Treatment Adherence

The level of on-treatment adherence to the study drug regimen will be determined by the total amount of study drug administered relative to the total amount of study drug expected to be administered during a subject's actual on-treatment period based on the study drug regimen.

The level of on-treatment adherence will be expressed as a percentage using the following formula:

On-Treatment Adherence (%) = 
$$\left(\frac{\text{Total Amount of Study Drug Administered}}{\text{Study Drug Expected to be Administered on Treatment}}\right) \times 100$$

Descriptive statistics for the level of on-treatment adherence with the number and percentage of subjects belonging to adherence categories (eg, < 80%,  $\ge 80\%$  to < 90%,  $\ge 90\%$  to < 120,  $\ge 120$ ) will be provided by treatment group for the Safety Analysis Set.

No formal statistical testing is planned.

A by-subject listing of study drug administration and drug accountability will be provided by subject ID number (in ascending order) and visit (in chronological order).

#### 4.3. Protocol Deviations

Subjects who did not meet the eligibility criteria for study entry, but enrolled in the study will be summarized. The summary will present the number and percentage of subjects who did not meet at least 1 eligibility criterion and the number of subjects who did not meet specific criteria by treatment group and overall based on the All Randomized Analysis Set. A by-subject listing will be provided for those subjects who did not meet at least 1 eligibility (inclusion or exclusion) criterion. The listing will present the eligibility criterion (or criteria if more than 1 deviation) that subjects did not meet and related comments, if collected.

Protocol deviations occurring after subjects entered the study are documented during routine monitoring. The number and percentage of subjects with major protocol deviations by deviation reason (eg, nonadherence to study drug, violation of key inclusion/exclusion criteria) will be summarized by treatment group and overall for the All Randomized Analysis Set for each individual study. A by-subject listing will be provided for those subjects with any major protocol deviation.

Similar summary and listing will be provided for major protocol deviations due to COVID-19.

#### 4.4. Missed and Virtual Visits due to COVID-19

A summary of subjects with missed or virtual visits due to the COVID-19 pandemic will be provided for each scheduled study visit by treatment group and overall for the All Randomized Analysis Set for each individual study. For each visit, the summary will present the number and percentage of subjects who missed the visit due to COVID-19 or had a virtual visit due to COVID-19.

An overall summary of the number and percentage of subjects with missed or virtual visits (eg, subjects with at least 1 missed or virtual visit, subjects with 1, 2, 3, or > 3 missed or virtual visits) due to the COVID-19 pandemic will be provided by treatment group and overall.

A by-subject listing of subjects with missed or virtual visits due to COVID-19 will be provided by subject ID number in ascending order.

Information regarding missed or virtual visits due to COVID-19 was collected as free text in the CRF comment fields. The determination of missing or virtual visits due to COVID-19 was done using Natural Language Processing (NLP) to search the CRF comment fields. A detailed explanation of the algorithm is given in Appendix 7.

# 5. BASELINE CHARACTERISTICS

## 5.1. Demographics and Other Baseline Characteristics

For the Induction Studies (Cohorts A and B), subject demographic variables and other baseline characteristics will be summarized by treatment group and overall using descriptive statistics for continuous variables and using the number and percentage of subjects for categorical variables. The summary of demographic data will be provided for the Safety Analysis Set.

- Age (years, on the date of first dose of the study drug)
- Age group ( $< 65 \text{ years}, \ge 65 \text{ years}$ )
- Sex at birth (female, male)
- Race
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Geographic region (United States [US], non-US)
- Weight
- Height
- Body mass index (BMI; in kg/m<sup>2</sup>)
- Smoking status (former, current, never)

For the Maintenance Study, the same demographic variables will be summarized by treatment group and overall. Baseline age from the Induction Study will be used for the Maintenance Study.

A by-subject demographic listing, including the informed consent date, will be provided by subject ID number in ascending order.

#### **5.2.** Baseline Disease Characteristics

For the Induction Studies (Cohorts A and B) and Maintenance Study, the following baseline disease characteristics will be summarized for the Safety Analysis Sets using descriptive statistics for continuous variables, and using number and percentage of subjects for categorical variables:

- Duration of CD (years) from date of diagnosis to first dosing date of study drug
- Duration of CD (< 1 year,  $\geq$  1 to < 3 years,  $\geq$  3 to < 7 years,  $\geq$  7 years)

- CDAI score (Induction Studies only)
- PRO2 subscores: liquid or very soft stool subscore and abdominal pain subscore (Induction Studies only)
  - Liquid or very soft stool subscore  $\geq 4$
  - Abdominal pain subscore (0 = None, 1 = Mild, 2 = Moderate, 3 = Severe)
  - Abdominal pain subscore  $\geq 2$
  - Liquid or very soft stool subscore  $\geq 4$  and abdominal pain subscore  $\geq 2$
- Total PRO2 score (Induction Studies only)
- Total SES-CD score (Induction Studies only)
- Number of available segments with SES-CD at Induction baseline
- Location of CD based on SES-CD at Induction baseline: ileum only, colon only, ileum and colon
- Complications of CD:
  - Fistula (yes, no)
  - Stricture (yes, no)
  - Abscess (yes, no)
- History of surgeries due to CD (yes, no)
- CCI
- CCI
- CCI
- CCI
- CD treatment history
  - Prior use of systemic corticosteroids (yes, no)
  - Prior use of immunomodulators (yes, no)
  - Number of prior exposures to biologic agent  $(0, 1, 2, \ge 3)$  as listed in Appendix 2

- Prior use of TNF- $\alpha$  antagonist as listed in Appendix 2 (yes, no) and for subjects with prior use:
  - Number of TNF-α antagonists used
    - 0 1
    - 0 2
    - $\circ \geq 3$
  - Worst outcome of prior use of TNF-α antagonist
    - Treatment failure
    - o Intolerance, including both allergic and non-allergic intolerance
    - o Other
- Prior use of vedolizumab (yes, no) and for subjects with prior use:
  - Worst outcome of prior use of vedolizumab
    - Treatment failure
    - Intolerance, including both allergic and non-allergic intolerance
    - Other
- Prior use of both TNF-α antagonist and vedolizumab (yes, no)
- Prior use of ustekinumab (yes, no) and for subjects with prior use:
  - Worst outcome of prior use of ustekinumab
    - Treatment failure
    - o Intolerance, including both allergic and non-allergic intolerance
    - o Other

<u>Note</u>: The worst outcome of a prior treatment is treatment failure, followed by intolerance, and then other outcomes.

- Prior failure of both TNF-α antagonist and vedolizumab
  - Yes (dual refractory, defined as those who have failed at least 2 classes of biologic therapies [any TNF-α antagonist and vedolizumab])
    - United States (US)/Korea Males
    - Subjects other than US/Korea Males

- No
  - US/Korea Males
  - Subjects other than US/Korea Males
- Concomitant treatment at baseline (or maintenance baseline for Maintenance Study)
  - Concomitant use of systemically absorbed corticosteroid and/or immunomodulator at baseline/maintenance baseline, including: a) systemically absorbed corticosteroid only, b) immunomodulator only, c) both, and d) neither;
  - Prednisone equivalent dose for subjects who are on systemically absorbed corticosteroid at baseline/maintenance baseline (mg/day)
  - Prednisone equivalent dose for subjects who are on systemically absorbed corticosteroid at baseline/maintenance baseline (> 0 to 10 mg/day, > 10 to 20 mg/day, > 20 30 mg/day, > 30 mg/day)
  - Concomitant use of 5-aminosalicylates (yes, no) at baseline/maintenance baseline

In addition, another baseline characteristics table for Maintenance Study using the FAS will be generated, including the above baseline characteristics except those marked as "Induction Studies only" and the following additional variables:

- CDAI score at maintenance baseline
- PRO2 subscores at maintenance baseline: abdominal pain and liquid or very soft stool subscores
- Total PRO2 score at Week 10
- Total SES-CD score at Week 10
- Clinical remission by CDAI (yes, no) at Week 10
- Clinical response by CDAI (yes, no) at Week 10
- Clinical remission by PRO2 (yes, no) at Week 10
- Endoscopic response (yes, no) at Week 10



# 5.3. Medical History

Medical history (disease-specific and general conditions) and IBD family history data will be collected at screening and presented in data listings.

General medical history data will be coded using the current version of Medical Dictionary for Regulatory Activities (MedDRA).

# 6. EFFICACY ANALYSES

#### 6.1. General Considerations

The efficacy analysis will be conducted on the FAS, defined in Section 3.1.2, unless otherwise specified.

The definitions of selected efficacy endpoints for each individual study (Cohort A Induction, Cohort B Induction, and Maintenance) are provided in Table 6-1. While the endoscopy will be read by both study site investigator and central reader, only the centrally-read endoscopic data will be used in the calculations of SES-CD scores and other related efficacy endpoints.

Appendix 6 includes a detailed definition of study treatment failure and the corresponding data handling rules for efficacy analysis.

Table 6-1. Definitions of Selected Efficacy Endpoints

| | | | 75.07.44 |
|---|---|---|---|
| Study | Type | Endpoint | Definition |
| Induction | EU: secondary<br>Non-EU: Co-primary | Clinical remission by<br>CDAI at Week 10 | CDAI score < 150 points at Week 10 |
| Induction | Co-primary | Endoscopic response at<br>Week 10 | ≥ 50% reduction from baseline in total SES-CD score at Week 10 based on central reading |
| Induction | EU: co-primary<br>Other: Secondary | Clinical remission by<br>PRO2 at Week 10 | Abdominal pain score ≤ 1 (on a scale of 0 to 3) and liquid or very soft stool (Bristol stool scale type 6 or 7) frequency ≤ 3 at Week 10 |
| Induction | Secondary | Clinical response by<br>CDAI at Week 10 | Reduction in CDAI score from Induction<br>baseline by at least 100 points or CDAI score<br>< 150 at Week 10 |
| Induction | CCI | CCI | CCI |
| Induction | EU: Secondary<br>Non-EU: CC | Both clinical remission by<br>PRO2 and endoscopic<br>response at Week 10 | Clinical remission by PRO2 and endoscopic response at Week 10 combined into a single endpoint on a patient level |
| Induction | CCI | CCI | CCI |
| Induction | CCI | CCI | CCI |
| Induction | CCI | CCI | CCI |
| Maintenance | Co-primary | Clinical remission by<br>CDAI at Week 58 | CDAI score < 150 points at Week 58 |

| Study | Type | Endpoint | Definition |
|---|---|---|---|
| Maintenance | Co-primary | Endoscopic response at<br>Week 58 | ≥ 50% reduction from Induction baseline in<br>total SES-CD score at Week 58 based on<br>central reading |
| Maintenance | Secondary | Clinical remission by<br>PRO2 at Week 58 | Abdominal pain score ≤ 1 (on a scale of 0 to 3) and liquid or very soft stool (Bristol stool scale type 6 or 7) frequency ≤ 3 at Week 58 |
| Maintenance | Secondary | Clinical response by<br>CDAI at Week 58 | Reduction in CDAI score from Induction<br>baseline by at least 100 points or CDAI score<br>< 150 at Week 58 |
| Maintenance | Non-EU: secondary | Sustained clinical<br>remission by CDAI at<br>Weeks 10 and 58 | Clinical remission by CDAI at both Week 10<br>and Week 58 |
| Maintenance | Non-EU: secondary | 6-month Corticosteroid-<br>free clinical remission by<br>CDAI at Week 58 | Clinical remission by CDAI with no corticosteroid use for the indication of CD for at least 6 months prior to Week 58 among subjects who are on corticosteroid at maintenance baseline (baseline of Maintenance Study). Subjects who weaned off steroids but required re-initiation within 6 months prior to Week 58 assessment will be considered to have not met this endpoint. |
| Maintenance | Secondary | Sustained clinical<br>remission by PRO2 at<br>Weeks 10 and 58 | Clinical remission by PRO2 at both Week 10 and Week 58 |
| Maintenance | Secondary | 6-month Corticosteroid-<br>free clinical remission by<br>PRO2 at Week 58 | Clinical remission by PRO2 with no corticosteroid use for the indication of CD for at least 6 months prior to Week 58 among subjects who are on corticosteroid at maintenance baseline (baseline of Maintenance Study). Subjects who weaned off steroids but required re-initiation within 6 months prior to Week 58 assessment will be considered to have not met this endpoint. |
| Maintenance | CCI | CCI | single endpoint on a patient level |
| Maintenance | EU: secondary<br>Non-EU: CC | Both clinical remission by<br>PRO2 and endoscopic<br>response at Week 58 | Clinical remission by PRO2 and endoscopic response at Week 58 combined into a single endpoint on a patient level |
| Maintenance | CCI | CCI | CCI |
| Maintenance | CCI | CCI | CCI |
| Maintenance | CCI | CCI | CCI |

CD = Crohn's Disease; CDAI = Crohn's Disease Activity Index; PRO2 = patient reported outcome consisting of 2 items: abdominal pain severity and liquid stool frequency; SES-CD = Simple Endoscopic Score for Crohn's Disease

Subjects who achieve either clinical remission by PRO2 or endoscopic response at Week 10 will be eligible to be re-randomized into the Maintenance Study.

# **Summary of Dichotomous Efficacy Endpoints**

For the Cohort A Induction Study, the Cohort B Induction Study, and the Maintenance Study, numbers and percentages of subjects achieving each of the dichotomous efficacy endpoints defined above, and numbers and percentages of subjects not achieving those endpoints for the following reasons will be summarized by treatment, in a hierarchy order with the first reason being the highest.

- 1) Data censored due to initiation or change of rescue medication
- 2) Subjects who do not meet the endpoint based on observed data
- 3) Subjects who do not meet the endpoint due to study drug discontinuation led by protocol-specified disease worsening (Maintenance Study only)
- 4) Subjects who do not have sufficient measurements to determine the endpoint due to study drug discontinuation for other reasons
- 5) Subjects who do not have sufficient measurements to determine the endpoint for other reasons

## **Non-Responder Imputation**

For analysis of all the above defined efficacy endpoints in Table 6-1, subjects who do not have sufficient measurements due to any reason (eg, study treatment failure, early study discontinuation) to determine the endpoint will be considered non-responders (ie, non-responder imputation).

#### 6.1.1. Calculation of CDAI and PRO2 Scores

The CDAI system is a composite index of 8 disease activity variables with scores ranging from 0 to over 600 based upon a composite of symptoms (eg, abdominal pain), signs (the presence of abdominal mass and weight), laboratory values (eg, hematocrit), and physician assessment amongst others. The CDAI has 3 PRO components: liquid or very soft stool frequency, abdominal pain, and general wellbeing. The clinical remission by CDAI endpoint is defined by the total CDAI score, calculated as a weighted sum of all 8 component subscores. If subjects have 3 or more of the 8 component subscores missing, then the subjects will be considered as having insufficient data to determine response status and their total CDAI score will be considered missing. If subjects have 1 or 2 CDAI components missing, then the missing component will be imputed by the LOCF method using the previous valid component score from the most recent analysis visit (ie, use the component score from Week 6 for missing

component at Week 10, or use the component score from Week 50 for missing component at Week 58. Scores from other post Induction baseline visits will not be used). If the component score from the most recent analysis visit is also missing, the missing value will be imputed with the corresponding component score at Induction baseline.

The PRO2 has 2 patient reported outcome components: liquid or very soft stool frequency subscore and abdominal pain subscore. If either subscore is missing, no imputation will be done, and the subject will be considered as having insufficient data to determine clinical remission status by PRO2 (or total PRO2 score) and treated as not meeting clinical remission. The clinical remission by PRO2 (or total PRO2 score) is defined by the PRO2 subscores as specified in Table 6-1.

For further information on the CDAI/PRO2 and calculation rules at screening and post-screening, reference is made to Appendix 3.

# 6.1.2. Calculation of SES-CD and Other Endoscopy Endpoints

The total SES-CD will be calculated at Screening (used as the baseline), Week 10, and Week 58. It is the sum of the values of the 4 variables (size of ulcers, ulcerated surface, affected surface and presence of narrowings) for 5 bowel segments (ileum, right colon, transverse colon, left colon and rectum). The detailed subscores for each variable of SES-CD are given in Appendix 5.

# **Endoscopic Response**

For each of the 5 bowel segments, if the subscore of a segment is missing at baseline, this segment will not be included in the calculation of the total SES-CD for all the visits for the purpose of evaluating endoscopic response. If the subscore of a segment is observed at baseline but missing at Week 10 (or Week 58), it will be imputed using a score of 12 (worst subscore from the sum of the 4 variables in a segment). This is the primary approach to impute missing data in a segment.

If the percentage reduction from baseline in total SES-CD is  $\geq$  50%, then the subject will be defined as achieving endoscopic response.

If the above criteria are not met, the subject will be considered as not achieving endoscopic response.





# 6.1.3. COVID-19 Impact on Primary Efficacy Endpoints

The number of subjects with the following categories due to COVID-19 will be summarized by treatment at Week 10 for Induction Studies and at Week 58 for Maintenance Study.

- Missed visit (including out of efficacy analysis window, as defined in Section 3.8.2)
- Delayed visit (occurring after the upper limit of the efficacy analysis visit window, as defined in Section 3.8.2)

For CDAI assessments, the number of subjects with the following categories due to COVID-19 will be summarized by treatment at Week 10 for Induction Studies and at Week 58 for Maintenance Study.

- Number of missed components (including out of analysis window, as defined in Section 3.8.2)
- Number of delayed components (occurring after the upper limit of the analysis visit window, as defined in Section 3.8.2)
- Number of virtually or locally conducted components. Only the following 3 components may
  be conducted virtually or locally: use of anti-diarrheal medications, hematocrit (from local
  laboratory), and weight (at home).

For SES-CD assessments, the number of subjects with the following categories due to COVID-19 will be summarized by treatment at Week 10 for Induction Studies and at Week 58 for Maintenance Study.

Missed ileocolonoscopy (including out of analysis window, as defined in Section 3.8.2)

• Delayed ileocolonoscopy (occurring after the upper limit of the analysis visit window, as defined in Section 3.8.2)

# 6.2. Primary Efficacy Endpoints

# 6.2.1. Definition of the Primary Efficacy Endpoints

## **EU-specific**:

The co-primary efficacy endpoints are the proportion of subjects achieving clinical remission by PRO2 at Week 10 and the proportion of subjects achieving endoscopic response at Week 10 for each Induction Study (Cohorts A and B), and the proportion of subjects achieving clinical remission by PRO2 at Week 58 and the proportion of subjects achieving endoscopic response at Week 58 for the Maintenance Study. Refer to Table 6-1 for the endpoint definitions.

#### Other (non-EU):

The co-primary efficacy endpoints are the proportion of subjects achieving clinical remission by CDAI at Week 10 and the proportion of subjects achieving endoscopic response at Week 10 for each Induction Study (Cohorts A and B), and the proportion of subjects achieving clinical remission by CDAI at Week 58 and the proportion of subjects achieving endoscopic response at Week 58 for the Maintenance Study. Refer to Table 6-1 for the endpoint definitions.

# 6.2.2. Statistical Hypotheses for the Primary Efficacy Endpoints

For each Induction Study (Cohorts A and B), the primary analysis will compare a filgotinib dose group to placebo on the proportion of subjects achieving clinical remission by CDAI at Week 10 and on the proportion of subjects achieving endoscopic response at Week 10. The primary statistical hypotheses at Weeks 10 for each Induction Study are listed in Section 3.5.2.1.

Similarly, for the Maintenance Study, the primary analysis will compare a filgotinib dose group to placebo among the subjects from Cohort A and Cohort B Induction Studies combined being treated with the same filgotinib dose in Induction Studies on the proportion of subjects achieving clinical remission by CDAI at Week 58 and on the proportion of subjects achieving endoscopic response at Week 58. The primary statistical hypotheses at Weeks 58 for the Maintenance Study are listed in Section 3.5.2.2.

For EU-specific analyses, for a filgotinib dose group to demonstrate a significant treatment effect over placebo, statistical significance needs to be achieved on both clinical remission by PRO2 and endoscopic response endpoints at the significance level as specified in Section 3.5. For other (non-EU) analyses, for a filgotinib dose group to demonstrate a significant treatment effect over placebo, statistical significance needs to be achieved on both clinical remission by CDAI and endoscopic response endpoints.

# 6.2.3. Estimands for the Primary Efficacy Endpoints

The EU-specific co-primary endpoints are:

- Clinical remission by PRO2
- Endoscopic response

The other (non- EU) co-primary endpoints are:

- Clinical remission by CDAI
- Endoscopic response

# 6.2.3.1. Clinical Remission by PRO2

The ICH E9 (R1) guidance {U. S. Department of Health & Human Services (DHHS) 2021} specifies that an estimand is characterized by five attributes (the treatment, the population, the subject level endpoint, handling of intercurrent events, and the population level summary).

Based on the definitions of the different types of estimands in the ICH E9 (R1), our primary estimate of clinical remission by PRO2 endpoint will use a composite estimand (Table 6-2). A second composite estimand is also proposed as a sensitivity analysis (Table 6-3).

Table 6-2. Composite Estimand 1 (Primary Analysis) for Clinical Remission by PRO2

| Attributes | Composite Estimand 1 |
|---|---|
| Treatment | Filgotinib 200 mg, filgotinib 100 mg, or placebo |
| Population | Full Analysis Set as defined in Section 3.1.2 |
| | PRO2 clinical remission status (Yes/No) at Week 10 for Induction Studies and at Week 58 for Maintenance Study |
| Subject level endpoint | If abdominal pain score ≤ 1 and liquid or very soft stool frequency ≤ 3, then the subject will be defined as achieving clinical remission at Week 10 or at Week 58, respectively. If the above remission criterion is not met or the PRO2 (any component) is missing, the subject will be considered as not achieving clinical remission by PRO2. |
| Handling of missing data due to intercurrent events | Subjects who meet treatment failure criteria (ie, take potentially effective medications other than study treatment as defined in Appendix 6) or prematurely discontinue from the study without available assessment result are considered as not achieving clinical remission by PRO2 |
| Population-level summary | Difference in proportions in clinical remission by PRO2, comparing a filgotinib dose group to placebo group |

Table 6-3. Composite Estimand 2 (Sensitivity Analysis) for Clinical Remission by PRO2

| Attributes | Composite Estimand 2 |
|---|---|
| Treatment | Filgotinib 200 mg, filgotinib 100 mg, or placebo |
| Population | Full Analysis Set as defined in Section 3.1.2 |
| Subject-level endpoint | PRO2 clinical remission status (Yes/No) at Week 10 for Induction Studies and at Week 58 for Maintenance Study |

| | If abdominal pain score ≤ 1 and liquid or very soft stool frequency ≤ 3, then the subject will be defined as achieving clinical remission at Week 10 or at Week 58, respectively. If the above remission criterion is not met, the subject will be considered as not achieving clinical remission by PRO2. If PRO2 is missing (any subcomponent), then data will be analyzed using MICE as outlined in section 6.2.5. |
|---|---|
| Handling of missing data due to intercurrent events | Subjects who meet treatment failure criteria (ie, take potentially effective medications other than study treatment as defined in Appendix 6) or prematurely discontinue from the study without available assessment result are considered as not achieving clinical remission by PRO2 |
| Population-level summary | Difference in proportions in clinical remission by PRO2, comparing a filgotinib dose group to placebo group |

# 6.2.3.2. Clinical Remission by CDAI

The ICH E9 (R1) guidance {U. S. Department of Health & Human Services (DHHS) 2021} specifies that an estimand is characterized by five attributes (the treatment, the population, the subject level endpoint, handling of intercurrent events, and the population level summary). Because the 8 components of CDAI come from different data sources, the CDAI data may have missing data at component level (only some components are missing) as well as at subject level (all 8 components are missing). Because of this complication, the definition of the estimand is expanded to include 2 additional attributes in addition to the 5 delineated above. These 2 additional attributes are: (1) the component level endpoint; and (2) the handling of missing data at component level endpoint.

Using this expanded definition of an estimand and based on the definitions of the different types of estimands in the ICH E9 (R1), our primary estimate of clinical remission by CDAI endpoint will use a composite estimand (Table 6-4). For this composite estimand (estimand 1), the handling of missing data will be expanded to the component level in addition to the subject level. A second composite estimand is also proposed as a sensitivity analysis (Table 6-5).

Table 6-4. Composite Estimand 1 (Primary Analysis) for Clinical Remission by CDAI

| Attributes | Composite Estimand 1 |
|---|---|
| Treatment | Filgotinib 200 mg, filgotinib 100 mg, or placebo |
| Population | Full Analysis Set as defined in Section 3.1.2 |
| Component-level endpoint | CDAI subscore for each component at Week 10 for Induction Studies and at Week 58 for Maintenance Study |
| Subject-level endpoint | CDAI clinical remission status (Yes/No) at Week 10 for Induction Studies and at Week 58 for Maintenance Study |
| | If CDAI < 150, then the subject will be defined as achieving clinical remission at Week 10 or at Week 58, respectively. If the above remission criterion is not met |

| | or the CDAI is missing, the subject will be considered as not achieving clinical remission by CDAI. |
|---|---|
| Handling of missing data (component-level endpoint) | If the subscore for 1 or 2 components are missing at Week 10 (or Week 58), then the subscore will be imputed using LOCF imputation method (see Section 6.1.1). If the subscores for 3 or more components are missing, then missing subscores will not be imputed, and the CDAI will be considered missing. |
| Handling of missing data due to intercurrent events (subject-level endpoint) | Subjects who meet treatment failure criteria (ie, take potentially effective medications other than study treatment as defined in Appendix 6) or prematurely discontinue from the study without available assessment result are considered as not achieving clinical remission by CDAI |
| Population-level summary | Difference in proportions in clinical remission by CDAI, comparing a filgotinib dose group to placebo group |

CDAI = Crohn's Disease Activity Index; LOCF = last observation carried forward

Table 6-5. Composite Estimand 2 (Sensitivity Analysis) for Clinical Remission by CDAI

| Attributes | Composite Estimand 2 |
|---|---|
| Treatment | Filgotinib 200 mg, filgotinib 100 mg, or placebo |
| Population | Full Analysis Set as defined in Section 3.1.2 |
| Subject-level endpoint | CDAI clinical remission status (Yes/No) at Week 10 for Induction Studies and at Week 58 for Maintenance Study |
| | If CDAI < 150, then the subject will be defined as achieving clinical remission at Week 10 or at Week 58, respectively. If the above remission criterion is not met, the subject will be considered as not achieving clinical remission by CDAI. If the CDAI is missing, then data will be analyzed using MICE as outlined in section 6.2.5. |
| Handling of missing data due to intercurrent events (subject-level endpoint) | Subjects who meet treatment failure criteria (ie, take potentially effective medications other than study treatment as defined in Appendix 6) or prematurely discontinue from the study without available assessment result are considered as not achieving clinical remission by CDAI |
| Population-level summary | Difference in proportions in clinical remission by CDAI, comparing a filgotinib dose group to placebo group |

CDAI = Crohn's Disease Activity Index

# 6.2.3.3. Endoscopic Response

Intercurrent events can impact subjects at the segment level (eg, stricture) or at the subject level (eg, early termination of the study) for SES-CD data. Similar to the estimand for clinical remission by CDAI, the definition of the estimand for endoscopic response is expanded to include 2 additional attributes. These 2 additional attributes are: (1) the segment level outcome to be measured; and (2) the handling of intercurrent events impacting the segment.

Using this expanded definition of an estimand and based on the definitions of the different types of estimands in the ICH E9(R1) guidance, the primary estimate of endoscopic response endpoint

will use a composite estimand (Table 6-6). A second composite estimand is also proposed as a sensitivity analysis (Table 6-7). For each estimand, the handling of missing data due to the intercurrent events will be expanded to the segment level in addition to the subject level.

Table 6-6. Composite Estimand 1 (Primary Analysis) for Endoscopic Response

| Attributes | Composite Estimand 1 |
|---|---|
| Treatment | Filgotinib 200 mg, filgotinib 100 mg, or placebo |
| Population | Full Analysis Set as defined in Section 3.1.2 |
| Segment-level outcome to be measured | SES-CD subscore for each segment at baseline and Week 10 for Induction<br>Studies and at Week 58 for Maintenance Study |
| | Endoscopic response status (Yes/No) at Week 10 for Induction Studies and at Week 58 for Maintenance Study |
| Subject-level outcome to be measured | If the percentage reduction of total SES-CD from Induction baseline is ≥ 50%, then the subject will be defined as achieving endoscopic response at Week 10 or at Week 58, respectively. If the above responder criterion is not met or total SES-CD is missing, the subject will be considered as not achieving endoscopic response. |
| Measure of intervention effect<br>& handling of missing data due<br>to intercurrent events<br>(segment-level outcome) | If the subscore of a segment is missing at baseline, this segment will not be included in the calculation of the total SES-CD for all the visits. If the subscore of a segment is observed at baseline, but missing at Week 10 or Week 58, it will be imputed using a score of 12 (worst subscore from the sum of the 4 variables in a segment). |
| Measure of intervention effect<br>& handling of missing data due<br>to intercurrent events (subject-<br>level outcome) | Subject who met treatment failure criteria (ie, take potentially effective medications rather than study treatment as defined in Appendix 6) or prematurely discontinued from study without available assessment result is considered a non-responder. |
| Population-level summary measure | Difference in proportions in endoscopic response, comparing a filgotinib dose group to placebo group |

SES-CD = Simple Endoscopic Score for Crohn's Disease

Table 6-7. Composite Estimand 2 (Sensitivity Analysis) for Endoscopic Response

| Attributes | Composite Estimand 2 |
|---|---|
| Treatment | Filgotinib 200 mg, filgotinib 100 mg, or placebo |
| Population | Full Analysis Set as defined in Section 3.1.2 |
| Segment-level outcome to be measured | SES-CD subscore for each segment at baseline and Week 10 for Induction<br>Studies and at Week 58 for Maintenance Study |
| Subject-level outcome to be measured | Endoscopic response status (Yes/No) at Week 10 for Induction Studies and at Week 58 for Maintenance Study |
| | If the percentage reduction of total SES-CD from Induction baseline is ≥ 50%, then the subject will be defined as achieving endoscopic response at |

| | Week 10 or at Week 58, respectively. If the above responder criterion is not met, the subject will be considered as not achieving endoscopic response. If total SES-CD is missing, then data will be analyzed using MICE as outlined in section 6.2.5. |
|---|---|
| Measure of intervention effect & handling of missing data due to intercurrent events (segment-level outcome) | All segments will be included in the total SES-CD calculation regardless of being missing or not. |
| Measure of intervention effect & handling of missing data due to intercurrent events (subject-level outcome) | Subject who met treatment failure criteria (ie, take potentially effective medications rather than study treatment as defined in Appendix 6) or prematurely discontinued from study without available assessment result is considered a non-responder. |
| Population-level summary measure | Difference in proportions in endoscopic response, comparing a filgotinib dose group to placebo group |

SES-CD = Simple Endoscopic Score for Crohn's Disease

# 6.2.4. Primary Analysis of the Primary Efficacy Endpoints

Primary analysis will be conducted according to the composite estimand 1 specified in Section 6.2.3.

For the individual Induction Studies (Cohort A and Cohort B), a stratified Cochran-Mantel-Haenszel (CMH) test will be used to compare the treatment effect between a filgotinib dose group (eg, 200 mg) and placebo. The CMH tests will be stratified by the following factors:

# Cohort A Induction Study:

- Number of prior exposures to biologic agent (0, 1, > 1) as listed in Appendix 2
- Concomitant use of oral, systemically absorbed corticosteroids at Day 1
- Concomitant use of immunomodulators at Day 1

#### Cohort B Induction Study:

- Number of prior exposures to biologic agent ( $\leq 1, > 1$ ) as listed in Appendix 2
- Concomitant use of oral, systemically absorbed corticosteroids at Day 1
- Concomitant use of immunomodulators at Day 1

For the Maintenance Study, a stratified CMH test will be used to compare the treatment effect between a filgotinib dose group and placebo among the subjects from Induction Cohorts A and B combined being treated with the same dose of filgotinib. The CMH test will be stratified by the following factors:

- History of exposure to a biologic agent, (Yes or No)
- Concomitant use of oral, systemically absorbed corticosteroids at maintenance baseline
- Concomitant use of immunomodulators at maintenance baseline

Stratification factors based on the clinical database will be used for the analysis. The stratified CMH chi-square p-value for each of the above comparison will be provided. Strata with low numbers of subjects might be aggregated for the analysis. The 2-sided 95% CI of clinical remission rate by CDAI and endoscopic response rate based on normal approximation method with a continuity correction will be provided for each treatment group. In addition, stratified proportion difference along with its 95% 2-sided CI using stratum-adjusted Mantel-Haenszel (MH) approach {Koch 1989} for each comparison will be provided as follows:

The stratified point estimates for difference in proportion of subjects achieving an endpoint between each filgotinib (F) treatment group and the placebo (P) group will be calculated following formula (1).

$$\hat{p}_F - \hat{p}_P = \frac{\sum W_h d_h}{\sum W_h} \tag{1}$$

where  $d_h = \hat{p}_{Fh} - \hat{p}_{Ph}$  is the difference in the proportion of subjects who achieved the endpoint between the filgotinib group and the placebo group in stratum h (h = 1, 2, ..., K), and  $W_h = \frac{n_{Fh}n_{Ph}}{n_{Fh}+n_{Ph}}$  is the weight based on the harmonic mean of sample size per treatment group for each stratum where  $n_{Fh}$  and  $n_{Ph}$  are the sample sizes of the filgotinib group and the placebo group in stratum h, respectively.

The 95% stratum-adjusted MH CIs will be calculated following formula (2).

$$\hat{p}_F - \hat{p}_P \pm Z_{1-\alpha/2} \cdot SE(\hat{p}_F - \hat{p}_P) \tag{2}$$

Where 
$$SE(\hat{p}_F - \hat{p}_P) = \frac{\sqrt{\sum W_h^2 \left(\frac{\hat{p}_{Fh}^*(1-\hat{p}_{Fh}^*)}{n_{Fh}-1} + \frac{\hat{p}_{Ph}^*(1-\hat{p}_{Ph}^*)}{n_{Ph}-1}\right)}}{\sum W_h}$$
,  $\hat{p}_{Fh}^* = \frac{m_{Fh} + 0.5}{n_{Fh} + 1}$ ,  $\hat{p}_{Ph}^* = \frac{m_{Ph} + 0.5}{n_{Ph} + 1}$ , and  $m_{Fh}$  and

 $m_{Ph}$  are the number of subjects who achieved the endpoint from the filgotinib group and the placebo group in stratum h, respectively.  $Z_{(1-\alpha/2)}$  is the 97.5% percentile of normal distribution with  $\alpha = 0.05$ .

If the computed lower confidence bound is less than -1, the lower bound is defined as -1. If the computed upper confidence bound is greater than 1, then the upper bound is defined as 1.

The significance level specified in Section 3.5 will be used to declare a statistically significant treatment effect for a filgotinib dose group.

Bar charts of the proportions of subjects achieving clinical remission by PRO2 (EU), CDAI (non-EU) and endoscopic response at Week 10 (for the Induction Studies) and Week 58 (for the Maintenance Study) will be provided by treatment group with corresponding p-values.

In addition, the proportion of subjects with percentage reduction of  $\geq 25\%$  from Induction baseline in total SES-CD score will be summarized for Week 10 (Induction Studies) and Week 58 (Maintenance Study), respectively. The number of available segments with SES-CD score at baseline and Week 10, and change from baseline at Week 10 for Induction Studies will be summarized. Similarly, the number of available segments with SES-CD score at Induction baseline and Week 58, and change from Induction baseline at Week 58 for Maintenance Study will be summarized. The score for each segment will be displayed in a data listing. If there is a missing segment score, the reason of missingness (if available) will be included.

# 6.2.5. Sensitivity Analyses for the Primary Efficacy Endpoints

# 6.2.5.1. Clinical Remission by PRO2 (EU-specific)

Sensitivity analysis will be conducted according to the composite estimand 2 specified in Section 6.2.3.

The multivariate imputation by chained equations (MICE) {Azur 2011} through regression model will be used to impute each missing subscore in PRO2. For Induction Studies, each subscore in PRO2 at baseline, Weeks 2, 4, 6, and 10, treatment, and stratification factors will be included in the imputation model using the Full Analysis Set. For the Maintenance Study, each subscore in PRO2 at maintenance baseline, Weeks 14, 20, 26, 34, 42, 50, and 58, treatment, and stratification factors will be included in the imputation model using the Full Analysis Set among the subjects from Induction Cohorts A and B combined being treated with the same dose of filgotinib.

For each imputed dataset, the clinical remission status by PRO2 will be derived. The subjects who met treatment failure criteria or prematurely discontinued from the study without available result from the study will be set as not achieving clinical remission in each imputed dataset. The parameters of interest for each imputed dataset will be estimated using a similar method as the primary approach. The results from multiple imputations will be combined using Rubin's rule {Rubin 1987}.

In addition, tipping point analysis with delta-adjusting pattern-mixture approach {Ratitch 2013} will be conducted to assess the robustness of analysis result under the MNAR (missing not at random) assumption. The proposed method will perform a series of analyses after adjusting for stratification factors with a range of different values of the shift parameter  $\delta$  applied to the imputed datasets at which the conclusion about the statistical significance of result will be altered. Specifically, the analysis is characterized by two-dimensional sequences (one sequence associated with missing data in the placebo group and the other associated with missing data in the filgotinib group). In the first step for both sequences, the missing data in both treatment groups are imputed under the missing at random (MAR) assumption. For each subsequent step of the placebo sequence, the missing data are imputed assuming incrementally more favorable than in the previous step of that sequence while holding the shift parameter constant in the filgotinib

group. Similarly, for each subsequent step of the filgotinib group sequence, the missing data are imputed assuming incrementally less favorable than in the previous step of that sequence while holding the shift parameter constant in the placebo group.

Appendix 8 provides sample SAS model statements for the tipping point analysis. Each  $\delta$  value is classified as either "altering the statistical significance conclusion" or "keeping the statistical significance conclusion unchanged." The tipping points that alter the statistical significance conclusion will be provided. The same analysis method for the primary analysis as specified in Section 0 will be applied when analyzing the adjusted data generated under different  $\delta$  values.

## 6.2.5.2. Clinical Remission by CDAI (other: non-EU)

Sensitivity analysis will be conducted according to the composite estimand 2 specified in Section 6.2.3.

The multivariate imputation by chained equations (MICE) {Azur 2011} through regression model will be used to impute the missing CDAI. If the subscore for at least 1 component is missing, then the CDAI is considered missing. For Induction Studies, the CDAI at baseline, Weeks 2, 4, 6, and 10, treatment, and stratification factors will be included in the imputation model using the Full Analysis Set. For the Maintenance Study, the CDAI at maintenance baseline, Weeks 14, 20, 26, 34, 42, 50, and 58, treatment, and stratification factors will be included in the imputation model using the Full Analysis Set among the subjects from Induction Cohorts A and B combined being treated with the same dose of filgotinib.

For each imputed dataset, the clinical remission status by CDAI will be derived. The subjects who met treatment failure criteria or prematurely discontinued from study without available result from study will be set as not achieving clinical remission in each imputed dataset. The parameters of interest for each imputed dataset will be estimated using a similar method as the primary approach. The results from multiple imputations will be combined using Rubin's rule {Rubin 1987}.

In addition, tipping point analysis with delta-adjusting pattern-mixture approach {Ratitch 2013} will be conducted to assess the robustness of analysis result under the MNAR (missing not at random) assumption. The proposed method will perform a series of analyses after adjusting for stratification factors with a range of different values of the shift parameter  $\delta$  applied to the imputed datasets at which the conclusion about the statistical significance of result will be altered. Specifically, the analysis is characterized by two-dimensional sequences (one sequence associated with missing data in the placebo group and the other associated with missing data in the filgotinib group). In the first step for both sequences, the missing data in both treatment groups are imputed under the missing at random (MAR) assumption. For each subsequent step of the placebo sequence, the missing data are imputed assuming incrementally more favorable than in the previous step of that sequence while holding the shift parameter constant in the filgotinib group. Similarly, for each subsequent step of the filgotinib group sequence, the missing data are imputed assuming incrementally less favorable than in the previous step of that sequence while holding the shift parameter constant in the placebo group.

Appendix 8 provides sample SAS model statements for the tipping point analysis. Each  $\delta$  value is classified as either "altering the statistical significance conclusion" or "keeping the statistical significance conclusion unchanged." The tipping points that alter the statistical significance conclusion will be provided. The same analysis method for the primary analysis as specified in Section 6.2.4 will be applied when analyzing the adjusted data generated under different  $\delta$  values.

# 6.2.5.3. Endoscopic Response

Sensitivity analysis will be conducted according to the composite estimand 2 specified in Section 6.2.3.

The MICE {Azur 2011} through regression model will be used to impute the missing segmental subscores. For Induction Studies, the segmental score at baseline and Week 10, treatment, and stratification factors will be included in the imputation model using the FAS. For the Maintenance Study, the segmental score at maintenance baseline and Week 58, treatment, and stratification factors will be included in the imputation model using the Full Analysis Set among the subjects from Induction Cohorts A and B combined being treated with the same dose of filgotinib.

For each imputed dataset, the percentage change from Induction baseline in the total SES-CD score will be calculated for each subject and the endoscopic response status will be derived. The subjects who met treatment failure criteria or prematurely discontinued from study without available result will be set as non-responders in each imputed dataset. The parameters of interest for each imputed dataset will be estimated using a similar method as the primary approach. The results from multiple imputations will be combined using Rubin's rule {Rubin 1987}.

In addition, tipping point analysis with delta-adjusting pattern-mixture approach {Ratitch 2013} will be conducted to assess the robustness of analysis result under the MNAR (missing not at random) assumption (see Section 6.2.5.1).

# 6.2.5.4. Clinical remission by PRO2 and Endoscopic Response

A cross tabulation will be created showing number and proportion of subjects with response at Week 58 (clinical remission and endoscopic response, clinical remission by PRO2 only, endoscopic response only, and no endoscopic response and no clinical remission by PRO2) by outcome at Week 10: clinical remission by PRO2 and endoscopic response, clinical remission by PRO2 alone, clinical endoscopic response only, and no endoscopic response and no clinical remission by PRO2). This table will be based on the Safety Analysis Set.

# 6.2.6. Analysis of the Primary Efficacy Endpoints for Japan Submission

The following analysis will be conducted as the primary analysis for evaluating the co-primary endpoints for the filgotinib 200 mg dose group in each Induction Study in order to support a Japanese marketing application.

Given the restriction in the US/Korea of only allowing dual refractory males to receive filgotinib 200 mg, there exists an inherent imbalance in each Induction Study between subjects randomized to filgotinib 200 mg and the placebo group with respect to US/Korea non-dual refractory males who will only be present in the placebo group, but not in the filgotinib 200 mg group. Recognizing this imbalance and the theoretical potential for non-dual refractory subjects to have better disease prognosis and a higher chance of response, an analysis excluding US/Korea non-dual refractory males from the placebo group in the FAS for each Induction Study will be conducted. Similar analysis method as specified in Section 6.2.4 will be used for the treatment comparison between the filgotinib 200 mg and the placebo group on clinical remission by CDAI and endoscopic response at Week 10.

The primary analysis to support Japanese marketing application to evaluate efficacy of the filgotinib 100 mg dose group in each Induction Study will still be based on all the subjects in the FAS.

# 6.2.7. Subgroup Analyses for the Primary and key secondary Efficacy Endpoints

The following subgroup analyses of the primary efficacy endpoints will be performed for each individual study (Cohort A Induction, Cohort B Induction, and Maintenance).

Subgroups based on study stratification factors include:

# **Cohort A Induction Study Stratification Factors:**

- Number of prior exposures to biologic agent as listed in Appendix 2  $(0, \ge 1)$
- Concomitant use of oral, systemically absorbed corticosteroids at Day 1 (yes, no)
- Concomitant use of immunomodulators at Day 1 (yes, no)

# **Cohort B Induction Study Stratification Factors:**

- Number of prior exposures to biologic agent as listed in Appendix 2 ( $\leq 1, \geq 1$ )
- Concomitant use of oral, systemically absorbed corticosteroids at Day 1 (yes, no)
- Concomitant use of immunomodulators at Day 1 (yes, no)

#### Cohort A and B Induction Studies Combined for Prior Exposure to Biologic Agent

• Number of prior exposures to biologic agent as listed in Appendix 2  $(0, \ge 1)$ 

# **Maintenance Study Stratification Factors:**

- History of exposure to a biologic agent (yes, no)
- Concomitant use of oral, systemically absorbed corticosteroids at maintenance baseline (yes, no)
- Concomitant use of immunomodulators at maintenance baseline (yes, no)

Other subgroups for each individual study include:

- Age group on the date of first dose of the study drug ( $< 65 \text{ years}, \ge 65 \text{ years}$ )
- Sex at birth (female, male)
- Race (Asian, Black or African American, White, and Other)
- Geographic region (US, non-US)
- CCI
- CCI
- Duration of CD (years from date of diagnosed to first dosing date of Induction study drug) (< 1 year, ≥ 1 to < 3 years, ≥ 3 to < 7 years, ≥ 7 years)
- Baseline disease activity (based on Induction baseline CDAI score) ( $< 300, \ge 300$ )
- Induction baseline SES-CD score ( $< 16, \ge 16$ )
- Previous exposure to TNF-α antagonist (yes, no)
- Prior TNF-α antagonist failure (yes, no)
- Previous exposure to vedolizumab (yes, no)
- Prior vedolizumab failure (yes, no)
- Dual refractory (yes, no)
- The following 4 subgroups:
  - US/Korean males who are dual refractory
  - US/Korean males who are not dual refractory
  - Non-US/Korean males (US/Korea females and subjects from countries other than US and Korea) who are dual refractory
  - Non-US/Korean males who are not dual refractory

For a subject, if the value of the grouping variable cannot be determined, this subject will be excluded from the corresponding subgroup analysis. Non-stratified risk difference between treatment groups will be evaluated for each of the subgroups using Fisher's exact test. A forest plot will graphically present the non-stratified risk difference and 95% CI using normal approximation with a continuity correction on the treatment differences (filgotinib – placebo) in each co-primary endpoint for each of the subgroups.

Additional subgroup analyses for geographic region may be added based on the distribution of study enrollment prior to study unblinding.

# 6.3. Secondary Efficacy Endpoints

# 6.3.1. Definition of the Secondary Efficacy Endpoints

#### 6.3.1.1. EU-specific

The key secondary efficacy endpoints are:

## Induction Studies (Cohorts A and B)

- The proportion of subjects achieving clinical remission by CDAI at Week 10
- The proportion of subjects achieving both clinical remission by PRO2 and endoscopic response (combined into a single endpoint on a patient level) at Week 10

#### Maintenance Study

- The proportion of subjects achieving clinical remission by CDAI at Week 58
- The proportion of subjects achieving sustained clinical remission by PRO2 at Weeks 10 and 58
- The proportion of subjects achieving both clinical remission by PRO2 and endoscopic response (combined into a single endpoint on a patient level) at Week 58
- The proportion of subjects achieving 6-month corticosteroid-free remission by PRO2 at Week 58

Refer to Table 6-1 for the endpoint definitions.

#### 6.3.1.2. Other (non-EU)

The key secondary efficacy endpoints are:

# Induction Studies (Cohorts A and B)

• The proportion of subjects achieving clinical remission by PRO2 at Week 10

The proportion of subjects achieving clinical response by CDAI at Week 10

# Maintenance Study

- The proportion of subjects achieving clinical remission by PRO2 at Week 58
- The proportion of subjects achieving clinical response by CDAI at Week 58
- The proportion of subjects achieving sustained clinical remission by CDAI at Weeks 10 and 58
- The proportion of subjects achieving 6 month corticosteroid-free clinical remission by CDAI at Week 58
- The proportion of subjects achieving sustained clinical remission by PRO2 at Weeks 10 and 58
- The proportion of subjects achieving 6 month corticosteroid-free clinical remission by PRO2 at Week 58

Refer to Table 6-1 for the endpoint definitions.

# 6.3.2. Analysis of the Secondary Efficacy Endpoints

The same primary statistical analysis method described in Section 6.2.4 for testing the primary efficacy endpoints will be utilized for testing the key secondary efficacy endpoints. The secondary efficacy endpoints will be tested in the order of clinical importance and interest and at the significance level as specified in Section 3.5.

Bar charts of the proportions of subjects achieving each of the key secondary efficacy endpoint by treatment group with corresponding p-values will be provided.














# 6.5. Cohorts A and B End-of-Induction Analysis

After all subjects from Cohorts A and B have completed the Week 10 visit or have terminated prior to Week 10 (and completed post-treatment assessments, if applicable) and corresponding data entry is complete, an End-of-Induction safety and efficacy analysis will be performed for DMC review including cumulative safety analysis and efficacy analysis on primary endpoints. Gilead blinded statistical programmers will provide the unblinded external statistician, who is independent of Gilead and not a member of Gilead's Study Management Team, with the datasets and programs necessary to complete the analysis. The unblinded external statistician will apply the unblinded treatment codes to the datasets and generate the unblinded analysis results.

Both cohorts will be examined independently by the DMC:

Taking into account data in Cohort A and Cohort B, if ALL the following 4 criteria are met for BOTH cohorts, the DMC may recommend overall study discontinuation.

- 2-sided p-value for filgotinib 200 mg vs placebo comparison is larger than 0.05 on clinical remission by CDAI at Week 10
- 2-sided p-value for filgotinib 100 mg vs placebo comparison is larger than 0.05 on clinical remission by CDAI at Week 10
- 2-sided p-value for filgotinib 200 mg vs placebo comparison is larger than 0.05 on endoscopic response at Week 10
- 2-sided p-value for filgotinib 100 mg vs placebo comparison is larger than 0.05 on endoscopic response at Week 10

If the condition above is not met from either cohort, the DMC may recommend that the study continues without modification.

## 6.6. Change from Protocol-Specified Efficacy Analyses





Subgroup analyses as defined for the co-primary endpoints, were added for all secondary endpoints.

#### 7. SAFETY ANALYSES

Unless otherwise specified, summaries of safety data will be provided for the Safety Analysis Set for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study, and will include data collected as specified below:

# <u>Induction Studies (Cohorts A and B)</u>

- No later than 30 days after the last dosing date of Induction Study, for subjects who did not take any study treatment from Maintenance Study, or
- On or before the first dosing date of Maintenance Study, for subjects who took any study treatment in Maintenance Study

#### Maintenance Study

• No later than 30 days after the last dosing date of Maintenance Study

#### 7.1. Adverse Events and Deaths

# 7.1.1. Adverse Event Dictionary

Clinical and laboratory AEs will be coded using a current version of MedDRA. System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

#### 7.1.2. Adverse Event Severity

The severity of AEs was grade using the modified Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. For each episode, the highest grade attained should be reported. If a CTCAE criterion does not exist, the adverse events are graded by the investigator as Grade 1, 2, 3, 4, or 5 according to toxicity criteria specified in the protocol. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings. The missing category will be listed last in the summary presentation.

## 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE eCRF to the question of "Related to Study Treatment." Relatedness will always reflect the investigator assessment of causality rather than the sponsor's. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-subject data listings will show the relationship as missing.

#### 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if AEs met the definitions of SAE specified in the study protocol. SAEs captured and stored in the clinical database will be reconciled with the safety database before data finalization.

# 7.1.5. Treatment-Emergent Adverse Events

# 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

# Induction Studies (Cohorts A and B)

- Any AEs with an onset date on or after the study drug start date for each Induction Study (Day 1) and
  - No later than 30 days after the last dosing date of Induction Study, for subjects who did not take any study treatment from Maintenance Study, or
  - Before the first dosing date of Maintenance Study, for subjects who took any study treatment in Maintenance Study
- Any AEs leading to premature discontinuation of Induction Study drug

#### Maintenance Study

- Any AEs with an onset date on or after the study drug start date for the Maintenance Study and no later than 30 days after last dosing date of Maintenance Study
- Any AEs leading to premature discontinuation of Maintenance Study drug

# 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dosing date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment-emergent. For first dosing date and last dosing date defined for Induction Studies (Cohorts A and B) and Maintenance Study, please refer to Section 3.8.1. The event is considered treatment-emergent if <u>both</u> of the following 2 criteria are met:

# <u>Induction Studies (Cohorts A and B)</u>

- The AE onset date is the same as or after the month and year (or year) of the first dosing date of study drug, and
- The AE onset date is the same as or before the month and year (or year) of the date corresponding to
  - 30 days after the last dosing date of Induction Study, for subjects who did not take any study treatment in Maintenance Study, or
  - The day before the first dosing date of Maintenance Study, for subjects who took any study treatment in Maintenance Study

#### Maintenance Study

- The AE onset date is the same as or after the month and year (or year) of the first dosing date of Maintenance Study, and
- The AE onset date is the same as or before the month and year (or year) of the date corresponding to 30 days after the last dosing date of Maintenance Study

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dosing date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and an incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dosing date of study drug will be considered treatment emergent.

#### 7.1.6. Summaries of Adverse Events and Deaths

Treatment-emergent AEs will be summarized based on the Safety Analysis Set for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study.

No formal statistical testing is planned.

#### 7.1.6.1. Summaries of AE Incidence

The number and percentage of subjects who experienced at least 1 TEAE will be provided and summarized by SOC, HLT, PT, and treatment group. For other AEs described below, summaries will be provided by SOC, PT, and treatment group:

- TEAEs of Grade 3 or higher (by maximum severity)
- TEAEs of Grade 2 or higher (by maximum severity)
- All TE treatment-related AEs
- TE treatment-related AEs of Grade 3 or higher (by maximum severity)

- TE treatment-related AEs of Grade 2 or higher (by maximum severity)
- All TE SAEs
- All TE treatment-related SAEs
- All TEAEs leading to premature discontinuation of study drug
- All TEAEs leading to premature discontinuation of study
- All TE SAEs leading to death (ie, outcome of death)
- All TEAEs leading to temporary dose interruption of study drug

A brief, high-level summary of AEs described above will be provided by treatment group presenting the number and percentage of subjects who reported the above AEs. All deaths observed in the study will be also included in this summary.

Multiple events will be counted only once per subject in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC and HLT within each SOC (if applicable), and then by PT in descending order of total frequency within each SOC. In addition, a summary of all AEs occurring at least 2% of subjects will be summarized by SOC and PT in order of descending frequency. For summaries by severity grade, the most severe grade will be used for those AEs that occurred more than once in an individual subject during the study.

In addition, the following tables will be generated and summarized by PT only, in descending order of total frequency:

- TEAEs
- TEAEs of Grade 3 or higher
- TEAEs of Grade 2 or higher
- TE SAEs
- TE treatment-related AEs
- TE treatment-related SAEs
- TEAEs leading to premature discontinuation of study drug

Data listings will be provided for the following:

- All AEs, indicating whether the event is treatment-emergent
- All AEs of Grade 3 or higher
- All AEs of Grade 2 or higher
- SAEs
- Deaths
- All AEs leading to death (ie, outcome of death)
- AEs leading to premature discontinuation of study drug
- AEs leading to premature discontinuation of study
- AEs leading to dose temporary interruption of study drug
- AEs related to COVID-19, as determined by the COVID-19 Standardised MedDRA Query (SMQ) narrow search

In addition, an XML file will be created to support EUDRACT reporting containing serious AEs, non-serious AEs and non-serious AEs occurring in at least 5% of subjects in at least one treatment arm, either at a system organ class level or at PT level (this XML file will be created in-house).

#### 7.1.7. Adverse Events of Interest

Adverse events of interest (AEI) include infections, malignancies (excluding nonmelanoma skin cancers), nonmelanoma skin cancers, gastrointestinal perforations, major adverse cardiovascular events (MACE), and thromboembolic events. Summaries of the following treatment-emergent AEI will be produced to enhance the analysis of safety data.

- Events of infections, presented in the following subcategories:
  - AEs of infections, utilizing all AEs in the MedDRA Infections and Infestations SOC
  - AEs of serious infections, using all AEs in the MedDRA Infections and Infestations SOC that are classified as SAEs
  - AEs of herpes zoster, utilizing an MST list developed by the Sponsor
  - AEs of opportunistic infections (SMQ), utilizing a narrow scope PTs

- AEs of malignancies, excluding nonmelanoma skin cancers, utilizing an MST list developed by the Sponsor
- AEs of nonmelanoma skin cancers, utilizing an MST list developed by the Sponsor
- AEs of gastrointestinal perforations, utilizing an MST list developed by the Sponsor
- AEs of MACE, utilizing a positively adjudicated event list, presented in the following subcategories (Section 7.1.7.1):
  - Cardiovascular (CV) death
  - Non-fatal myocardial infarction (MI)
  - Non-fatal stroke
- AEs of arterial systemic thromboembolism (ASTE), utilizing a positively adjudicated event list (Section 7.1.7.1)
- AEs of venous thromboembolism (VTE), utilizing a positively adjudicated event list (Section 7.1.7.1)

A list of all AE PTs is provided in Appendix 9.

The number and percentage of subjects with a reported event will be summarized for each treatment group by PT for each AEI category. A data listing for each category of AEI will also be provided.

A by-subject listing for subjects with potential events for adjudication. For each AE, it will be described if the AE was adjudicated for a specific category (cardiovascular death, myocardial infarction, stroke, arterial systemic thromboembolism and venous thromboembolism) and their respective adjudication results (NA if not adjudicated for a specific category) will be provided.

A by-subject listing of thromboembolic history and risk factors will be provided for subjects with potential events for adjudication (MACE, ASTE, and VTE).

# 7.1.7.1. Cardiovascular Safety Endpoint Adjudication Committee

An independent cardiovascular safety endpoint adjudication committee (CVEAC) will be formed to periodically review and adjudicate all potential MACE and thromboembolic events in a blinded manner. To identify potential MACE and thromboembolic events, the following AEs will be sent for adjudication. Please refer to the Cardiovascular Event Adjudication Charter for more details.

All AEs leading to death

- CV events (meeting seriousness criteria), utilizing an MST list developed by the Sponsor
- MI, utilizing a narrow scope SMQ
- Unstable angina (meeting hospitalization criteria), utilizing an MST list developed by the Sponsor
- Transient ischemic attack, utilizing an MST list developed by the Sponsor
- Stroke, utilizing an MST list developed by Sponsor
- Cardiac failure (meeting hospitalization criteria), utilizing an MST list developed by the Sponsor
- Percutaneous coronary intervention, utilizing an MST list developed by the Sponsor
- Embolic and thrombotic events, utilizing a narrow scope SMQ

The CVEAC will review the above AEs, and related clinical data to adjudicate whether the criteria for MACE (CV death, MI, and/or stroke), ASTE, and VTE have been met for each AE.

# 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the Safety Analysis Set for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study.

The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7. Test results from hemolyzed samples will not be included in the analysis, but they will be listed in by-subject laboratory listings.

A by-subject listing for laboratory test results will be provided by subject ID number and time point in chronological order for hematology, serum chemistry, urinalysis, lipid profile, and serum immunoglobulin separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the Common Terminology Criteria for Adverse Events (CTCAE) severity grade will be flagged in the data listings, as appropriate.

Hematocrit results collected from local laboratories due to COVID-19 impact will not be included in the safety laboratory summary but will be included in the listing with a flag to indicate which records were collected at local laboratories.

No formal statistical testing is planned.

#### 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics will be provided by treatment group for each laboratory test specified in the study protocol within hematology and chemistry panels, and also laboratory tests from lipids panel (under fasting status) including total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides, non-HDL cholesterol (total cholesterol minus HDL cholesterol), LDL/HDL ratio, and total immunoglobulin (Ig), IgA, IgM, and IgG, as follows for each Induction Study:

- Baseline values
- Values at each postbaseline time point
- Change from baseline at each postbaseline time point

In addition, descriptive statistics for the laboratory tests described from above will be provided by treatment group for the Maintenance Study:

- maintenance baseline values
- Values at each postbaseline time point after maintenance baseline
- Change from maintenance baseline at each postbaseline time point after maintenance baseline

A baseline laboratory value will be defined as the last measurement obtained on or prior to the date of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the visit value minus the baseline value. A maintenance baseline laboratory value will be defined as the last measurement obtained on or prior to the date of first dose of study drug for the Maintenance Study, and change from maintenance baseline will be defined as the visit value minus the maintenance baseline value. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; SD values will be displayed to the reported number of digits plus 1.

Median (Q1, Q3) of the observed change from baseline (or maintenance baseline) values for aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, alkaline phosphatase, serum creatinine, creatinine clearance, creatine phosphokinase, white blood cell count, absolute neutrophils, absolute lymphocytes, hemoglobin, platelets, fasting total cholesterol, fasting LDL, fasting HDL, total Ig, IgG, IgA and IgM, will be plotted using a line plot by treatment group and visit.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

# 7.2.2. Graded Laboratory Values

Modified CTCAE 4.03 (see Appendix 6 of the protocol) will be used for assigning toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (ie, increased, decreased) will be presented separately.

## 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

# <u>Induction Studies (Cohorts A and B)</u>

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, and

- No later than 30 days after the last dosing date of Induction Study, for subjects who did not take any study treatment from Maintenance Study, or
- On or before the first dosing date of Maintenance Study, for subjects who took any study treatment in Maintenance Study

#### Maintenance Study

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from maintenance baseline at any post maintenance baseline time point after first dosing date of Maintenance Study, no later than 30 days after the last dosing date of Maintenance Study drug.

# 7.2.2.2. Treatment-Emergent Marked Laboratory Abnormalities

#### Induction Studies (Cohorts A and B)

Treatment-emergent marked laboratory abnormalities are defined as values that increase at least 3 toxicity grades from baseline at any postbaseline time point, and

- No later than 30 days after the last dosing date of Induction Study, for subjects who did not take any study treatment from the Maintenance Study, or
- On or before the first dosing date of Maintenance Study, for subjects who took any study treatment in the Maintenance Study

#### Maintenance Study

Treatment-emergent marked laboratory abnormalities are defined as values that increase at least 3 toxicity grades from maintenance baseline at any post maintenance baseline time point after the first dosing date of Maintenance Study, no later than 30 days after the last dosing date of Maintenance Study.

# 7.2.2.3. Summaries of Laboratory Abnormalities

Laboratory data that are categorical will be summarized using the number and percentage of subjects in the study with the given response at baseline and each scheduled postbaseline time point for Cohort A Induction Study, Cohort B Induction Study, and at maintenance baseline and each scheduled time point after maintenance baseline for Maintenance Study.

The following summaries (number and percentage of subjects) for treatment-emergent laboratory abnormalities will be provided by laboratory test and treatment group for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study. Subjects will be categorized according to the most severe postbaseline abnormality grade for a given laboratory test:

- Graded laboratory abnormalities
- Grade 3 or higher laboratory abnormalities
- Marked laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of subjects with nonmissing postbaseline values.

A by-subject listing of treatment-emergent Grade 3 or 4 laboratory abnormalities will be provided by subject ID number and time point in chronological order. This listing will include all test results that were collected throughout the study for the laboratory test of interest, with all applicable severity grades displayed.

# 7.2.3. Liver-Related Laboratory Evaluations

Liver-related abnormalities after initial study drug dosing will be examined and summarized using the number and percentage of subjects who were reported to have the following laboratory test values for postbaseline measurements for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study:

- AST: (a) > 3 times of upper limit of the normal range (ULN); (b) > 5 × ULN;
   (c) > 10 × ULN; (d) > 20 × ULN
- ALT: (a)  $> 3 \times ULN$ ; (b)  $> 5 \times ULN$ ; (c)  $> 10 \times ULN$ ; (d)  $> 20 \times ULN$
- AST or ALT  $> 3 \times ULN$  and total bilirubin  $> 2 \times ULN$

For individual laboratory tests, subjects will be counted once based on the most severe postbaseline values. For both the composite endpoint of AST or ALT and total bilirubin, subjects will be counted once when the criteria are met at the same postbaseline visit date. The denominator is the number of subjects in the Safety Analysis Set who have nonmissing postbaseline values of all relevant tests at the same postbaseline visit date. A listing of subjects who met at least 1 of the above criteria will be provided.

# 7.2.4. Complete Blood Count-Related Laboratory Evaluations

Complete blood count-related abnormalities such as anemia, leucopenia, neutropenia, lymphopenia, and thrombocytopenia after initial study drug dosing will be examined and summarized using the number and percentage of subjects who were reported to have the following laboratory test values for postbaseline measurements for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study, respectively.

The list of laboratory tests to be examined is:

- Hemoglobin
- White blood cell count
- Absolute neutrophil count
- Lymphocyte count
- Platelet count

For each of the above laboratory test, the following will be summarized:

- Postbaseline worsening CTCAE grade from baseline
- Baseline value of less than Grade 3 and increase to Grade 3 or 4 at worst postbaseline
- Baseline value of less than Grade 3 and increase to Grade 4 at worst postbaseline

For Maintenance Study, maintenance baseline will be used in the summaries described above.

#### 7.2.5. Shifts Relative to the Baseline Value

Shift tables will be presented by showing change in CTCAE grade for hemoglobin, platelet count, white blood cell count, absolute lymphocyte count, absolute neutrophils, triglycerides, and total cholesterol.

Shift tables will be presented by showing change in lab normal range (low, normal, and high) for hematocrit, absolute monocyte count, absolute eosinophil count, and absolute basophil count. In addition, shift tables for fasting LDL and HDL will be presented using the following National Cholesterol Education Program (NCEP) ATP III categories {National Cholesterol Education Program (NCEP) 2001}:

- For LDL (mg/dL):  $< 100, 100-129, 130-159, 160-189, and \ge 190$
- For HDL (mg/dL):  $< 40, \ge 40$  to  $< 60, \text{ and } \ge 60$

In all shift tables, the number and proportion of subjects for each category of each laboratory result will be summarized by its baseline/maintenance baseline category for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study.

For Induction Studies, shift tables will be presented for Week 10. For Maintenance Study, shift tables will be presented for Weeks 26 and 58.

# 7.3. Body Weight and Vital Signs

Descriptive statistics will be provided by treatment group for body weight, BMI and vital signs (resting blood pressure [systolic blood pressure and diastolic blood pressure], respiratory rate, pulse, and temperature) as follows for each Induction Study:

- Baseline value
- Values at each postbaseline time point
- Change from baseline at each postbaseline time point

In addition, descriptive statistics will be provided by treatment group for the Maintenance Study as follows:

- Maintenance baseline values
- Values at each time point after maintenance baseline
- Change from maintenance baseline at each time point after maintenance baseline

A baseline value will be defined as the last available value collected on or prior to the date of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value. A maintenance baseline value will be defined as the last measurement obtained on or prior to the date of first dose of study drug for the Maintenance Study, and change from maintenance baseline will be defined as the visit value minus the maintenance baseline value. Body weight and vital signs measured at unscheduled visits will be included for the baseline/maintenance baseline value selection.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3. No formal statistical testing is planned.

A by-subject listing of vital signs will be provided by subject ID number and time point in chronological order. Body weight, height, and BMI will be included in the vital signs listing, if space permits. If not, they will be provided separately.

Body weight results measured by subjects at home from virtual visits due to COVID-19 impact will not be included in the vital signs summary, but will be included in the listing with a flag to indicate which records were collected at home.

#### 7.4. Prior and Concomitant Medications

Medications reported at screening and during the study will be coded using the current version of the World Health Organization (WHO) Drug dictionary.

#### 7.4.1. Prior Medications

Prior medications are defined as any medication taken before a subject took the first dose of Induction Study drug for Induction Studies, and the first dose of Maintenance Study drug for Maintenance Study.

General prior and CD-specific prior medications will be summarized separately by preferred name using the number and percentage of subjects for each treatment group and overall. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered by 2<sup>nd</sup> WHO ATC level and PT in descending overall frequency (for both ATC level and PT). For drugs with the same frequency, sorting will be done alphabetically.

For the purposes of analysis, any medication with a start date prior to the first dosing date of study drug will be included in the prior medication summary regardless of when the stop date is. If a partial start date is entered the medication will be considered prior unless the month and year (if day is missing) or year (if day and month are missing) of the start date are after the first dosing date. Medications with a completely missing start date will be included in the prior medication summary, unless otherwise specified.

Summaries will be based on the Safety Analysis Set for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study. No formal statistical testing is planned.

#### 7.4.2. Concomitant Medications

General concomitant and CD-specific concomitant medications are defined as medications taken while a subject took study drug. Use of concomitant medications will be summarized by 2<sup>nd</sup> WHO ATC level and preferred name using the number and percentage of subjects in descending overall frequency (for both ATC level and PT). For drugs with the same frequency, sorting will be done alphabetically. A subject reporting the same medication more than once will be counted only once when calculating the number and percentage of subjects who received that medication. The summary will be ordered by PT in descending overall frequency. For drugs with the same frequency, sorting will be done alphabetically.

First dosing date and last dosing date for Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study are defined in Section 3.8. For the purposes of analysis, any medication with a start date prior to or on the first dosing date of study drug and continued to take after the first dosing date, or started after the first dosing date but prior to or on the last dosing date of study drug will be considered concomitant medications. Medications started and stopped on the same day as the first dosing date or the last dosing date of study drug will also be considered concomitant. Medications with a stop date prior to the date of first dosing date of study drug or a start date after the last dosing date of study drug will be excluded from the concomitant

medication summary. If a partial stop date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) prior to the date of first study drug administration will be excluded from the concomitant medication summary. If a partial start date is entered, any medication with the month and year (if day is missing) or year (if day and month are missing) after the study drug stop date will be excluded from the concomitant medication summary. Medications with completely missing start and stop dates will be included in the concomitant medication summary, unless otherwise specified. Summaries will be based on the Safety Analysis Set. No formal statistical testing is planned.

All prior and concomitant medications (other than per-protocol study drugs) will be provided in a by-subject listing sorted by subject ID number and administration date in chronological order.

# 7.5. Electrocardiogram Results

A shift table of the investigators' assessment of ECG results at each visit compared with baseline (or maintenance baseline) values will be presented by treatment group for each Induction Study and Maintenance Study, using the following categories: normal; abnormal, not clinically significant; abnormal, clinically significant. The number and percentage of subjects in each cross-classification group of the shift table will be presented. Subjects with a missing value at baseline (or maintenance baseline) or postbaseline will not be included in the denominator for percentage calculation.

No formal statistical testing is planned.

A by-subject listing for ECG assessment results will be provided by subject ID number and time point in chronological order.

# 7.6. Other Safety Measures

A data listing will be provided for subjects who become pregnant during the study.

## 7.7. Changes from Protocol-Specified Safety Analyses

The following overall (Induction and Maintenance) safety analysis, indicated in the protocol, will not be conducted for this study. Details of the pooled analyses will be specified in the analysis plan for integrated safety summary.

## Overall (Induction and Maintenance)

All safety data collected on or after the first dose of study drug administration for the entire study (Day 1) up to 30 days after permanent discontinuation of study drug will be summarized by treatment group according to the study drug received.

# 8. PHARMACOKINETIC ANALYSES

The pharmacokinetic analyses are detailed in the pharmacokinetic analysis plan (PKAP) (see appendix 10).

Additional PK analysis may be performed and exposure-response relationships may be explored.



## 10. REFERENCES

- Azur MJ, Stuart EA, Frangakis C, Leaf PJ. Multiple Imputation by Chained Equations: What is it and how does it work? International journal of methods in psychiatric research 2011;20 (1):9.
- Bretz F, Maurer W, Brannath W, Posch M. A Graphical Approach to Sequentially Rejective Multiple Test Procedures. Stat Med 2009;28:586-604.
- Daperno M, D'Haens G, Van Assche G, Baert F, Bulois P, Maunoury V, et al. Development and validation of a new, simplified endoscopic activity score for Crohn's disease: the SES-CD. Gastrointestinal endoscopy 2004;60 (4):505-12.
- Khanna R, Zou G, D'Haens G, Feagan BG, Sandborn WJ, Vandervoort MK, et al. A retrospective analysis: the development of patient reported outcome measures for the assessment of Crohn's disease activity. Aliment Pharmacol Ther 2015;41 (1):77-86.
- Koch GG, Carr GJ, Amara IA, Stokes ME, Uryniak TJ. Categorical Data Analysis. Chapter 13 in Berry, D.A. (ed.). Statistical Methodology in the Pharmaceutical Sciences. New York: Marcel Dekker, Inc., 1989:pp. 414-21.
- National Cholesterol Education Program (NCEP). Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) Executive Summary. National Institute of Health May, 2001.
- Ratitch B, O'Kelly M, Tosiello R. Missing data in clinical trials: from clinical assumptions to statistical analysis using pattern mixture models. Pharm Stat 2013;12 (6):337-47.
- Rubin DB. Multiple Imputation for Nonresponse in Surveys. New York, NY: John Wiley & Sons, Inc; 1987.
- Sandborn WJ, Feagan BG, Hanauer SB, Lochs H, Lofberg R, Modigliani R, et al. A review of activity indices and efficacy endpoints for clinical trials of medical therapy in adults with Crohn's disease. Gastroenterology 2002;122 (2):512-30.
- U. S. Department of Health & Human Services (DHHS), Food and Drug Administration (FDA), Center for Drug Evaluation amd Research (CDER), Center for Biologic Evaluation and Research (CBER). E9(R1) Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials. Guidance for Industry. Revision 1. May. 2021.

# 11. SOFTWARE

SAS® Software Version 9.4 (SAS Institute Inc., Cary, NC, USA) is to be used for all programming of tables, listings, and figures.

nQuery + nTerim Version 4.0 (Statistical Solutions, Cork, Ireland) was used for sample size and power calculation.

# 12. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| Original Final Draft<br>(7 September 2016) | | | |
| | 1.1, 1.2 | Modified to include biologic-experienced subjects in cohort A | To be consistent with the most updated protocol |
| | 1.3, 3.5 | Modified multiple testing strategy to<br>allow alpha recycling between the two<br>tested filgotinib doses | To be consistent with the most updated protocol |
| | 3.1 | Modified definition for Per-Protocol<br>Analysis Sets | To better conduct Per-Protocol analysis |
| | 3, 7 | Added Cohorts A and B pooled safety summary | To support safety evaluation of study<br>drug across Induction Studies |
| Final Draft 0.2 | 3, 7 | Clarified overall safety summaries only include adverse events and laboratory abnormalities including data collected across Cohort A Induction Study, Cohort B Induction Study and Maintenance Study | To support safety evaluation of study<br>drug across Induction and Maintenance<br>Studies |
| (13 March 2019) | 5 | Modified the list of variables to be<br>summarized in baseline characteristic<br>tables | To provide better characterization of the investigated patient populations |
| | CCI | CCI | To support the primary and secondary endpoints |
| | 7 | Clarified AEs of interest to be summarized | To better address safety concerns |
| | 7 | Added summary of complete blood count-related laboratory evaluations | To better address safety concerns |
| | Appendix 1 | Updated Schedule of Assessments | To align with the most updated Protocol<br>Amendment |
| | Global | Administrative and editorial changes<br>have been made throughout the SAP,<br>where appropriate | To improve clarity and consistency |

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| | 1.1, 1.2, 1.3, | Modified study objectives randomization stratification factors for Induction Cohort A and Maintenance Study, study power and some of the efficacy endpoints | To be consistent with the most updated protocol |
| | 3.1.3, 7.1, 7.2 | Deleted overall (Induction and<br>Maintenance) safety analysis set and<br>corresponding analysis for AE and<br>laboratory results | To focus on the purpose of this SAP, which is to conduct analyses separately for each study (Induction Cohort A, Induction Cohort B, and Maintenance). Any details about pooled analyses will be specified in the analysis plan for the integration safety summary. |
| | 3.5 | Modified the alpha control strategy | To be consistent with the most updated protocol |
| | 3.9, 4, 6.1.3,<br>7.2, 7.3,<br>Appendix 7 | Added assessment of COVID-19 impact | To better understand the COVID-19 impact on subject disposition and missing data |
| | 4.2, 7 | Deleted extent of study drug exposure<br>and safety analysis for Cohorts A and B<br>combined | To better streamline CSR process and will conduct these analyses in the integrated safety summary when appropriate |
| | 6.1.1 | Modified the LOCF method to impute<br>the missing CDAI components by using<br>only available values from two visits:<br>most recent analysis visit or Induction<br>baseline | To use a more conservative approach per FDA feedback |
| Final Draft 0.3 | 6.1.2 | Modified the imputation method for SES-CD by using the worst score | To use a more conservative and reasonable approach per FDA feedback |
| (01 April 2021) | 6.2.3 | Added estimands | To clearly state the strategy to handle intercurrent events |
| | 6.2.4 | Used stratum-adjusted proportion<br>difference estimate and corresponding<br>95% CI instead of non-stratified<br>proportion difference estimate and<br>corresponding 95% CI | To be consistent with the way how the p-value is generated (stratified CMH test) |
| | 6.3.3, 6.2.5 | Deleted some imputation methods on missing data as sensitivity analyses | Some of these imputation methods are not the best strategies to handle intercurrent events in the estimands framework for the study |
| | 6.5 | Modified the criteria to stop the study<br>based on End of Induction Analysis<br>results | To be consistent with the most updated protocol |
| | 6.5 | Deleted the language regarding Gilead Executive team to review the End of Induction analysis results in parallel with DMC review | To better protect the integrity of the study data and reduce potential bias in final analysis |
| | 7.1 | Deleted subgroup analysis for adverse events | To better streamline CSR process and will conduct these analyses in the integrated safety summary when appropriate |
| | 7.1.7 | Added adverse event of interest for MACE, ASTE, and VTE based on positively adjudicated events by the cardiovascular safety endpoint adjudication committee | To be consistent with the most updated protocol |

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| | Appendix 7<br>to 12 | Deleted the list of preferred terms for<br>each category of adverse events of<br>interest in Appendix 7 to 12 in previous<br>version | To reduce the burden to keep track of<br>the list of preferred terms due to<br>MedDRA up-versioning. The lists will<br>be provided in the CSR. |
| | Appendix 7 | Added appendix for determining missing and virtual visits due to COVID-19 | To provide details of the determination algorithm |
| | Global | Administrative and editorial changes<br>have been made throughout the SAP,<br>where appropriate | To improve clarity and consistency |
| | 3.8.3 | Added the data handling rule for shift tables in safety endpoints | To use a conservative rule for shift tables in safety endpoints |
| | 4.1 | Added key study dates table | To provide information for the clinical study report |
| | 4.5 | Added overall assessment of COVID-19 impact | To address the overall COVID-19 impact at subject level |
| | 5.2 | Added summary of each abdominal pain subscore | To better assess the baseline characteristics of the analysis population |
| | 5.2 | Added the number of available segments with SES-CD score for Maintenance study | In response to comments from FDA |
| Version 1.0 | 6.2.4 | Added summary of the number of<br>available segments with SES-CD score at<br>Induction baseline and post Induction<br>baseline, and change from Induction<br>baseline | In response to comments from FDA |
| (07 February 2022) | 6.2.5 | Added tipping point analysis as a<br>sensitivity analysis for the primary<br>endpoints | To assess the robustness of analysis result under the MNAR (missing not at random) assumption. |
| | CCI | CCI | CCI |
| | Appendix 8 | Added the SAS programming for the tipping point analysis for binary endpoint | To provide clear guidance on the tipping point analysis |
| | Global | Editorial changes or clarification<br>languages have been provided<br>throughout the SAP, where appropriate | To improve clarity and consistency |
| Version 2.0<br>(xx January 2022) | Global | This SAP is a combination of the SAP for submission within EU and the SAP for submission outside EU. Objectives for both regions and corresponding analyses methods are combined in this SAP | To have one SAP covering all regions |
| | 3.4 and 6.2.7 | Add subgroups for key secondary endpoints in addition to the co-primary endpoints | To further explore consistency of the results |

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| | 3.8.2 | Gaps between analyses visit windows were removed by extending the windows | To make sure all data is included in the analyses |
| | 4.2.1 | Improved on the calculation of extent of exposure | To cover all possible scenarios of (partially) missing data |
| | 4.2.2 | Modified the calculation of treatment<br>adherence + modified the treatment<br>adherence categories | To be able to summarize overdoses |
| | 4.3 | Removed tabulation of minor protocol deviations | Because the database will not allow this summary |
| | 4.5<br>7.1.6 | Remove overall assessment of COVID-<br>19 pandemic impact<br>Added a listing on the COVID-19 related<br>AEs | To avoid duplication in the listings. All aspects of the removed listing were covered in other more detailed listings, except for the COVID-19 AEs, for which a listing was added in section 7.1.6 |
| | 5.2 | Add additional categories for baseline prednisone equivalent dose | To better characterize baseline prednisone equivalent dose |
| | 6.2.5.4 | Added a cross-tabulation of CDAI remission and SES-CD response at Week 58 versus Week 10 | Not all subjects entering the Maintenance study achieved CDAI remission. The cross-tabulation was added to explore those subjects |
| | 6.2.7 | - Added subgroup for prior exposure to biologic agents in Cohorts A and B combined - subgroup on number of prior exposure combined categories with low numbers for Cohort A | Cohort A includes both subjects with and without prior experience to biologic agents. Cohort B only has subjects with prior exposure. Therefore, the best comparison between those with and without treatment experience is the comparison combining both Cohorts. To avoid subgroups with very low numbers |
| | 6.6 | Updated to include all changes to protocol-specific efficacy analyses | Because the list was incomplete |
| | 7.1.6 | Added a summary of AEs with prespecified cut-off added a listing for COVID-19 related AEs | - To streamline CSR writing (table with<br>cut-off in the body of the CSR and the<br>complete table in the CSR appendices)<br>- to describe all aspects of the pandemic |
| | 7.4 | Change the sorting order of prior and concomitant therapies | To streamline CSR writing |
| | 8<br>Appendix 10 | Description of PK analyses replaced by the PKAP in appendix 10 Additional PK parameters were added | To allow for a better flow of the SAP To characterize the pharmacokinetics in more detail |
| | Appendix 9 | Add the list of preferred terms based on the latest MeDRA version | Even though previously removed to reduce the burden of updating the list with each MedDRA up-versioning, it was decided to put the lists back in based on the latest MedDRA version. |
| | Global | The EU-specific SAP and the SAP for non-EU submission were combined into 1 SAP | To have 1 SAP covering all submissions |

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| | Global | Editorial changes or clarification languages have been provided throughout the SAP, where appropriate | To improve clarity and consistency |

# 13. APPENDIX

| Appendix 1. | Schedule of Assessments |
|---|---|
| Appendix 2. | List of Biologics for CD Treatment |
| Appendix 3. | Crohn's Disease Activity Index (CDAI) and Patient Reported Outcomes – 2 items (PRO2) |
| Appendix 4. | Calculation of Standard Body Weight |
| Appendix 5. | Simple Endoscopic Score for Crohn's Disease (SES-CD) |
| Appendix 6. | Study Treatment Failure Rules |
| Appendix 7. | Determining Missing and Virtual Visits due to COVID-19 |
| Appendix 8. | SAS Programming for Tipping Point Analysis for Binary Endpoint |

# Appendix 1. Schedule of Assessments

| Period | Screen | | | | | | | | | | Treat | ment | | | | | | | | | Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | PTxa | ET |
| Week | | 0 | 2 | 4 | 6 | 10 | 11 | 14 | 17 | 20 | 23 | 26 | 30 | 34 | 38 | 42 | 46 | 50 | 54 | 58 | | |
| Study Day | -30 to -1 | 1 | 15 | 29 | 43 | 71 | 78 | 99 | 120 | 141 | 162 | 183 | 211 | 239 | 267 | 295 | 323 | 351 | 379 | 407 | | |
| Visit Window<br>(±) | | | ±3 | ±3 | ±3 | ±2 | ±3 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±3 | ±3 | |
| Written<br>Informed<br>Consent | X | | | | | | | | | | | | | | | | | | | | | |
| Medical History<br>&<br>Demographics | X | | | | | | | | | | | | | | | | | | | | | |
| Crohn's Disease<br>& Treatment<br>History | X | | | | | | | | | | | | | | | | | | | | | |
| 12-lead ECG | X | | | | | X | | | | | | X | | | | | | | | X | | Xb |
| Review of<br>Inclusion/<br>Exclusion<br>Criteria | Х | X | | | | | | | | | | | | | | | | | | | | |
| Complete<br>Physical Exam <sup>c</sup> | X | | | | | | | | | | | | | | | | | | | | | |
| Symptom-<br>directed Exam <sup>c</sup><br>(as needed) | | X | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | X | X |
| Vital Signs | X | X | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | X | X |
| Height | X | | | | | | | | | | | | | | | | | | | | | |
| Weight | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | X | X |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | X | X |
| Randomization | | X | | | | | X | | | | | | | | | | | | | | | |

| Period | Screen | | | | | | | | | | Treati | ment | | | | | | | | | Follow | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | PTx <sup>a</sup> | ET |
| Week | | 0 | 2 | 4 | 6 | 10 | 11 | 14 | 17 | 20 | 23 | 26 | 30 | 34 | 38 | 42 | 46 | 50 | 54 | 58 | | |
| Study Day | -30 to -1 | 1 | 15 | 29 | 43 | 71 | 78 | 99 | 120 | 141 | 162 | 183 | 211 | 239 | 267 | 295 | 323 | 351 | 379 | 407 | | |
| Visit Window<br>(±) | | | ±3 | ±3 | ±3 | ±2 | ±3 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±3 | ±3 | |
| Study Drug<br>Dispensing | | X | | X | | | X | X | | X | | X | | X | | X | | X | | | | |
| Ileocolonoscopy<br>(with Biopsies) <sup>d</sup> | X | | | | | X | | | | | | | | | | | | | | X | | |
| Local<br>Endoscopic<br>Assessment <sup>e</sup> | X | | | | | X | | | | | | | | | | | | | | X | | |
| SES-CD | X | | | | | X | | | | | | | | | | | | | | X | | |
| CDAIf | X | | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | | X |
| PRO2 <sup>f</sup> | X | | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | | X |
| Abdominal pain assessment <sup>g</sup> | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | | X |
| Anchor<br>Questions | X | | | | | | | | | | | | | | | | | | | | | |
| Patient Global<br>Impression<br>Scales <sup>h</sup> | | X | | | | X | | | | | | | | | | | | | | X | | |
| eDiary<br>instruction &<br>review <sup>i</sup> | X | X | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | |
| Stool for <i>C. diff</i> toxin, pathogenic <i>E. coli</i> , <i>Salmonella</i> spp, <i>Shigella</i> spp, <i>Campylobacter</i> spp or <i>Yersinia</i> spp testing j | X | | | | | | | | | | | | | | | | | | | | | |


| Period | Screen | | | | | | | | | | Treat | ment | | | | | | | | | Follow | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | PTxa | ET |
| Week | | 0 | 2 | 4 | 6 | 10 | 11 | 14 | 17 | 20 | 23 | 26 | 30 | 34 | 38 | 42 | 46 | 50 | 54 | 58 | | |
| Study Day | -30 to -1 | 1 | 15 | 29 | 43 | 71 | 78 | 99 | 120 | 141 | 162 | 183 | 211 | 239 | 267 | 295 | 323 | 351 | 379 | 407 | | |
| Visit Window<br>(±) | | | ±3 | ±3 | ±3 | ±2 | ±3 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±3 | ±3 | |
| Stool O&P j | X | | | | | | | | | | | | | | | | | | | | | |
| Urine drug<br>screen <sup>k</sup> | X | | | | | | | | | | | | | | | | | | | | | |
| Urinalysis | X | X | | | | X | | | | | | | | | | | | | | X | | |
| Pregnancy Test <sup>l</sup> | X | X | | X | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| TB <sup>m</sup> | X | | | | | | | | | | | | | | | | | | | | | |
| Chest x-ray n | X | | | | | | | | | | | | | | | | | | | | | |
| HBV, HCV,<br>HIV screening <sup>o</sup> | X | | | | | | | | | | | | | | | | | | | | | |
| HBV DNA<br>monitoring<br>(Japan) <sup>p</sup> | | | | X | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| HBV DNA<br>monitoring<br>(other regions) <sup>p</sup> | | | | | | X | | | | X | | | | X | | | | X | | X | | |
| Hematology | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | X | X |
| Chemistry | X | X | X | X | X | X | | X | | X | | X | | X | | X | | X | | X | X | X |
| Lipid profile (fasting) <sup>q</sup> | | X | | | | X | | | | | | X | | | | | | | | X | | X |

| Period | Screen | | | | | | | | | | Treat | ment | | | | | | | | | Follov | v-Up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | PTxa | ET |
| Week | | 0 | 2 | 4 | 6 | 10 | 11 | 14 | 17 | 20 | 23 | 26 | 30 | 34 | 38 | 42 | 46 | 50 | 54 | 58 | | |
| Study Day | -30 to -1 | 1 | 15 | 29 | 43 | 71 | 78 | 99 | 120 | 141 | 162 | 183 | 211 | 239 | 267 | 295 | 323 | 351 | 379 | 407 | | |
| Visit Window<br>(±) | | | ±3 | ±3 | ±3 | ±2 | ±3 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±3 | ±3 | |
| Serum<br>immunoglobulin | | X | | X | | X | | | | | | X | | | | | | | | X | X | X |
| Blood<br>TCR/BCR<br>repertoire<br>sample <sup>rp</sup> | | X | | X | | X | | | | | | X | | | | | | | | X | | |
| PK collection (sparse) s | | | | X | | X | | | | | | X | | | | | | | | X | | |
| CCI | İ | 1 | | | | | l | l | ı | | 1 | | 1 | 1 | ı | | ı | ı | | ı | | |
| PK substudy <sup>u</sup> | | | | 2 | X | | | | | | | | | | | | | | | | | |

- a. The Post-Treatment (PTx) visit should occur 30 days after the last dose of study drug. Only subjects who roll over into the LTE study (GS-US-419-3896/GLPG0634-CL-310) will not complete PTx assessments.
- b. For subjects who terminate prior to Week 10.
- c. A complete physical examination (PE) including, vital signs, body weight, and height will be performed at screening. A symptom directed PE may be done at other time points.
- d. Once a subject meets all other eligibility criteria (centrally calculated CDAI, PRO2 and labs), perform the screening full video ileocolonoscopy with biopsies within 14 days prior to Day 1 visit.
- e. The investigator (ie local endoscopist) may enter endoscopic assessment data based on the SES-CD in the eCRF (see Appendix 5). The locally read SES-CD score may not be used for eligibility or assessing endoscopic response for primary efficacy analysis, and it is not a substitute for the centrally read score,
- f. The screening CDAI will be used to determine subject eligibility for the study on Day 1. The CDAI patient reported outcomes of stool frequency and abdominal pain will be used to derive the PRO2 score.
- h. Patient global impression change (PGI-C) should be assessed at Weeks 10 and 58 only. Patient global impression of severity (PGI-S) should be assessed at Day 1, Weeks 10 and 58.
- i. Subjects should begin filling out the e-Diary the day of their initial screening visit and continue to fill it out throughout the remainder of the study.
- j. Stool samples should be collected to rule out infectious causes when disease worsens.
- k. Positive cocaine test disqualifies subject; positive amphetamines, barbiturates, benzodiazepines, and opioids require medical monitor review.
- 1. All females meeting the childbearing potential criteria must have a serum pregnancy testing at screening and a urine pregnancy test must be completed in clinic every 4 weeks at a minimum. If any pregnancy test is positive, study drug should be immediately interrupted and the subject should have a serum pregnancy test in clinic.
- m. Proof of no active or untreated latent TB at screening. Subjects who are diagnosed with latent TB at screening must initiate an adequate course of prophylaxis as per local standard of care for a minimum of 4 weeks prior to randomization. Subject may initiate study drug dosing only after consultation with the medical monitor.
- n. Chest x-ray (views as per local guidelines) taken at screening or within the 3 months prior to screening (with the report or films available for investigator review) without evidence of active or latent TB infection
- o. Hepatitis B surface Ag, surface Ab and core Ab, reflex HBV DNA, Hepatitis C Ab, reflex HCV RNA, HIV Ag/Ab, reflex HIV 1/2 Ab at Screening (Protocol Section 6.2.1).
- p. In Japan, subjects with negative HBsAg, positive HBcAb and/or positive HBsAb at Screening require HBV DNA monitoring every 4 weeks in accordance with local guidelines (Protocol Section 6.2.1). In other regions, subjects with negative HBsAg and positive HBcAb require HBV DNA monitoring every 3 months in accordance with local guidelines (Protocol Section 6.2.1)
- q. Fasting means no food or drink, except water, for 8 hours
- TCR: T-cell receptor; BCR: B-cell receptor.
- s. This PK sample at Weeks 10 and 58 are collected at pre-dose (within 2 hours prior to dosing). The PK sample at Week 4 is collected post-dose dose (at least 30 minutes and up to 3 hours after study drug dosing. For this visit, it is preferred that study drug dosing is in clinic. The PK sample at Week 26 can be collected at any time without regard to dosing. For these visits, the time of dose taken on the day of and the dose taken prior to the PK sample being drawn will be noted in the eCRF.
- t. 🗀
- u. Subjects who consent to optional PK substudy will have an additional plasma PK sample at any single visit from Week 2 to 10, collected pre-dose and at 0.5, 1, 2, 3, 4 and 6 hours after supervised dosing in the clinic. For all visits with PK sampling, the time of dose taken prior to and on the day of visit will be noted in the eCRF


# **Appendix 2.** List of Biologics for CD Treatment

The drug names of biologics considered as CD treatment are listed below.

| No. | Drug Class | Drug Name |
|---|---|---|
| 1 | TNF-α antagonist | Adalimumab |
| 2 | TNF-α antagonist | Certolizumab/Certolizumab Pegol |
| 3 | TNF-α antagonist | Infliximab |
| 4 | TNF-α antagonist | TNF-α antagonist biosimilar (to adalimumab,<br>Certolizumab/Certolizumab Pegol, or infliximab) |
| 5 | Integrin antagonist | Natalizumab |
| 6 | Integrin antagonist | Vedolizumab |
| 7 | Interleukin antagonist | Ustekinumab |

# Appendix 3. Crohn's Disease Activity Index (CDAI) and Patient Reported Outcomes – 2 items (PRO2)

The total CDAI score is a weighted sum of all 8 variables as specified in Table 13-1, and the PRO2 scores will be assessed according to Table 13-2 and Table 13-3. Details for the calculations of CDAI and PRO2 scores at screening and post-screening visits are provided in this appendix.

Table 13-1. Calculation of Total CDAI Score

| Variable no. | Variable | Variable description | Multiplier |
|---|---|---|---|
| 1 | Liquid or very soft stool | Daily stool count is summed for 7 days | 2 |
| 2 | Abdominal pain | Sum of 7 days of daily ratings as $0 = \text{none}$ , $1 = \text{mild}$ , $2 = \text{moderate}$ , $3 = \text{severe}$ | 5 |
| 3 | General wellbeing | Sum of 7 days of daily ratings as<br>0 = generally well, 1 = slightly below par,<br>2 = poor, 3 = very poor, 4 = terrible | 7 |
| 4 | Complications | Number of listed complications: | 20 each |
| 5 | Use of anti-diarrheal medications | Use of diphenoxylate or loperamide or other opiate for diarrhea $0 = \text{No}, 1 = \text{Yes}$ | 30 |
| 6 | Abdominal mass | 0 = none, 2 = questionable, 5 = definite | 10 |
| 7 | Hematocrit* | Males: 47 – Hct [%] Females: 42 – Hct [%] *Result must be greater than or equal to 0. If negative result enter 0 | 6 × difference |
| 8 | Weight* | Percentage deviation from standard weight (1 – weight / standard weight) × 100 *Limit of -10 (Result must be greater than or equal to -10) | 1 |
| CDAI score | | | TOTAL |

CDAI = Crohn's Disease Activity Index; Hct = hematocrit {Sandborn 2002}
Table 13-2. Calculation of PRO2 Components

| Variable no. | Variable | Variable Description |
|---|---|---|
| 1 | Liquid or very soft stool | Mean of the daily (liquid or very soft) stool count for 7 days |
| 2 | Abdominal pain | Mean of 7 days of daily ratings as 0 = none, 1 = mild, 2 = moderate, 3 = severe |

{Khanna 2015}

Each PRO2 subscore will be rounded to the nearest integer (eg, 2) in the determination of subject eligibility for the study and calculation of endpoints.

Table 13-3. Calculation of Total PRO2 score

| Variable no. | Variable | Variable Description | Multiplier |
|---|---|---|---|
| 1 | Liquid or very soft stool | Mean of the daily (liquid or very soft) stool count for 7 days | 2 |
| 2 | Abdominal pain | Mean of 7 days of daily ratings as 0 = none, 1 = mild, 2 = moderate, 3 = severe | 5 |
| Total PRO2 scoreg | | | TOTAL |

{Khanna 2015}

The 3 patient-reported outcome components for CDAI (and each subscore for PRO2) are determined using an electronic daily diary, which collects subject reported components directly. Given that the ileocolonoscopy procedure (including protocol-directed and non-protocol-directed procedures) may impact the validity of the diary data, diary data collected 1 day prior to and on the day of the procedure will not be used in the calculation of CDAI and PRO2 subscores for all visits. Those days are called non-evaluable days.

#### Calculation of CDAI and PRO2 Scores at Screening

Ileocolonoscopy is required to be performed during screening. The calculations of CDAI and PRO2 at screening are specified below:

- 1) Define T-Day 1 = subject activation date on the electronic diary device during screening
- 2) Define a 10-day window using T-Day 1 as the anchor date, and the window starts the day after T-Day 1 and ends 10 days after T-Day 1.
- 3) For each CDAI patient-reported outcome component, if there are 7 or more evaluable records within the 10-day window, take the **sum** of the 7 evaluable records closest to T-Day 1. For

each PRO2 component, take the **average** of the 7 evaluable records within the 10-day window closest to T-Day 1.

- a) If there are 4 or more (but less than 7) evaluable records within this 10-day window, the average of the available records will be taken, and then multiplied by 7 for the corresponding CDAI patient-reported component. For the corresponding PRO2 component, the average of the available records will be taken.
- b) If subjects do not have at least 4 evaluable records within this 10-day window, the corresponding CDAI patient-reported component and PRO2 component will not be calculated and will be considered as missing.

A schema of this approach and some examples are included below for further illustration:

Figure 13-1. Selection of Diary Data for the Calculation at Screening



Table 13-4. Calculation of CDAI Patient-Reported Outcome Components and PRO2 Scores at Screening

| | D | Diary Day Looking Forward from subject activation date (T-Day) | | | | | | | | Sum of 7 Days<br>(CDAI | Average<br>of | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Example | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | Days for<br>Calculation | Patient-Reported<br>Component) | 7 Days<br>(PRO2) |
| Diary<br>Subscore 1 | 1 | 2 | M | 1 | 2 | 2 | M | 0 | 1 | 2 | 2,3,5,6,7,9,10 | 9.0 | 1.3 |
| Diary<br>Subscore 2 | М | М | 1 | M | 2 | 1 | M | 2 | M | M | 4,6,7,9 | 10.5 | 1.5 |
| Diary<br>Subscore 3 | 2 | M | M | 0 | M | 2 | M | M | M | M | 2,5,7 | Missing | Missing |
| Diary<br>Subscore 4 | 1 | 2 | 1 | 1 | X | IL | 3 | 3 | 1 | 2 | 2,3,4,5,8,9,10 | 12.0 | 1.7 |

M = Missing. IL = Ileocolonoscopy day; X = non-evaluable (due to preparation for ileocolonoscopy). Days are named relative to subject activation date on electronic diary device during screening (T-Day 1). Rounding of subscores into one decimal place is for displaying purpose only. When calculating the total CDAI scores, the subscores will not be rounded.

- 4) For the non-diary components (ie, complications, use of anti-diarrheal medications, abdominal mass, hematocrit, and weight) of the CDAI, in the case of multiple records collected during screening, the value collected on the same date as T-Day 1 will be used; otherwise, the earliest valid value during screening (for re-screened subjects, most recent screening period will be used first before using previous screening period) will be used. If no valid value is available during screening, then the value on Day 1 will be used.
- 5) The CDAI total score at screening is based on a weighted sum (rounded to the nearest integer) of all 8 components (no rounding applied to the subscore for each component when calculating the CDAI total score, but the subscore will be displayed with one decimal place for displaying purpose). The weight (multiplier) of each component is specified in Table 13-1. For example, if the sum of the 7-day scores for abdominal pain is 10, then the abdominal pain CDAI subscore is 10 x 5 = 50, where 5 is the multiplier for abdominal pain. The CDAI total score will be set to 0 in the case the calculation leads to a CDAI total score of < 0.
- 6) The PRO2 subscores at screening are based on the calculation of liquid or very soft stool frequency and abdominal pain subscores individually (rounded to the nearest integer).

#### Calculation of CDAI and PRO2 Scores at Post-Screening Visits

The calculations of CDAI and PRO2 scores at post-screening visits are specified below:

- 1) CDAI and PRO2 are not assessed on Day 1 and Week 11 by the study sites, but for baseline (or maintenance baseline) summary purpose, the PRO2 subscore and Total PRO2 score will be calculated for Day 1 and Week 11. Both screening and Day 1 values will be considered for the derivation of Induction baseline for PRO2 subscores and total PRO2 score. Similarly, both Weeks 10 and 11 values will be considered for the derivation of maintenance baseline for PRO2 subscores and total PRO2 score. CDAI at Day 1 and Week 11 will not be calculated, and CDAI at screening will be Induction baseline, and at Week 10 will be maintenance baseline.
- 2) The visit date will be used as the anchor day for post-screening visits. The visit date for each analysis visit will be selected among all scheduled visits and unscheduled visits where CDAI were assessed within the analysis window as defined in Section 3.8.2. For Day 1, the date of visit from the nominal visit Day 1 will be used. Only diary data collected on evaluable days within a 10-day window which starts 10 days prior to the visit date (V-Day 1) and ends on the day prior to V-Day 1 will be used for calculation.
- 3) If there are 7 or more evaluate records within the 10-day window, take the **sum** of the 7 evaluable records closest to V-Day 1 for the corresponding CDAI subject-reported component. For the corresponding PRO2 component, take the **average** of the 7 evaluable records within the 10-day window closest to V-Day 1.
  - a) If there are 4 or more (but less than 7) evaluable records within this 10-day window, the average of the available records will be taken, and then multiplied by 7 for the corresponding CDAI patient-reported component. For the corresponding PRO2 component, the average of the available records will be taken.
  - b) If subjects do not have at least 4 evaluable records within this 10-day window, the corresponding CDAI patient-reported component, and the corresponding PRO2 component will not be calculated and will be considered as missing for that visit.

A schema of this approach and some examples are included below for further explanation:

Figure 13-2. Selection of Diary Data for the Calculation at Post-Screening Visits



Table 13-5. Calculation of CDAI Patient-Reported Outcome Components and PRO2 Scores at Post-Screening Visits

| | Dia | Diary Day Looking Backwards from Visit Date (V-Day) | | | | | | | - | Sum of 7 Days<br>(CDAI | Average | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Example | -10 | -9 | -8 | -7 | -6 | -5 | -4 | -3 | -2 | -1 | Days for<br>Calculation | Patient-Reported<br>Component) | of 7 Days<br>(PRO2) |
| Diary<br>Subscore 1 | 1 | 2 | 2 | M | 0 | 1 | 2 | 2 | 1 | X | -2,-3,-4,-5,-6,-<br>8,-9 | 10.0 | 1.4 |
| Diary<br>Subscore 2 | M | M | 1 | M | X | IL | 2 | 2 | 1 | M | -2,-3,-4, -8 | 10.5 | 1.5 |
| Diary<br>Subscore 3 | M | M | 1 | X | IL | M | M | 2 | 1 | M | -2,-3,-8 | Missing | Missing |
| Diary<br>Subscore 4 | 0 | M | 2 | 2 | 1 | 0 | M | 2 | X | IL | -3,-5,-6,-7,-8,-10 | 8.2 | 1.2 |

M = Missing; IL = Ileocolonoscopy day; X = non-evaluable (due to preparation for ileocolonoscopy). Days are named relative to visit date (V-Day 1), where V-Day -1 is the day prior to V-Day 1. Rounding of subscores into one decimal place is for displaying purpose only. When calculating the total CDAI scores, the subscores will not be rounded.

- 4) The CDAI total score for a specific visit is based on a weighted sum (rounded to the nearest integer) of all 8 components. The CDAI total score will be set to 0 in the case the calculation leads to a CDAI total score of < 0. Each component will be selected within the analysis window as defined in
- 5) If subjects have 3 or more of the 8 CDAI components missing, then the subjects will be considered as having insufficient data to determine response status and their total CDAI score will be considered missing. If at least 1 out of the 6 complications under the complication component is missing, then the complication component will be considered missing.

- a) If subjects have 1 or 2 CDAI components missing, then the missing component will be imputed by the LOCF method using the previous valid component score calculated from the most recent analysis visit (ie, use the component score from Week 6 for missing component at Week 10, or use the component score from Week 50 for missing component at Week 58. Scores from other post Induction baseline visits will not be used). If the component score from the most recent analysis visit is also missing, the missing value will be imputed with the corresponding component score at Induction baseline.
  - The PRO2 subscores for a specific visit are based on the evaluation of liquid or very soft stool frequency and abdominal pain subscores individually (rounded to the nearest integer) within the analysis window as defined in Section 3.8.2. If either subscore is missing, no imputation will be done and the subject will be considered as having insufficient data to determine clinical remission status and treated as not meeting clinical remission.
- 6) The total PRO2 score for a specific visit is the sum (rounded to the nearest integer) of liquid or very soft stool subscore (without rounding) × 2 and abdominal pain subscore (without rounding) × 5 within the analysis window as defined in Section 3.8.2. If either subscore is missing, no imputation will be done, and the subject will be considered as having insufficient data to determine clinical remission status and treated as not meeting clinical remission by total PRO2 score.

#### **Source of Information Used for Calculation**

The sources of information used for the calculations of CDAI and PRO2 subscores and total PRO2 score as described above are given in Table 13-6 (the calculated scores from ERT data will not be used for data analysis). Hematocrit results collected from local laboratories and body weight measured at home due to COVID-19 impact will be used in CDAI calculation.

Table 13-6. Sources of Information for Calculating CDAI and PRO2 Scores

| Variable in Calculation | Data Source |
|---|---|
| Ileocolonoscopy Procedure Date | ILEODAT in ILEO dataset from eCRF data for Screening, Week 10 and Week 58; QSTEST = "Date of Colonoscopy" in CDAI dataset from vendor ERT data for the rest of the visits |
| Visit Date | VISITDAT in VISDT dataset from eCRF data |
| Subject Activation Date on<br>Electronic Device | QSORRES in CDAI dataset with QSTEST="Date of Visit" and Visit="Screening" from vendor ERT data |
| Stool Frequency Diary Data | QSSTRESN in DIARY dataset with QSTESTCD="SOFSTOOL" from vendor ERT data |
| Abdominal Pain Diary Data | QSSTRESN in DIARY dataset with QSTESTCD="ABDPAIN" from vendo<br>ERT data |
| Subject Standard Weight | SEX_STD in DM dataset and HEIGHT_STD in VSPERF dataset from eCRF data will be used to determine the standard weight based on Appendix 4. |
| Subject Actual Weight | WEIGHT_STD in VSPERF dataset from eCRF data |
| Hematocrit Value | CNVRESN in COVLAB dataset with LBTEST="Hematocrit" from vendor Covance data or LBORRES in LB_HEM dataset with LBTEST="Hematocrit" from eCRF data if collected in local laboratory due to COVID-19 impact |

Note: eCRF = electronic case report form(s). ERT is the vendor that electronically collects patient and investigator reported outcomes.

#### Appendix 4. Calculation of Standard Body Weight

The following table will be used to determine the standard body weight for each subject. Height from the eCRF will be used and is assumed to be measured without shoes.

| | Wom | nen | |
|---|---|---|---|
| Height in <i>cm</i><br>(in shoes)* | Standard Weight<br>in <i>kg</i> | Height in <i>cm</i> (in shoes)* | Standard Weight<br>in <i>kg</i> |
| 127 | 41.2 | 163 | 60.2 |
| 128 | 41.7 | 164 | 60.7 |
| 129 | 42.3 | 165 | 61.3 |
| 130 | 42.8 | 166 | 61.9 |
| 131 | 43.3 | 167 | 62.4 |
| 132 | 43.8 | 168 | 62.9 |
| 133 | 44.4 | 169 | 63.4 |
| 134 | 44.9 | 170 | 63.9 |
| 135 | 45.4 | 171 | 64.5 |
| 136 | 45.9 | 172 | 65.0 |
| 137 | 46.4 | 173 | 65.5 |
| 138 | 47.0 | 174 | 66.0 |
| 139 | 47.5 | 175 | 66.6 |
| 140 | 48.0 | 176 | 67.2 |
| 141 | 48.6 | 177 | 67.7 |
| 142 | 49.1 | 178 | 68.3 |
| 143 | 49.6 | 179 | 68.8 |
| 144 | 50.2 | 180 | 69.3 |
| 145 | 50.7 | 181 | 69.8 |
| 146 | 51.2 | 182 | 70.3 |
| 147 | 51.8 | 183 | 70.8 |
| 148 | 52.3 | 184 | 71.3 |
| 149 | 52.8 | 185 | 71.8 |
| 150 | 53.1 | 186 | 72.3 |
| 151 | 54.1 | 187 | 72.8 |
| 152 | 54.5 | 188 | 73.3 |
| 153 | 55.0 | 189 | 73.8 |
| 154 | 55.4 | 190 | 74.3 |
| 155 | 55.9 | 191 | 74.9 |
| 156 | 56.4 | 192 | 75.4 |
| 157 | 57.0 | 193 | 76.0 |
| 158 | 57.5 | 194 | 76.5 |
| 159 | 58.1 | 195 | 77.0 |
| 160 | 58.6 | 196 | 77.6 |
| 161 | 59.1 | 197 | 78.1 |

Version 2.0

| 162 | 59.6 | 198 | 78.6 |
|-----|------|-----|------|

<sup>\*</sup> add 2.0 cm if shoeless. Please round height to a whole number and select the appropriate standard weight (eg, height 157.4 cm will be rounded to 157 cm; 157.5 cm will be rounded to 158 cm.)

| Men | | | |
|---|---|---|---|
| Height in <i>cm</i><br>(in shoes)* | Standard Weight<br>in <i>kg</i> | Height in <i>cm</i> (in shoes)* | Standard Weight<br>in <i>kg</i> |
| 142 | 54.4 | 179 | 71.9 |
| 143 | 54.9 | 180 | 72.4 |
| 144 | 55.4 | 181 | 73.0 |
| 145 | 55.8 | 182 | 73.6 |
| 146 | 56.3 | 183 | 74.3 |
| 147 | 56.8 | 184 | 74.8 |
| 148 | 57.2 | 185 | 75.5 |
| 149 | 57.7 | 186 | 76.2 |
| 150 | 58.2 | 187 | 76.9 |
| 151 | 58.6 | 188 | 77.6 |
| 152 | 59.1 | 189 | 78.2 |
| 153 | 59.6 | 190 | 78.8 |
| 154 | 60.0 | 191 | 79.6 |
| 155 | 60.5 | 192 | 80.4 |
| 156 | 61.0 | 193 | 81.2 |
| 157 | 61.4 | 194 | 82.1 |
| 158 | 61.9 | 195 | 82.9 |
| 159 | 62.2 | 196 | 83.8 |
| 160 | 62.6 | 197 | 84.7 |
| 161 | 62.9 | 198 | 85.4 |
| 162 | 63.3 | 199 | 86.1 |
| 163 | 63.7 | 200 | 86.7 |
| 164 | 64.1 | 201 | 87.4 |
| 165 | 64.6 | 202 | 88.0 |
| 166 | 65.0 | 203 | 88.8 |
| 167 | 65.5 | 204 | 89.4 |
| 168 | 66.0 | 205 | 90.1 |
| 169 | 66.6 | 206 | 90.7 |
| 170 | 67.1 | 207 | 91.4 |
| 171 | 67.6 | 208 | 92.1 |
| 172 | 68.1 | 209 | 92.7 |
| 173 | 68.7 | 210 | 93.4 |
| 174 | 69.2 | 211 | 94.1 |
| 175 | 69.7 | 212 | 94.8 |

Version 2.0

| 176 | 70.3 | | 213 | 95.5 |
|-----|------|---|-----|------|
| 177 | 70.8 | • | 214 | 96.1 |
| 178 | 71.3 | | | |

<sup>\*</sup> add 2.0 cm if shoeless. Please round height to a whole number and select the appropriate standard weight (eg, height 157.4 cm will be rounded to 157 cm; 157.5 cm will be rounded to 158 cm.)

#### Appendix 5. Simple Endoscopic Score for Crohn's Disease (SES-CD)

| | ore | | | |
|---|---|---|---|---|
| Variables | 0 | 1 | 2 | 3 |
| Size of ulcers (cm) | None | Aphthous ulcers (diameter 0.1-0.5) | Large ulcers (diameter 0.5-2) | Very large ulcers (diameter > 2) |
| Ulcerated Surface (%) | None | < 10 | 10-30 | > 30 |
| Affected surface (%) | Unaffected segment | < 50 | 50-75 | > 75 |
| Presence of narrowings | None | Single, can be passed | Multiple, can be passed | Cannot be passed |

Total SES-CD: sum of the values of the 4 variables for the 5 bowel segments. Values are given to each variable and for every examined bowel segment (eg, rectum, left colon, transverse colon, right colon, and ileum) {Daperno 2004}

#### **Appendix 6.** Study Treatment Failure Rules

Study treatment failure rules apply to treatment failure that occurs during the course of the study. Study treatment failure rules will be applied to all efficacy endpoints, unless otherwise specified. All efficacy data will be censored (set to missing) after treatment failure criteria are met, regardless of the observed data. Subjects who do not have sufficient measurements after censoring to determine the dichotomized endpoint(s) will be considered non-responder for corresponding endpoint(s). Study treatment failure rules override other data handling rules.

Subjects who have any of the following events will be considered a study treatment failure after the earliest event through the end of the Induction Study (if the event occurred during Induction) or through the end of the Maintenance Study (if the event occurred during Maintenance), regardless of the actual efficacy data collected. Induction baseline will be referenced when calculating the potentially effective use for Induction Studies, and Maintenance baseline will be referenced when calculating the potentially effective use for Maintenance Study.

#### 1) Potentially effective corticosteroid use

Potentially effective corticosteroids, for the purpose of this SAP, are corticosteroids that may impact the disease under study. **Potentially effective corticosteroids** include the following corticosteroids when administered for the indication of CD:

#### a) Commencement of:

Any steroid administered intramuscularly (IM), intravenously (IV), orally (PO), or rectally (PR) at any dose for 7 or more continuous days

- This rule applies regardless if a change in drug, dose, or route (from IM to IV to PO or PR or vice versa) occurs within the seven continuous days; and it includes oral steroids with intended local actions (eg, budesonide)
- b) Escalation of concomitant steroid dose above the baseline dose for 7 or more continuous days. The baseline steroid dose is defined as the dose at Day 1 of induction if the escalation occurs in the Induction Study, or Day 1 of maintenance (maintenance baseline) if the escalation occurs in the Maintenance Study. Prednisone equivalent dose will be used to determine escalation of concomitant systemic steroid dose even if there is a change in drug or route. For steroids with predominant local effect (eg, budesonide or any rectally administered steroid), the dose escalation rule will apply to scenarios where the post-baseline dose is above the baseline dose via the same drug and the same route for 7 or more continuous days.

Potentially effective steroid use only includes use of steroids administered via routes that are IM, PO, IV, or PR. The below steroids will **not** be considered potentially effective steroids regardless of indication for use:

- A) ocular steroids (ie, eye drops)
- B) topical steroids (eg, cutaneously applied solely to the skin, or topically applied to the nasal mucosa)
- C) inhaled steroids (eg, inhalational fluticasone for asthma)
- D) intra-articular steroids (steroids administered directly into a joint)
- E) neuraxial steroids (steroids administered into the epidural or spinal space)

#### 2) Potentially effective immunomodulator use

Commencement of a different class of oral, IM, SC, or IV immunomodulator drugs (where the subject was not previously taking concomitant immunomodulators of the same class on Day 1 of induction or maintenance), including but not limited to 6-MP, azathioprine, MTX, 6-thioguanine, and prohibited immunomodulators including but not limited to cyclosporine, leflunomide, tacrolimus, thalidomide regardless of dose, for 7 continuous days. The use of an immunomodulator will be considered potentially effective when it is administered for the indication of CD.

#### 3) Potentially effective biologic agent use

Commencement of a biologic agent including but not limited to TNF- $\alpha$  antagonists, IL-12/23 antagonists, and vedolizumab (or similar agents), regardless of indication for use and duration.

#### Appendix 7. Determining Missing and Virtual Visits due to COVID-19

This appendix describes the clinical trial site collection of COVID-19 data pertaining to missed/virtual visits and the data processing algorithm used to determine which visits were missing and which visits were virtual.

#### Data collection

A COVID-19 supplement to the eCRF Completion Guidelines was provided by data management to instruct clinical trial sites with respect to data entry expectations pertaining to scenarios related to the COVID-19 pandemic. If a visit was missed, sites should enter "Visit missed due to COVID-19." If an in-person visit was conducted virtually, sites should enter "Virtual visit due to COVID-19."

#### Determination of Missed and Virtual visits

Natural Language Processing (NLP) was used to search the CRF comment fields to identify instances of "COVID-19" (or synonyms, see Table 13-7) and "Virtual" (or synonyms, see Table 13-7). The search terms are maintained in a global lookup table and can be modified to tune the NLP model. For any comments with COVID-19 search terms, assign "Missed visit" or "Virtual visit" as follows:

- i) If COVID-19 terms are identified through NLP and the visit date is missing, then result is "Missed Visit."
- ii) If COVID-19 and Virtual terms are identified through NLP for a visit, then result is "Virtual Visit". When there are multiple records for the same subject and the same visit, NLP will be based on multiple records to ensure that only 1 unique visit type (either Missing Visit or Virtual Visit) is assigned for all the records belong to the same visit for a subject.
- iii) Otherwise the visit type is missing.

Table 13-7. Examples of Search Terms for "COVID-19" and "Virtual" Used to Identify Missed and Virtual Visits

| Search terms for "COVID-19" | Search terms for "Virtual" |
|-----------------------------|----------------------------|
| COVID19 | VIRTUAL |
| CORONA | TELEMED |
| CORONAVIRUS | TELEHEALTH |
| PANDEMIC | TELEPHONE |
| OUTBREAK | REMOTE |
| CRISIS | TELEMEDICINE |
| LOCKDOWN | TELECONSULTATION |

| <b>T</b> 7 | | $^{\circ}$ |
|------------|---------|------------|
| 1/ | ersion | , , |
| v | CISIOII | Z.() |

| QUARANTINE | TELEPHONICALLY |
|------------|----------------|
| SHELTER | PHONE |
| | HOME VISIT |
| | ZOOM |
| | SKYPE |

#### Appendix 8. SAS Programming for Tipping Point Analysis for Binary Endpoint

The following **%tp\_binary** macro generates multiple imputed data and a set of the shift parameters that adjust the imputed values will be examined.

```
/*--- Delta-Adjusting Method for Tipping Point Analysis for Binary Endpoint
/*--- Generate imputed data set for specified shift parameters
/*--- data= input data set
/*--- smin= min shift parameter for active drug
/*--- smax= max shift parameter for active drug
/*--- sinc= increment of the shift parameter for active drug
/*--- pmin= min shift parameter for placebo drug
/*--- pmax= max shift parameter for placebo drug
/*--- pinc= increment of the shift parameter for placebo drug
/*--- trt= treatment group indicator
/*--- out= output imputed data set
                                                                                 ---*/
/*______*/
%macro tp binary( data=, smin=, smax=, sinc=, pmin=, pmax=, pinc=, trt=, out=);
       data &out;
       set null;
       run:
/*----*/
       %let nease pbo = %sysevalf( (&pmax-&pmin)/&pinc, ceil );
       %do pc=0 %to &ncase pbo;
       %let pj= %sysevalf( &pmin + &pc * &pinc);
               /*----*/
               %let ncase= %sysevalf( (&smax-&smin)/&sinc, ceil );
               /*----*/
               %do jc=0 %to &ncase;
               %let sj= %sysevalf( &smin + &jc * &sinc);
                       proc mi data=&data seed=14823 nimpute=20 out=outmi;
                              var trt01pn strat1V strat2V strat3V RESP;
                              class trt01pn strat1V strat2V strat3V RESP;
                              monotone logistic (RESP / link=glogit);
                              mnar adjust(RESP (event='1') / adjustobs=(trt01pn="&trt") shift= &sj)
                                      adjust(RESP (event='1') / adjustobs=(trt01pn='3') shift= &pj);
                              run;
               data outmi;
```

```
set outmi;
Shift_Trt= &sj;
Shift_Pbo= &pj;
run;

data &out;
set &out outmi;
run;

%end;
%mend tp_binary;
```

#### Appendix 9. MST lists for AEs of Interest

Herpes Zoster - Galapagos Search Term List MedDRA Version 25.0


## Nonmelanoma Skin Cancers - Galapagos Search Term List MedDRA Version 25.0


### Gastrointestinal Perforations - Galapagos Search Term List MedDRA Version 25.0


#### Unstable Angina - Galapagos Search Term List MedDRA Version 25.0


### Transient Ischemic Attack - Galapagos Search Term List MedDRA Version 25.0


## Transient Ischemic Attack - Galapagos Search Term List MedDRA Version 25.0


Stroke - Galapagos Search Term List MedDRA Version 25.0


Stroke - Galapagos Search Term List MedDRA Version 25.0


### Cardiac Failure - Galapagos Search Term List MedDRA Version 25.0


### Cardiac Failure - Galapagos Search Term List MedDRA Version 25.0


# Percutaneous Coronary Intervention - Galapagos Search Term List MedDRA Version 25.0

# Percutaneous Coronary Intervention - Galapagos Search Term List MedDRA Version 25.0


GLPG0634-CL-MACE, 20DEC22:15:49

# Percutaneous Coronary Intervention - Galapagos Search Term List MedDRA Version 25.0


GLPG0634-CL-MACE, 20DEC22:15:49

Specific AE directly associated with the pathogen causing COVID-19 - Galapagos Search Term List MedDRA Version 25.0  $\,$ 


GLPG0634-CL-MACE, 20DEC22:15:49

### Appendix 10. PKAP



# PHARMACOKINETIC ANALYSIS PLAN

Combined Phase 3, Double-blind, Randomized, Placebo-Controlled Studies Evaluating the Efficacy and Safety of Filgotinib in the Induction and Maintenance of Remission in Subjects with Moderately to Severely Active Crohn's Disease

Galapagos NV Generaal De Wittelaan L11 A3 2800 Mechelen Belgium

Protocol Identification: GS-US-419-3895

Pharmacokinetic Analysis Plan

Version: 1.0

Date: December 20, 2022

#### PHARMACOKINETIC ANALYSIS PLAN

#### **REPORT TITLE:**

Combined Phase 3, Double-blind, Randomized, Placebo-Controlled Studies Evaluating the Efficacy and Safety of Filgotinib in the Induction and Maintenance of Remission in Subjects with Moderately to Severely Active Crohn's Disease

QPS PROJECT NO.

2260-2202CRS

CLIENT PROTOCOL NO.

GS-US-419-3895

#### **CONTRIBUTING SCIENTISTS:**

PPD

Sr. Principal Clinical Pharmacokineticist II

Global Data Services

QPS, LLC

#### **TESTING FACILITY:**

QPS, LLC 3 Innovation Way, Suite 240 Newark, DE 19711

#### **SPONSOR:**

Galapagos NV

Generaal De Wittelaan L11 A3

2800 Mechelen, Belgium

#### **SPONSOR REPRESENTATIVES:**



Sr Director Clinical Pharmacology Galapagos NV

# Signature Page



Page

# **TABLE OF CONTENTS**

| 1. | | ATIONS AND DEFINITIONS OF TERMS | |
|---|---|---|---|
| 2. | INTRODUCTION | | 22 |
| 3. | STUDY BACKGROU | OUND | 23 |
| 4. | PKAP OBJECTIVE | | 24 |
| 5. | SUMMARY OF STU | UDY DESIGN | 25 |
| 6. | PHARMACOKINET | TIC ANALYSIS PLAN | 26 |
| | <ul><li>6.2. Pharmacokine</li><li>6.3. Data Handling</li></ul> | y Analysis Setnetic Parameters Estimationng Proceduresvaluations of PK Parameters | 26<br>27 |
| 7. | REPORT | | 30 |
| 8. | TABLES AND LISTI | ΓINGS | 35 |
| | | scriptive Statistics of Plasma Concentrations of Filgotinib ar | |
| | Table 14.4.1.1.Descrip Oral Adminis | riptive Statistics of Plasma Concentrations of Filgotinib Follostration of 200 mg Filgotinib at One Visit Between Week 2 h Moderately to Severely Active Crohn's Disease | owing Once Daily<br>and Week 10 in |
| | Table 14.4.1.2.Descrip | riptive Statistics of Plasma Concentrations of Filgotinib Follosistration of 100 mg Filgotinib at One Visit Between Week 2 h Moderately to Severely Active Crohn's Disease | owing Once Daily<br>and Week 10 in |
| | Table 14.4.1.3 Do | Descriptive Statistics of Plasma Concentrations of GS-82984 Administration of 200 mg Filgotinib at One Visit Between Wats with Moderately to Severely Active Crohn's Disease | 5 Following Once<br>Veek 2 and Week |
| | Table 14.4.1.4 Do | Descriptive Statistics of Plasma Concentrations of GS-82984 Administration of 100 mg Filgotinib at One Visit Between Wats with Moderately to Severely Active Crohn's Disease | 5 Following Once Veek 2 and Week |
| | Table 14.4.1.5.Descrip<br>Oral Adminis | riptive Statistics of Plasma Concentrations of Filgotinib Folkistration of 200 or 100 mg Filgotinib in Subjects with Modern's Disease - Cohort A | owing Once Daily rately to Severely |
| | Table 14.4.1.6.Descrip<br>Oral Adminis | riptive Statistics of Plasma Concentrations of Filgotinib Follostration of 200 or 100 mg Filgotinib in Subjects with Mode n's Disease - Cohort B | owing Once Daily rately to Severely |
| | Oral Adminis | riptive Statistics of Plasma Concentrations of Filgotinib Folloistration of 200 or 100 mg Filgotinib in Subjects with Mode n's Disease - Maintenance Study | rately to Severely |
| | Daily Oral Ac<br>Severely Acti | Descriptive Statistics of Plasma Concentrations of GS-82984 Administration of 200 or 100 mg Filgotinib in Subjects with tive Crohn's Disease - Cohort A | Moderately to39 |
| | Table 14.4.1.9 Do<br>Daily Oral Acti<br>Severely Acti | Descriptive Statistics of Plasma Concentrations of GS-82984<br>Administration of 200 or 100 mg Filgotinib in Subjects with<br>tive Crohn's Disease - Cohort B | 5 Following Once<br>Moderately to39 |
| | Daily Oral Ad | Descriptive Statistics of Plasma Concentrations of GS-82984 Administration of 200 or 100 mg Filgotinib in Subjects with tive Crohn's Disease - Maintenance Study | Moderately to |

| Table 14.4.2 Descriptive Statistics of Plasma Filgotinib and Metabolite GS-829845 |
|---|
| Pharmacokinetic Parameters |
| Table 14.4.2.1 Descriptive Statistics of Plasma Pharmacokinetic Parameters of Filgotinib |
| Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between |
| Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease .40 |
| Table 14.4.2.2 Descriptive Statistics of Plasma Pharmacokinetic Parameters of Filgotinib |
| Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between |
| Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease.41 |
| Table 14.4.2.3 Descriptive Statistics of Plasma Pharmacokinetic Parameters of GS-829845 |
| Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between |
| Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease.41 |
| Table 14.4.2.4 Descriptive Statistics of Plasma Pharmacokinetic Parameters of GS-829845 |
| Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between |
| Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease .42 |
| Listing 16.4.1 |
| Metabolite GS-829845 |
| Listing 16.4.1.1 Individual Plasma Concentrations of Filgotinib Following Once Daily Oral |
| Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in |
| Subjects with Moderately to Severely Active Crohn's Disease |
| Listing 16.4.1.2 Individual Plasma Concentrations of Filgotinib Following Once Daily Oral |
| Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in |
| Subjects with Moderately to Severely Active Crohn's Disease |
| Listing 16.4.1.3 Individual Plasma Concentrations of GS-829845 Following Once Daily Oral |
| Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in |
| Subjects with Moderately to Severely Active Crohn's Disease |
| Listing 16.4.1.4 Individual Plasma Concentrations of GS-829845 Following Once Daily Oral |
| Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in |
| Subjects with Moderately to Severely Active Crohn's Disease |
| Listing 16.4.2. Individual Plasma Filgotinib and Metabolite GS-829845 |
| Pharmacokinetic Parameters 43 |
| Listing 16.4.2.1 Individual Plasma Pharmacokinetic Parameters of Filgotinib Following Once |
| Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease |
| Listing 16.4.2.2 Individual Plasma Pharmacokinetic Parameters of Filgotinib Following Once |
| Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease |
| Listing 16.4.2.3Individual Plasma Pharmacokinetic Parameters of GS-829845 Following Once |
| Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease44 |
| Listing 16.4.2.4 Individual Plasma Pharmacokinetic Parameters of GS-829845 Following Once |
| Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease44 |
| Figure 16.4.3 Individual Subject Plasma |
| Concentration-Time Graphs45 |
| Figure 16.4.3.1 Individual Plasma Filgotinib Concentration – Time Profiles Following Once |
| Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease |
| Figure 16.4.3.2 Individual Plasma Filgotinib Concentration – Time Profiles Following Once |
| Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease |
| Figure 16.4.3.3Individual Plasma Filgotinib Concentration – Time Profiles Following Once |
| Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours46 |

| Figure 16.4.3.4 Individual Plasma Filgotinib Concentration – Time Profiles Following On | ice |
|---|---|
| Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Wee | k |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours | 47 |
| Figure 16.4.3.5 Individual Plasma GS-829845 Concentration - Time Profiles Following On | ice |
| Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Wee | k |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease | |
| Figure 16.4.3.6 Individual Plasma GS-829845 Concentration – Time Profiles Following On | ice |
| Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Wee | k |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease | 47 |
| Figure 16.4.3.7 Individual Plasma GS-829845 Concentration – Time Profiles Following On | ice |
| Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Wee | k |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours | |
| Figure 16.4.3.8 Individual Plasma GS-829845 Concentration – Time Profiles Following On | ice |
| Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Wee | k |
| 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours | 47 |

# LIST OF TABLES AND FIGURES

| Table 14.2.1. | Subjects Not Included in the Pharmacokinetic Analysis (if Applicable)30 |
|---|---|
| Figure 14.2.1. | Mean (± SD) Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease |
| Figure 14.2.2. | Mean (± SD) Plasma GS-829845 Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease |
| Figure 14.2.3. | Mean (± SD) Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours |
| Figure 14.2.4. | Mean (± SD) Plasma GS-829845 Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours |
| Figure 14.2.5. | Median (Q1, Q3) Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease |
| Figure 14.2.6. | Median (Q1, Q3) Plasma GS-829845 Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease |
| Figure 14.2.7. | Median (Q1, Q3) Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours |
| Figure 14.2.8. | |

# 1. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|---|---|
| AM | Arithmetic mean |
| %AUC <sub>extrap</sub> | Percentage of extrapolated AUC (%AUC <sub>t-∞</sub> ), (1-[AUC <sub>0-t</sub> /AUC <sub>0-inf</sub> ])*100 |
| $\mathrm{AUC}_{0	ext{-tau}}$ | Area under the concentration-time curve within dosing interval, calculated by linear up/log down trapezoidal method. |
| BLQ | Below the lower limit of quantification |
| $C_{\text{max}}$ | Maximum observed plasma concentration |
| CD | Crohn's disease |
| CL <sub>ss</sub> /F | Apparent total body clearance at steady state |
| $C_{\text{tau}}$ | The concentration in plasma at the end of a dosing interval |
| CV% | Percentage coefficient of variation |
| GM | Geometric mean |
| Н | Hour |
| IBD | Inflammatory bowel disease |
| (IL)-6 | Interleukin |
| JAKs | Janus kinases |
| LLOQ | Lower limit of quantification |
| Max | Maximum |
| Min | Minimum |
| MRcmax | Metabolic ratio of C <sub>max</sub> |
| MRctau | Metabolic ratio of C <sub>tau</sub> |
| MRauctau | Metabolic ratio of AUC <sub>0-tau</sub> |
| PD | Pharmacodynamics |

| Abbreviation | Definition |
|------------------|---------------------------------------------------|
| PK | Pharmacokinetic(s) |
| Q1 | 1 <sup>st</sup> quartile |
| Q3 | 3 <sup>rd</sup> quartile |
| RA | Rheumatoid arthritis |
| SD | Standard deviation |
| $T_{\text{max}}$ | Time of the maximum observed plasma concentration |
| TYKs | Tyrosine kinases |
| UC | Ulcerative colitis |

#### 2. INTRODUCTION

This Pharmacokinetic Analysis Plan (PKAP) for GS-US-419-3895 study has been developed according to the study design described in the study protocol Amendment 9 dated on 02 December 2021 with the purpose of establishing a framework for pharmacokinetic (PK) analysis in which answers to the protocol objectives may be obtained in a rigorous fashion, without bias or analytical deficiency.

The purpose of this plan is two-fold:

- To determine the types of analyses and presentations of data that will form the basis for conclusions to be reached;
- To define in detail how the data will be handled and analyzed, adhering to commonly accepted standards and practices of PK and biostatistical analysis in the pharmaceutical industry and QPS SOPs.

The PK parameters and statistical results outlined herein will be reported in a PK Section that will be included to the Clinical Study Report (CSR).

.

#### 3. STUDY BACKGROUND

Crohn's disease (CD) is a relapsing and remitting form of inflammatory bowel disease (IBD) that causes gastrointestinal signs and symptoms of diarrhea, abdominal pain, weight loss, and the passage of blood or mucous per rectum. The inflammation of CD can involve the mucosal surface of the gastrointestinal tract and penetrate through the full thickness of the gastrointestinal wall, including the serosal surface. Crohn's disease is characterized by phenotype and location of involved bowel. The phenotypes include inflammatory, stricturing, and penetrating subtypes. Stricture formation can result in intestinal obstruction requiring surgical management. Over time, patients with repeated surgeries are at risk for developing short bowel syndrome and/or intestinal failure.

Janus kinases (JAKs) are intracellular cytoplasmic tyrosine kinases (TYKs) that transduce cytokine signaling from membrane receptors through signal transducer and activator of transcription (STAT) to the nucleus of cells. JAK inhibitors block the signaling of various cytokines, growth factors, and hormones, including the proinflammatory cytokine interleukin (IL)-6. Four different types of JAKs are known, JAK1, JAK2, JAK3, and TYK2 which interact with different sets of membrane receptors. Inhibition of JAKs is a promising therapeutic option for a range of inflammatory conditions including rheumatoid arthritis (RA) and CD.

Filgotinib (GS-6034, formerly known as GLPG0634) is a potent and selective inhibitor of JAK1. Filgotinib is approved in the European Union (EU), Japan, and Great Britain for treatment of moderate to severe active RA in adult patients. It is also approved for the treatment of moderately to severely active ulcerative colitis (UC) in adults in the EU, and is currently under regulatory review for the treatment of UC in Japan and Great Britain. The compound has shown good preliminary efficacy in CD patients in Phase 2 studies.

In humans, filgotinib is metabolized to form one major active metabolite, GS-829845. Though the potency of this metabolite is lower than the parent molecule, the overall exposure and peak plasma concentration in humans is higher than seen in all tested animal species. As a consequence, dedicated pharmacology and toxicology studies have been performed with GS-829845. Results from pharmacodynamics (PD) testing in healthy volunteers suggest that the clinical activity of filgotinib could result from the combination of the parent molecule and the metabolite.

For further information on filgotinib, refer to the current Investigator's Brochure (IB).

# 4. **PKAP OBJECTIVE**

• To assess the PK characteristics of filgotinib and its metabolite GS-829845.

#### 5. SUMMARY OF STUDY DESIGN

These are combined Phase 3 double-blind, randomized, placebo-controlled studies to evaluate the efficacy and safety of filgotinib in the induction and maintenance of clinical remission, as well as, endoscopic response in subjects with moderately to severely active CD.

Subjects who are biologic-naïve or biologic-experienced will be enrolled in Cohort A and subjects who are biologic-experienced will be enrolled in Cohort B, respectively. Treatment assignments will be randomized within each Cohort.

#### **Treatment Regimen (Cohorts A and B Induction Studies)**

Subjects who meet protocol eligibility criteria will be assigned to the respective Cohort and subsequently randomized in a blinded fashion in a 1:1:1 ratio to 1 of 3 treatments as follows:

**Treatment 1:** filgotinib 200 mg oral tablet and placebo-to-match (PTM) filgotinib 100 mg oral tablet, once daily

**Treatment 2**: filgotinib 100 mg oral tablet and PTM filgotinib 200 mg oral tablet, once daily **Treatment 3**: PTM filgotinib 200 mg oral tablet and PTM filgotinib 100 mg oral tablet, once daily

Note: US and Korea males who have not failed at least two biologic therapies (any TNF $\alpha$  antagonist and vedolizumab) will be randomized in a 1:1 ratio to either filgotinib 100 mg or matching placebo.

The sparse PK samples at Week 4 are collected pre-dose, and post-dose (at least 30 minutes and up to 3 hours after study drug dosing). For this visit, it is preferred that study drug dosing is done in clinic. The PK sample at Weeks 26 can be collected at any time without regard to dosing. The PK sample at Weeks 10 and 58 are collected at pre-dose (within 2 hours prior to dosing).

The optional PK substudy will be performed in a subset of subjects (approximately 16 subjects on 200 mg treatment and 16 subjects on 100 mg treatment in the substudy) who provide a separate informed consent. In the PK substudy, the daily dose of study drug should be administered under supervision in the clinic (at one visit between Week 2 and Week 10, inclusive), and the PK substudy will have additional plasma PK samples at any single visit from Week 2 to Week 10, collected pre-dose, and at 0.5, 1, 2, 3, 4 and 6 hours after supervised dosing in the clinic. If a sub-study PK sample is scheduled to be collected at the same time as a sparse PK sample, only one sample should be collected.

For all visits with PK sampling, the time of dose taken prior to and on the day of visit will be noted in the eCRF. Plasma concentrations of filgotinib and its metabolite (GS-829845) will be analyzed.

#### 6. PHARMACOKINETIC ANALYSIS PLAN

#### 6.1. PK Substudy Analysis Set

The primary analysis set for intensive PK analyses will be the PK substudy analysis set for each Induction Study (Cohorts A and B), which includes all subjects in the Safety Analysis Set from the corresponding Induction Study who have enrolled into the PK substudy, and have dense concentration data to provide interpretable results for the specific parameters of interest for the analyte under evaluation.

The primary analysis set for general PK analyses will be defined separately for each individual study (Cohort A Induction Study, Cohort B Induction Study, and Maintenance Study). For each study, the PK analysis set includes all subjects in the corresponding Safety Analysis Set who have at least 1 non-missing plasma concentration data for filgotinib and/or its metabolite GS-829845.

#### 6.2. Pharmacokinetic Parameters Estimation

The plasma PK parameters for filgotinib and its metabolite (GS-829845) will be derived by non-compartmental analysis of the plasma concentration-time profiles based on actual blood sampling times [h] (relative to the corresponding administration time) rounded to two decimal digits and negative pre-dose times set to zero. The plasma PK parameters will be computed using Phoenix WinNonlin 6.3 or higher. The nominal times will be used to present in the individual concentration listings or tables and the mean concentration-time figures.

The following plasma PK parameters of filgotinib and its metabolite (GS-829845) will be calculated as data allows. The definition for each PK variable is listed in the following tables:

| C <sub>max</sub> | The maximum observed plasma concentration |
|---|---|
| T <sub>max</sub> | The time to reach $C_{max}$ |
| C <sub>tau</sub> | The concentration in plasma at the end of a dosing interval |
| AUC <sub>0-tau</sub> | Area under the concentration-time curve within dosing interval, |
| | calculated by linear up/log down trapezoidal method. A 24 hour data |
| | point will be based on imputation of the predose value of filgotinib and |
| | its metabolite (GS-829845). |
| CL <sub>ss</sub> /F | Apparent total body clearance at steady state, calculated as |
| | Dose/AUC <sub>0-tau</sub> , on steady state, for parent compound only |
| MRcmax | Metabolic ratio of GS-829845 C <sub>max</sub> / filgotinib C <sub>max</sub> * (425.51/357.43) |
| MRctau | Metabolic ratio of GS-829845 C <sub>tau</sub> / filgotinib C <sub>tau</sub> * (425.51/357.43) |
| MRauctau | Metabolic ratio of GS-829845 AUC <sub>0-tau</sub> / filgotinib AUC <sub>0-tau</sub> * |
| | (425.51/357.43) |

The substudy PK analysis population will be used for the analyses. Individual subject listings will be provided. For substudy PK analysis, mean and individual plasma concentration-time

profiles for filgotinib and its metabolite (GS-829845) will be presented graphically for each treatment.

The measured individual plasma concentrations of filgotinib and its metabolite (GS-829845) will be used to directly obtain  $C_{max}$  and  $T_{max}$  for substudy PK analysis.

The concentration in plasma at the end of a dosing interval (C<sub>tau</sub>), where tau is 24 h, was also determined. To estimate AUC<sub>0-tau</sub>, the concentration observed in the predose sample (collected at steady-state) will be assumed as the same 24h post-dose.

For general PK analysis, descriptive statistics for plasma concentrations of filgotinib and its metabolite GS-829845 will be listed and summarized per timepoint and per treatment for Cohort A, Cohort B, and maintenance study.

#### 6.3. Data Handling Procedures

Only subjects included in the PK substudy analysis set and only samples obtained in this substudy will be included in the summary statistics for PK parameters. All analyses will be performed on data available at the time point considered. In summary tables, the number of subjects with missing data will be presented unless otherwise specified. In the calculation of percentages, subjects with missing data will not be considered in numerator or denominator unless otherwise specified.

#### **Missing Concentrations:**

Samples will be treated as missing for PK data analysis, if:

- Blood samples are collected but no bioanalytical data are reported;
- Missed PK sample collections;
- Samples are collected but the sampling time and/or dosing time are not recorded;
- Samples whose identities are uncertain due to possible handing or labelling errors conducted in the clinical site or bioanalytical labs;
- Sample is diluted and below the quantifiable limits.

#### **Protocol Deviations and/or Violations**

The data for subjects with significant protocol deviations and/or violations will be cautiously evaluated. If the deviation or violation has a significant impact on the filgotinib and its metabolite (GS-829845) PK profile, the data for those subjects should be excluded from the study's statistical evaluation by the pharmacokineticist and the reason for excluding individual data points will be recorded. Filgotinib and its metabolite (GS-829845) concentration data and PK parameters derived for those subjects will not be determined and reported.

#### Below the Lower Limit of Quantification Limit (BLQ)

PK concentration values and PK parameter values below the lower limit of quantitation (BLQ) will be presented as "BLQ" in the data listings. BLQ values will be treated as 1/2 of the lower limit of quantitation (LLOQ) for calculation of geometric mean and CV%, and will be treated as 0 for all other summary statistics. Unexpected BLQ samples or samples whose identity is

uncertain due to possible handling or labeling errors can be treated as missing at the judgment of the pharmacokineticist and noted accordingly.

#### Data exclusion due to vomiting:

In regard to the data from subjects who experience emesis during the PK sampling period (i.e. in the period "predose until the last sample (6 hrs post dose), if vomiting occurs at or before 2 times median  $T_{max}$  under the same treatment, the time course of the study for filgotinib and its metabolite GS-829845 will be excluded from pharmacokinetic statistical analysis.

#### Data Format (significant figures and decimal points)

PK concentrations and PK parameters will be reported to 3 significant figures for individual concentrations and parameters and summary statistics, with the exception of  $T_{max}$  (2 decimal places), coefficient of variation (CV%, 1 decimal place), and the number of subjects (N, 0 decimal place).

#### 6.4. Statistical Evaluations of PK Parameters

For each individual study (Cohort A Induction Study, Cohort B Induction Study and Maintenance Study), plasma concentrations of filgotinib and its metabolite GS-829845 will be listed and summarized by treatment using descriptive statistics (eg, sample size, arithmetic mean, geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum).

For the subjects at the substudy, individual concentrations and PK parameters of filgotinib and its metabolite GS-829845 will be listed. Mean concentrations and PK parameters of filgotinib and its metabolite GS-829845 will be summarized descriptively. Individual and mean concentration-time profiles will be presented on semi-logarithmic and linear formats as mean  $\pm$  SD and median (Q1, Q3) by treatment.

For descriptive statistics of pharmacokinetic parameters and concentration data, sample size, arithmetic mean, geometric mean, % coefficient of variation, standard deviation, median, 1<sup>st</sup> quartile [Q1] (for concentration data only), 3<sup>rd</sup> quartile [Q3] (for concentration data only), minimum, and maximum, will be given.

Plasma concentrations for the subjects at each individual study and substudy will be listed by subject and nominal sampling time and summarized by nominal sampling time and treatment using descriptive statistics. Similarly, calculated plasma PK parameters for substudy will be listed by subject and summarized by treatment using descriptive statistics.

# 7. REPORT

The following tables and figures will be generated.

Table 14.2.8. Subjects Not Included in the Pharmacokinetic Analysis (if Applicable)

| Subject | Treatment | Dose level | Comments |
|---------|-----------|------------|----------|

Figure 14.2.3. Mean (± SD) Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

**Linear Scale (Mock Figure)** 



## Semi-logarithmic Scale (Mock Figure)



Figure 14.2.4. Mean (± SD) Plasma GS-829845 Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

Figure 14.2.5. Mean (± SD) Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours

Linear Scale (Mock Figure)



Semi-logarithmic Scale (Mock Figure)



Figure 14.2.6. Mean (± SD) Plasma GS-829845 Concentration – Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours

- Figure 14.2.7. Median (Q1, Q3) Plasma Filgotinib Concentration Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease
- Figure 14.2.8. Median (Q1, Q3) Plasma GS-829845 Concentration Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease
- Figure 14.2.9. Median (Q1, Q3) Plasma Filgotinib Concentration Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease 0 to 24 hours
- Figure 14.2.10. Median (Q1, Q3) Plasma GS-829845 Concentration Time Profiles Following Once Daily Oral Administration of 100 or 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease 0 to 24 hours

#### 8. TABLES AND LISTINGS

Descriptive statistics plasma filgotinib and its metabolite GS-829845 concentrations will be provided in Tables 14.4.1. Descriptive statistics plasma pharmacokinetic parameters of filgotinib and its metabolite GS-829845 will be included in Tables 14.4.2. The individual subject filgotinib and its metabolite GS-829845 plasma concentration will be included in in Listing 16.4.1. The individual subject filgotinib and its metabolite GS-829845 plasma pharmacokinetic parameters will be included in in Listing 16.4.2. The individual subject filgotinib and its metabolite GS-829845 plasma concentration time plots will be included in in Figures 16.4.3.

#### Table 14.4.1. Descriptive Statistics of Plasma Concentrations of Filgotinib and Metabolite GS-829845

# Table 14.4.1.1. Descriptive Statistics of Plasma Concentrations of Filgotinib Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

| | | Plasma Concentration (ng/mL) over Nominal Time (h) | | | | | |
|---|---|---|---|---|---|---|---|
| Subject | Pre-dose | 0.5 | 1 | 2 | 3 | 4 | 6 |
| N | | | | | | | |
| AM | | | | | | | |
| SD | | | | | | | |
| Min | | | | | | | |
| Q1 | | | | | | | |
| Median | | | | | | | |
| Q3 | | | | | | | |
| Max | | | | | | | |
| CV% | | | | | | | |

AM: Arithmetic Mean; SD: Standard Deviation; Min: Minimum; Q1: 1<sup>st</sup> Quartile; Q3: 3<sup>rd</sup> Quartile; Max: Maximum; GM: Geometric Mean; CV%: Arithmetic CV which is equal to SD/AM\*100.


- Table 14.4.1.2. Descriptive Statistics of Plasma Concentrations of Filgotinib Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease
- Table 14.4.1.3. Descriptive Statistics of Plasma Concentrations of GS-829845 Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease
- Table 14.4.1.4. Descriptive Statistics of Plasma Concentrations of GS-829845 Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease


Table 14.4.1.5. Descriptive Statistics of Plasma Concentrations of Filgotinib Following Once Daily Oral Administration of 200 or 100 mg Filgotinib in Subjects with Moderately to Severely Active Crohn's Disease - Cohort A

| | 2.0 | 10 ma | | | | 10 | 0 | | |
|---|---|---|---|---|---|---|---|---|---|
| | 200 mg | | | | | 100 mg | | | |
| Week 4 predose | Week<br>4<br>0.5-3<br>hr | Week<br>10<br>predose | Week<br>26<br>anytime | Week<br>58<br>predose | Week 4 predose | Week 4<br>0.5-3 hr | Week<br>10<br>predose | Week<br>26<br>anytime | Weel<br>58<br>predos |
| Week 4 predose | 4<br>0.5-3 | 10 | 26 | 58 | Week 4 predose | | 10 | 26 | 5 |
| | Week 4 predose | Week 4 predose 0.5-3 | Week 4 predose 4 Week 10 predose | Week 4 predose 4 Week Week 26 26 anytime | Week 4 predose 4 Week Week Week 10 26 58 26 anytime predose | Week 4 predose 4 | Week 4 predose 4 | Week 4 predose Week Week Week Week Week Week 4 predose Week 4 Week | Week 4 predose 4 |

AM: Arithmetic Mean; SD: Standard Deviation; Min: Minimum; Q1: 1<sup>st</sup> Quartile; Q3: 3<sup>rd</sup> Quartile; Max: Maximum; GM: Geometric Mean; CV%: Arithmetic CV which is equal to SD/AM\*100.

Note: if a sub-study PK sample is scheduled to be collected at the same time as a sparse PK sample, only one sample should be collected.


| Table 14.4.1.6. | Descriptive Statistics of Plasma Concentrations of Filgotinib Following Once Daily Oral Administration of 200 or 100 mg Filgotinib in Subjects with Moderately to Severely Active Crohn's Disease - Cohort B |
|---|---|
| Table 14.4.1.7. | Descriptive Statistics of Plasma Concentrations of Filgotinib Following Once Daily Oral Administration of 200 or 100 mg Filgotinib in Subjects with Moderately to Severely Active Crohn's Disease - Maintenance Study |
| <b>Table 14.4.1.8.</b> | Descriptive Statistics of Plasma Concentrations of GS-829845 Following Once Daily Oral Administration of 200 or 100 mg Filgotinib in Subjects with Moderately to Severely Active Crohn's Disease - Cohort A |
| <b>Table 14.4.1.9.</b> | Descriptive Statistics of Plasma Concentrations of GS-829845 Following Once Daily Oral Administration of 200 or 100 mg Filgotinib in Subjects with Moderately to Severely Active Crohn's Disease - Cohort B |
| Table 14.4.1.10. | Descriptive Statistics of Plasma Concentrations of GS-829845 Following Once Daily Oral Administration of 200 or 100 mg Filgotinib in Subjects with Moderately to Severely Active Crohn's Disease - Maintenance Study |


Table 14.4.2. Descriptive Statistics of Plasma Filgotinib and Metabolite GS-829845 Pharmacokinetic Parameters

Table 14.4.2.1. Descriptive Statistics of Plasma Pharmacokinetic Parameters of Filgotinib Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

| Subject | C <sub>max</sub> | T <sub>max</sub> | Ctau | AUC <sub>0-tau</sub> | CL <sub>ss</sub> /F |
|---|---|---|---|---|---|
| | (ng/mL) | (h) | (ng/mL) | (ng*h/mL) | (L/h) |

N
AM
SD
Min
Median
Max
CV%
GM

AM: Arithmetic Mean; SD: Standard Deviation; Min: Minimum; Max: Maximum; GM: Geometric Mean; CV%: Arithmetic CV which is equal to SD/AM\*100. Note: To estimate AUC<sub>0-tau</sub>, the concentration of 24h post-dose is based on imputed predose value.


| <b>Table 14.4.2.2.</b> | Descriptive Statistics of Plasma Pharmacokinetic Parameters of Filgotinib Following Once Daily Oral |
|---|---|
| | Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with |
| | Moderately to Severely Active Crohn's Disease |

Table 14.4.2.3. Descriptive Statistics of Plasma Pharmacokinetic Parameters of GS-829845 Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

| Subject | Cmax | $T_{max}$ | Ctau | AUC <sub>0-tau</sub> | MRcmax | MRctau | MRauctau |
|---|---|---|---|---|---|---|---|
| | (ng/mL) | (h) | (ng/mL) | (ng*h/mL) | | | |

N

AM

SD

Min

Median

Max

CV%

GM

AM: Arithmetic Mean; SD: Standard Deviation; Min: Minimum; Max: Maximum; GM: Geometric Mean; CV%: Arithmetic CV which is equal to SD/AM\*100. Note: To estimate AUC<sub>0-tau</sub>, the concentration of 24h post-dose is based on imputed predose value.

MRcmax: Metabolic ratio of GS-829845 C<sub>max</sub> / filgotinib C<sub>max</sub> \* (425.51/357.43)

MRctau: Metabolic ratio of GS-829845 C<sub>tau</sub> / filgotinib C<sub>tau</sub> \* (425.51/357.43)

MRauctau: Metabolic ratio of GS-829845 AUC<sub>0-tau</sub> / filgotinib AUC<sub>0-tau</sub> \* (425.51/357.43)


Table 14.4.2.4. Descriptive Statistics of Plasma Pharmacokinetic Parameters of GS-829845 Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

Listing 16.4.1. Individual Plasma Concentrations of Filgotinib and Metabolite GS-829845

Listing 16.4.1.1. Individual Plasma Concentrations of Filgotinib Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

| | Plasma Concentration (ng/mL) over Nominal Time (h) | | | | | | |
|---|---|---|---|---|---|---|---|
| Subject | Pre-dose | 0.5 | 1 | 2 | 3 | 4 | 6 |


- Listing 16.4.1.2. Individual Plasma Concentrations of Filgotinib Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease
- Listing 16.4.1.3. Individual Plasma Concentrations of GS-829845 Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease
- Listing 16.4.1.4. Individual Plasma Concentrations of GS-829845 Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease
- Listing 16.4.2. Individual Plasma Filgotinib and Metabolite GS-829845 Pharmacokinetic Parameters
- Listing 16.4.2.1. Individual Plasma Pharmacokinetic Parameters of Filgotinib Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

| Subject | Cmax | T <sub>max</sub> | Ctau | AUC <sub>0-tau</sub> | CL <sub>ss</sub> /F |
|---|---|---|---|---|---|
| | (ng/mL) | (h) | (ng/mL) | (ng*h/mL) | (L/h) |

Note: To estimate AUC<sub>0-tau</sub>, the concentration of 24h post-dose is based on imputed predose value.


Listing 16.4.2.2. Individual Plasma Pharmacokinetic Parameters of Filgotinib Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

Listing 16.4.2.3. Individual Plasma Pharmacokinetic Parameters of GS-829845 Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

| Subject | Cmax | $T_{max}$ | Ctau | AUC <sub>0-tau</sub> | MRcmax | MRctau | MRauctau |
|---|---|---|---|---|---|---|---|
| | (ng/mL) | (h) | (ng/mL) | (ng*h/mL) | | | |

Note: To estimate  $AUC_{0\text{-}tau}$ , the concentration of 24h post-dose is based on imputed predose value.

MRcmax: Metabolic ratio of GS-829845  $C_{max}$  / filgotinib  $C_{max}$  \* (425.51/357.43) MRctau: Metabolic ratio of GS-829845  $C_{tau}$  / filgotinib  $C_{tau}$  \* (425.51/357.43)

MRauctau: Metabolic ratio of GS-829845 AUC0-tau / filgotinib AUC0-tau \* (425.51/357.43)

Listing 16.4.2.4. Individual Plasma Pharmacokinetic Parameters of GS-829845 Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease


Figure 16.4.3. Individual Subject Plasma Concentration-Time Graphs

Figure 16.4.3.1. Individual Plasma Filgotinib Concentration – Time Profiles
Following Once Daily Oral Administration of 200 mg Filgotinib at
One Visit Between Week 2 and Week 10 in Subjects with
Moderately to Severely Active Crohn's Disease

## **Linear Scale (Mock Figure)**



#### Semi-logarithmic Scale (Mock Figure)



Figure 16.4.3.2. Individual Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease

Figure 16.4.3.3. Individual Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 200 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours

#### **Linear Scale (Mock Figure)**



#### **Semi-logarithmic Scale (Mock Figure)**



Figure 16.4.3.4. Individual Plasma Filgotinib Concentration – Time Profiles Following Once Daily Oral Administration of 100 mg Filgotinib at One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours

Figure 16.4.3.5. Individual Plasma GS-829845 Concentration – Time Profiles
Following Once Daily Oral Administration of 200 mg Filgotinib at
One Visit Between Week 2 and Week 10 in Subjects with Moderately
to Severely Active Crohn's Disease

Figure 16.4.3.6. Individual Plasma GS-829845 Concentration – Time Profiles
Following Once Daily Oral Administration of 100 mg Filgotinib at
One Visit Between Week 2 and Week 10 in Subjects with Moderately
to Severely Active Crohn's Disease

Figure 16.4.3.7. Individual Plasma GS-829845 Concentration – Time Profiles
Following Once Daily Oral Administration of 200 mg Filgotinib at
One Visit Between Week 2 and Week 10 in Subjects with Moderately
to Severely Active Crohn's Disease – 0 to 24 hours

Figure 16.4.3.8. Individual Plasma GS-829845 Concentration – Time Profiles Following Once Daily Oral Administration of 100 mg Filgotinib at

One Visit Between Week 2 and Week 10 in Subjects with Moderately to Severely Active Crohn's Disease – 0 to 24 hours